



# **Reproductive Medicine Network**

Funded by Eunice Kennedy Shriver NICHD

# Males, Antioxidants, and Infertility (MOXI) Trial

Protocol Leader: Anne Z. Steiner, MD, MPH Data and Coordination Leader: Heping Zhang, PhD

Version: 4.0

Prepared by:

The RMN Data Coordination Center

Collaborative Center for Statistics in Science

Yale University School of Public Health

300 George Street, Suite 523

New Haven, CT 06511

(203) 785-5185

Last updated October 12, 2016

# **Protocol Subcommittee**

Group email address: <a href="mailto:rmn.moxi@mailman.yale.edu">rmn.moxi@mailman.yale.edu</a>

| Name | E-mail |
|---------------------------|------------------------------|
| Anne Z. Steiner, MD, MPH | anne_steiner@med.unc.edu |
| Matt Coward, MD | mcoward@med.unc.edu |
| Esther Eisenberg, MD, MPH | eisenbes@mail.nih.gov |
| Stephen A. Krawetz, PhD | steve@compbio.med.wayne.edu |
| Puneet Masson, MD | Puneet.Masson@uphs.upenn.edu |
| Nanette Santoro, MD | nanette.santoro@ucdenver.edu |
| Jim Smith, MD, MS | SmithJF@urology.ucsf.edu |
| Peter Snyder, MD | pjs@mail.med.upenn.edu |
| J. C. Trussell, MD | ictrussell1@verizon.net |
| Heping Zhang, PhD | heping.zhang@yale.edu |

# **Table of Contents**

| 1 | ACRONYMS | 6 |
|----------------|-----------------------------|----|
| 2 | STUDY SYNOPSIS | 8 |
| 2.1 | Objectives | 8 |
| 2.2 | PATIENT POPULATION | 8 |
| 2.3 | STUDY DESIGN | 8 |
| 2.4 | Treatment | 8 |
| 2.5 | PRIMARY OUTCOME | 9 |
| 2.6 | SECONDARY OUTCOME | 9 |
| 2.7 | INTERNAL PILOT | 9 |
| 2.8 | STATISTICAL ANALYSIS | 9 |
| 2.9 | REGULATORY COMPLIANCE | 10 |
| 3 | BACKGROUND AND SIGNIFICANCE | 11 |
| 3.1 | BACKGROUND | 11 |
| 3.2 | SIGNIFICANCE | 13 |
| 3.3 | INNOVATION | 14 |
| 4 | OBJECTIVES | 15 |
| 4.1 | Primary Aim | 15 |
| 4.2 | SECONDARY AIM | |
| 4.3 | TERTIARY AIMS | |
| 4.4 | INTERNAL PILOT | 15 |
| 5 | STUDY DESIGN | 17 |
| 5.1 | OVERVIEW AND SCHEMA | 17 |
| 5.2 | STUDY POPULATION | |
| 5.2.1 | Inclusion Criteria | |
| 5.2.2 | Exclusion Criteria | |
| 5.2.3 | Study Termination Criteria | |
| 5.2.4 | Rationale for Criteria | 19 |
| 5.3 | RECRUITMENT | 20 |
| 5.4 | SCREENING | 21 |
| 5.5 | INFORMED CONSENT | |
| 5.6 | TREATMENT PROTOCOLS | |
| 5.6.1 | J | |
| 5.6.2 | | |
| 5.6.3 | | |
| 5.6.4 | | |
| 5.7 | STUDY FLOW: | |
| 5.7.1 | Screening: | |
| 5.7.2 | | |
| 5.7.3 | | |
| 5.7.4 | | |
| 5.7.5 | | |
| 5.7.6 | | |
| 5.7.7 | | |
| 5.7.8<br>5.7.9 | | |
| 5.7.9 | · . | |
| 6 | DATA COLLECTION | 32 |

| 6.1 | SPECIMEN COLLECTION, PROCESSING, AND SHIPMENT | |
|---|---|---|
| 6.1.1 | Semen Collection | 32 |
| 6.1.2 | Semen analysis | 33 |
| 6.1.3 | DNA integrity testing | 33 |
| 6.1.4 | SCSA | 33 |
| 6.1.5 | TUNEL | |
| 6.1.6 | COMET | |
| 6.2 | COMPLIANCE | |
| 6.2.1 | | |
| 6.3 | DIETARY ASSESSMENT | |
| 6.4 | MALE URINARY TESTING FOR ENVIRONMENTAL CONTAMINANTS | 35 |
| 6.5 | STRESS BIOMARKER TESTING | 35 |
| 6.6 | MALE LABORATORY TESTING (CENTRAL CORE LABORATORY) | |
| 6.7 | MALE SUNSCREEN USAGE | |
| 6.8 | QUALITY OF LIFE (QOL) MEASURES | |
| 6.9 | EARLY PREGNANCY ULTRASOUND | |
| 6.10 | ASCERTAINMENT OF PREGNANCY OUTCOMES | |
| 6.11 | Pregnancy Registry | |
| 6.12 | BIOLOGIC REPOSITORY | |
| 6.13 | CENTRAL CORE LABORATORY | |
| 7 | DATA ANALYSIS | 38 |
| 7.1 | INTERNAL PILOT | 38 |
| 7.2 | PRIMARY AND SECONDARY OUTCOMES | |
| 7.3 | SAMPLE SIZE AND STATISTICAL POWER | |
| 8 | TECHNICAL ASPECTS | 42 |
| 8.1 | REPORTING ADVERSE EVENTS | 42 |
| 8.2 | DATA COLLECTION AND MANAGEMENT (INCLUDING QUALITY ASSURANCE/COMPLIANCE MEASURES) | |
| 8.2.1 | Data Entry and Forms | |
| 8.2.2 | Features of Data Management System | |
| 8.2.3 | Data Security | |
| 8.2.4 | | |
| 8.3 | STUDY MONITORING | |
| 8.4 | DATA AND SAFETY MONITORING BOARD | |
| 8.5 | REPORTING | |
| 8.6 | OBLIGATION OF THE INVESTIGATOR | |
| 8.6.1 | IRB Review | |
| 8.6.2 | | |
| 8.7 | REGULATORY REQUIREMENTS | |
| 8.8 | PROTOCOL AMENDMENTS. | |
| 8.9 | TIMELINE | |
| 9 | RMN PUBLICATIONS POLICY | 51 |
| 9.1 | MAIN STUDY | 51 |
| 9.1.1 | Major Publications | |
| 9.1.2 | Minor Publications | |
| 9.2 | ANCILLARY STUDY | |
| 9.2.1 | Publication Policy on Ancillary Papers | |
| 9.3 | PILOT STUDY | |
| 9.4 | RELATED PUBLICATIONS. | |
| 9.5 | OUTSIDE STUDIES | |
| 9.6 | Presentations | |
| 9.7 | TIMELINES | |
| 9.8 | NICHD CLEARANCE | |

| 10 | REFERENCES | 59 |
|---|---|---|
| 11 | INFORMED CONSENT | 65 |
| 11.1 | Informed Consent Template – Male Partners | |
| 11.2 | INFORMED CONSENT TEMPLATE – FEMALE PARTNERS | |
| 12 | APPENDIX A: MALE MEDICAL HISTORY QUESTIONNAIRE | |
| 13 | APPENDIX B: FEMALE MEDICAL HISTORY QUESTIONNAIRE | |
| 14 | APPENDIX C: LIST OF PROHIBITED CONCOMITANT MEDICATIONS | |
| 15 | APPENDIX D: REVIEW OF ANTIOXIDANT FORMULATIONS | |
| 15.1<br>15.2 | COMMERCIALLY AVAILABLE FORMULATIONS | |
| 16 | APPENDIX E: RISK FACTORS FOR GENETIC DISORDERS | 138 |
| 17 | APPENDIX F: FEMALE SEXUAL FUNCTION INDEX (FSFI) | 140 |
| 18 | APPENDIX G: SF-12V2 HEALTH SURVEY | 145 |
| 19 | APPENDIX H: PATIENT HEALTH QUESTIONNAIRE (PHQ-9) | 148 |
| 20 | APPENDIX I: FERTIQOL | 150 |
| 21 | APPENDIX J: EPWORTH SLEEPINESS SCALE | 151 |
| 22 | APPENDIX K: STOP BANG QUESTIONNAIRE | 152 |
| 23 | APPENDIX L: FEMALE SEXUAL DISTRESS SCALE (FSDS- REVISED 2005) | 153 |
| 24 | APPENDIX M: INTERNATIONAL INDEX OF ERECTILE FUNCTION (IIEF) | 154 |
| 25 | APPENDIX N: DIET HISTORY QUESTIONNAIRE II | 157 |
| 26 | APPENDIX O: AUTOMATED SELF-ADMINISTERED 24-HOUR RECALL (ASA24) | 197 |
| 27 | APPENDIX P: QADAM QUESTIONNAIRE | 208 |
| 28 | APPENDIX Q: PSYCHOSEXUAL DAILY QUESTIONNAIRE | 209 |
| 29 | APPENDIX R: SUN EXPOSURE AND BEHAVIOUR INVENTORY (SEBI V2) | |
| 30 | APPENDIX S: INVESTIGATOR SIGNATURE OF AGREEMENT | 214 |
| 31 | APPENDIX T: DATA AND SAFETY MONITORING PLAN | |
| Figur | re 1: Schema for the Participation Timeline | 17 |
| Figur | re 2: SAE flowchart | 44 |
| Table | e 1: Overview of Timing and Content of Data Collection for Primary Cohort | 32 |
| | e 2: Sample size estimates under a variety of assumptions | |
| | 23: Power for subgroup analyses | |
| | e 4: Types of Serious Adverse Events and Their Reporting Requirements | |
| | e 6: RMN Publication Authorship | |
| | e 7: Authorship Order of the RMUs and Outside Sites | |

# 1 Acronyms

| Assisted Reproductive Technologies | ART | Intrauterine Insemination | IUI |
|---|---|---|---|
| Advisory Board | АВ | Investigational New Drug | IND |
| American Congress of Obstetricians and Gynecologists | ACOG | National Institute of Child Health and<br>Human Development | NICHD |
| Assessment of Multiple Intrauterine Gestations from Ovarian Stimulation | AMIGOS | Ovarian Hyperstimulation Syndrome | OHSS |
| Clinical Report Form | CRF | Principal Investigator | PI |
| Clomiphene Citrate | СС | Progesterone | P4 |
| Code of Federal Regulations | CFR | Protected Health Information | PHI |
| Data and Safety Monitoring Board | DSMB | Quality Control | QC |
| Data Coordination Center | DCC | Randomized Controlled Trial | RCT |
| Deoxyribonucleic Acid | DNA | Reactive oxygen species | ROS |
| DNA fragmentation index | DFI | Reproductive Medicine Network | RMN |
| Ectopic Pregnancy | EP | Reproductive Medicine Unit | RMU |
| Follicle Stimulating Hormones | FSH | Serious Adverse Event | SAE |
| Food and Drug Administration | FDA | Single cell gel electrophoresis | Comet |
| Health Insurance Portability and Accountability Act | HIPAA | Sperm Chromatin Structure Analysis | SCSA |
| Human Chorionic Gonadotropin | hCG | Terminal Deoxynucleotide Transferase-<br>mediated dUTP Nick-end Labeling | TUNEL |

| Human Investigation Committee | ніс | Time to Conceive | ттс |
|---|---|---|---|
| Identification | ID | Total and Free Testosterone | T, FT |
| In Vitro Fertilization | IVF | Ultrasound | U/S |
| Institutional Review Board | IRB | University of North Carolina | UNC |
| Intracytoplasmic sperm injection | ICSI | | |

# 2 Study Synopsis

## 2.1 Objectives

The objective of the Males, Antioxidants, and Infertility (MOXI) Trial is to examine whether treatment of infertile males with an antioxidant formulation improves male fertility. The central hypothesis is that treatment of infertile males with antioxidants will improve sperm structure and function, resulting in higher fertilization rates and improved embryo development, leading to higher pregnancy and live birth rates. Findings from this research will be significant in that they will likely lead to an effective, non-hormonal treatment modality for male infertility. An effective treatment for men would also reduce the treatment burden on the female partner, lower costs, and provide effective alternatives to couples with religious or ethical contraindications to ART. If antioxidants do not improve pregnancy rates, but do improve sperm motility and DNA integrity, they could allow for couples with male factor infertility to use less intensive therapies such as intrauterine insemination. Male fertility specialists currently prescribe antioxidants based on the limited data supporting their use. A negative finding, lack of any benefit, would also alter current treatment of infertile males.

# 2.2 Patient population

The population will consist of 790 heterosexual couples, who have been attempting to conceive for ≥12 months, recruited from the Reproductive Medicine Network (RMN) clinical sites and their surrounding communities over a two-year period.

## 2.3 Study design

This will be a multi-center, randomized, placebo-controlled trial of antioxidant formulation, ConceptionXR Motility Support Formulation by Theralogix ("ConceptionXR") for the male partner. The randomization scheme will be stratified by participating site. The study will contain an internal pilot study.

## 2.4 Treatment

790 male subjects will be equally randomized via computer-generated randomization to receive:
A) ConceptionXR Motility Support Formulation (Theralogix) containing an antioxidant combination including Vitamin C, Vitamin E, folic acid, selenium, zinc, and L-carnitine by oral ingestion twice daily or B) a placebo by oral ingestion twice daily in a double-blinded fashion. Treatment assignments will be randomized within each site by varying block size design. Treatment will occur for a minimum of 3 months and a maximum of 6 months. Couples will attempt to conceive naturally during the first 3 months and with clomiphene citrate with intrauterine insemination in months 4 through 6.

## 2.5 Primary outcome

The primary outcome will be live birth rate following up to 6 months of treatment with antioxidants as compared to placebo.

# 2.6 Secondary outcome

The secondary outcomes will be pregnancy rate, miscarriage rate, time to pregnancy, and semen parameters and DNA fragmentation at 3 months of treatment with an antioxidant as compared to placebo.

#### 2.7 Internal Pilot

We will be conducting an internal pilot study with a three-fold objective. The objective of the internal pilot is 1) to determine the distribution of the semen abnormalities in the study population, 2) to examine the effect of our antioxidant formulation on male semen parameters and DNA integrity at 3 months of treatment compared to controls, and 3) to determine the feasibility of the proposed recruitment paradigm. The first 120 men enrolled in the MOXI trial will be included in the internal pilot. Assuming we fail to reject the null hypothesis that motility and DNA fragmentation percentage do not differ between the two treatment groups (antioxidant and placebo) at 3 months, the MOXI trial will stop enrolling subjects. Assuming we reject the null hypothesis that motility and DNA fragmentation percentage do not differ between the two treatment groups (antioxidant and placebo) at 3 months, the MOXI trial will continue. As the primary outcome will not be analyzed for the pilot, adjustments in significance levels will not be required for the primary analyses. Feasibility will be assessed by recruitment pace. We anticipate that the pilot enrollment will be completed by 6 months. If we fail to meet this pace, the recruitment strategies may need to be altered or the study stopped at the conclusion of the pilot.

# 2.8 Statistical Analysis

The primary outcome is a live birth resulting from a pregnancy that is conceived within the 6 months from initiation of treatment. Live birth is defined as a delivery of a live infant after 20-weeks gestation. Secondary outcomes include pregnancy, defined by a positive home pregnancy test within the 6 months of treatment. We will conduct an intent-to-treat analysis. Cumulative incidence of live birth and pregnancy will be compared between those couples randomized to antioxidants and those couples randomized to placebo. In addition, discrete-time hazard models will be used to compare time-to-pregnancy between the two treatment groups. Subsequent subgroup analyses will be conducted to assess for effect modification by type of baseline sperm abnormality (asthenospermia, high DNA fragmentation, oligospermia).

After transformations, if needed, semen parameter measures will be analyzed using a generalized linear mixed model (including random effects for site if necessary) or generalized linear model (if fixed effects for site are used). Interaction terms will be used to determine the

extent to which the change in semen parameter measures differs by type of baseline sperm abnormality (asthenospermia, high DNA fragmentation, oligospermia). If there is evidence of effect modification, change estimates will be determined for each type of baseline sperm abnormality.

For the power analysis, we assume live birth rates of 35% in the antioxidant group and 25% in the control group, and 17% drop-out. Under these assumptions, the power by using a two-sided chi square test at  $\alpha$ =0.05 would be 0.80.

# 2.9 Regulatory Compliance

The DCC is working with the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) to ensure that clinical study data and regulatory requirements are met regarding the Food and Drug Administration (FDA) code for federal regulations and Investigational New Drug (IND) submissions.

This trial is registered on http://www.clinicaltrials.gov (NCT # 02421887), and has been issued IND # 125753.

# 3 Background and Significance

# 3.1 Background

A variety of pathologic conditions including infection (1), varicocele (2), and cancer (3), along with environmental exposures including organic chemicals (4), pharmaceuticals, smoking (5), and radiation appear to increase oxidative stress, measured as reactive oxygen species (ROS), in semen. The sperm plasma membrane and nuclear genomes are highly susceptible to damage due to ROS due to high levels of polyunsaturated fatty acids, deficiencies in intracellular antioxidant enzymes, and limited capacity for DNA repair in sperm (6). ROS cause lipid peroxidation and thereby structural modifications to the membrane, which have been shown to interfere with sperm motility, the acrosome reactions, and sperm-oocyte fusion (7). ROS damage the nuclear and mitochondrial genome by causing single and double DNA breaks, chemical modifications of bases, DNA crosslinks, and DNA protein crosslinks (8). Damaged DNA may be repaired by endogenous repair mechanisms; however, if these are overwhelmed, the damaged DNA will be integrated into the embryo. It has been proposed that this damaged DNA will impair embryonic development, lead to pregnancy loss, or result in birth defects or morbidity in the offspring.

Given that ROS negatively affect the sperm plasma membrane, which is important for fertilization, and sperm DNA, which is important for normal embryonic and fetal development, it is logical that ROS will diminish a sperm's capacity to fertilize or lead to impaired embryo development. Clinically this would be observed as reduced fertility and greater pregnancy loss in female partners of men with elevated levels of ROS. While ROS are not commonly measured in semen, ROS damage to sperm, as measured by loss of motility and DNA fragmentation, can be quantified. Sperm motility can be measured using a standard semen analysis. DNA integrity is measured using a number of assays including Terminal Deoxynucleotide Transferase-mediated dUTP Nick-end Labeling (TUNEL), Sperm Chromatin Structure Analysis (SCSA), and single cell gel electrophoresis (Comet).

In fact, previous studies have shown that low sperm motility and high DNA fragmentation, as measured by the SCSA, are associated with a longer time-to-pregnancy among couples trying to conceive (9). Sperm motility lower than 32% is associated with 2.5 times the odds of infertility (10). Evenson et al. found that couples that did not conceive had 30% more DNA fragmentation compared to couples that conceived within 3 months of attempt (9). DNA fragmentation was also greater among those couples that did not conceive with intrauterine insemination and intracervical insemination compared to those that did conceive (11-13). DNA fragmentation levels have not consistently been associated with live birth rates following ART. Some studies have shown that fertilization and pregnancy rates are lower with high DNA fragmentation (14-20), while others have not shown an association (11, 17, 21, 22). These discrepancies may be

due to the variety of assays used to measure DNA fragmentation, the use of ICSI (ROS plasma membrane damage may be mitigated with intracytoplasmic sperm injection) (13-15, 23-25), and the variety of cut-off values used to define high DNA fragmentation. In addition, sperm preparation techniques may decrease the percentage of sperm with fragmented DNA in the aliquots of sperm used for *in vitro fertilization* (26).

Vitamin C, E, and other naturally occurring antioxidants are low molecular mass ROS scavengers found in semen (27). Low levels of seminal vitamin C are associated with poor semen quality (27). Seminal concentrations of antioxidants are lower in men with infertility compared to fertile men (28-30). As antioxidants appear to lower ROS and ROS appear to negatively affect fertility, antioxidants have been proposed as a treatment for male factor infertility.

The limited data suggest that antioxidants improve sperm motility and reduce DNA fragmentation. A previous observational study showed that a health conscious diet is associated with a decrease in sperm DNA fragmentation, suggesting that natural antioxidants are beneficial to sperm (31). However, another observational study using food frequency questionnaires failed to find an association between any antioxidant measure and DNA fragmentation, perhaps because the cohort was comprised of healthy volunteers (32). Studies of supplements have tended to show an improvement in semen parameters with the use of antioxidants. Benefits of Vitamin C (33), selenium (34), N-acetylcysteine (35), L-carnitine (36), and Zinc (37) on sperm motility have been seen after 3 months of treatment. Unfortunately, most of these studies have been small and heterogeneous. While most studies included only infertile men, some included those with normal baseline semen parameters and some with abnormal baseline semen parameters. Only one clinical trial has compared DNA integrity between men treated with antioxidants (Vitamin C and Vitamin E) and a control group (38). This study of 64 men found that after 2 months of treatment, men who received antioxidants had on average 14% (10.1-17.5%) less fragmented sperm. DNA integrity needs to be assessed in addition to traditional semen parameters as a significant number of men will have high levels of DNA fragmentation despite a normal semen analysis (39-41).

The paternal genome is thought to be activated between cleavage stage and blastocyst stage during embryonic development. It has been suggested that sperm DNA fragmentation will alter embryonic development in these later stages (42). Aberrant embryo development could lead to miscarriage or subsequent congenital abnormalities. Meta-analyses of previous studies examining the association between DNA fragmentation and miscarriage suggest that high DNA damage as measured by TUNEL assay is associated with an increase in the risk of miscarriage (Mantel-Hansel Risk ratio (random effects model) 3.94 (95% CI 2.54, 6.32)(43). The association was not as strong when the SCSA was used as the measure of DNA fragmentation (RR 1.47, 95% CI 1.04, 2.09). Only one underpowered study examined the relationship between miscarriage and DNA fragmentation among couples conceiving naturally (9). It is impossible to determine

the amount of DNA fragmentation in the fertilizing sperm *in vivo* and *in vitro* as assays to assess sperm DNA integrity preclude their use. Thus it is assumed that the overall percentage of sperm with DNA damage in a given ejaculate reflects the probability that the DNA from the sperm that fertilized the egg was damaged. It is possible that the probability of an embryologist selecting a sperm with DNA fragmentation to fertilize an oocyte *in vitro* would differ from the probability that a sperm with DNA fragmentation would fertilize an oocyte *in vivo*.

Clinical studies of the use of antioxidants in the treatment of male infertility have been encouraging. A recent meta-analysis found that use of antioxidants by males with infertility was associated with 4.85 times the odds (95% CI 1.92-12.24) of live birth following ART compared to men who did not use antioxidants (44). While these findings are encouraging, they fail to provide a definitive answer as to whether antioxidants improve male fertility. The meta-analysis included 3 studies for a total of 214 participants and the quality of the evidence was graded as low. These studies examined the antioxidants vitamin E (45, 46) and zinc (47), while studies using pregnancy as an outcome have shown L-carnitine to be promising (36, 48). Finally, these studies all used antioxidants in combination with ART; it is certainly possible that the response to antioxidants will differ with *in vivo* fertilization.

## 3.2 Significance

Although clinical trials suggest that antioxidants have a positive effect on sperm motility, DNA integrity, and pregnancy rates in couples undergoing assisted reproductive technologies, there are significant gaps in our knowledge of their impact on fertility (44). Gaps exist due to limitations in existing literature. 1) A variety of antioxidants at varying doses and duration have been used, precluding a strong conclusion as to whether a specific regimen is beneficial. 2) Most studies have had small sample sizes, usually less than 50 subjects. 3) Studies have utilized heterogeneous populations, limiting ability to combine results of multiple studies. 4) Most studies have used changes in semen parameters or DNA integrity as the endpoint, rather than clinical outcomes. 5) Studies have used antioxidants in conjunction with *in vitro* fertilization with intracytoplasmic sperm injection (ICSI) when measuring effectiveness. This has precluded the possibility of studying antioxidant effects on *in vivo* fertilization, which relies on normal sperm function. Our proposed study will improve generalizability, but still allow for sufficient power to determine benefit among subgroups, and will look at reproductive endpoints including pregnancy, miscarriage, and live birth.

Findings from this research will be significant in that they will likely lead to an effective, natural treatment modality for men with abnormal sperm. An effective, inexpensive, non-invasive treatment for male subfertility would be of significant benefit, as no such treatment has been clinically validated. An effective treatment for men would also reduce the treatment burden on the female partner, lower costs, and provide effective alternatives to couples with religious or ethical contraindications to ART. Even if antioxidants are found not to be of benefit to any

subgroup, this research will help us better understand the reproductive impact of sperm DNA integrity, leading to treatments that could improve fertility, pregnancy outcomes, and offspring health.

Another important possible benefit of antioxidant use in males is their potential to reduce offspring morbidity. Increasing evidence highlights a link between paternal age and offspring morbidities including autism (49), schizophrenia (50), and sporadic autosomal dominant disorders (51). It is possible that these disorders may be attributable to DNA fragmentation due to increased ROS in aging males (15, 52). While the proposed study will not directly address the therapeutic benefits of antioxidants in the prevention of these morbidities, it will address a potential mechanism and possibly suggest a preventative therapy by providing information about relationships between chronological age, DNA fragmentation, and relative effectiveness of antioxidant therapy in treating DNA fragmentation.

#### 3.3 Innovation

This proposal is innovative in that it 1) focuses on male infertility, 2) examines both primary clinical outcomes such as live birth, and intermediate outcomes, such as semen parameters, 3) seeks to discover a cure for male infertility that does not require ART, and 4) will use the highest quality study design, an adequately powered, randomized controlled trial. While biologic evidence supports the hypothesis that antioxidants would improve male fertility, our unique study design will allow the RMN to ultimately determine if antioxidants improve male fertility without the use of ART.

# 4 Objectives

# 4.1 Primary Aim

Our primary aim is to compare live birth rates in infertile couples (≥12 months of infertility) following up to 6 months of male treatment with antioxidants, as compared to placebo. This is a randomized, multi-center trial in which couples receive clomiphene citrate and IUI in the second half of treatment. The primary outcome measure will be cumulative incidence of live birth of pregnancies conceived following up to 6 months of male treatment with the antioxidant formulation or placebo.

# 4.2 Secondary Aim

We will assess secondary outcomes including cumulative pregnancy rates with pregnancy defined as a positive pregnancy test, clinical pregnancy rates defined as presence of a fetus with cardiac activity, miscarriage rate, defined as the loss of a pregnancy prior to 20-weeks gestation, and time to pregnancy. In addition, we will examine changes in semen parameters and DNA fragmentation at 3 months of treatment.

## 4.3 Tertiary Aims

Subsequent subgroup analyses will be conducted to assess for effect modification by type of baseline sperm abnormality (oligospermia, asthenospermia, high DNA fragmentation). Additional questions that can be addressed with this cohort could include:

- 1. Do high levels of DNA fragmentation increase the risk of miscarriage?
- 2. Does DNA fragmentation increase with paternal age?
- 3. Does DNA fragmentation increase time to pregnancy (and decrease fecundability)?
- 4. How do SCSA and TUNEL assays for DNA fragmentation compare?

#### 4.4 Internal Pilot

While there are a number of small randomized controlled trials showing that antioxidants improve semen parameters and a few that show that they increase pregnancy rates following ART, the studies vary tremendously in their choice of antioxidant and formulation. There are a number of commercial products marketed to improve male fertility. No trials have been published in peer-reviewed journals using any of these formulations. We have chosen a commercial antioxidant formulation, which includes the antioxidants that appear to improve semen parameters based on the existing literature. For this reason, we will be conducting an internal pilot study.

The objective of the internal pilot is to examine the effect of our antioxidant formulation, ConceptionXR, on male semen parameters and DNA integrity at 3 months of treatment compared to controls. We hypothesize that motility will be significantly higher and DNA fragmentation

significantly lower among those men treated with antioxidants compared to placebo. A secondary objective of the internal pilot is to determine the feasibility of recruitment into a male fertility study. A tertiary objective, which will only be assessed if we fail to meet the primary and secondary objectives of the internal pilot, would be to compare live birth rates and pregnancy rates.

# 5 Study Design

#### 5.1 Overview and Schema

To achieve our objective, we will conduct the Males, Antioxidants, and Infertility (MOXI) Trial, a randomized controlled trial of the effect of antioxidants on semen parameters and male fertility. Couples will be recruited from the clinics and will undergo a screening visit. At the female screening visit, she will provide consent, complete a questionnaire and any necessary screening tests, provide a blood sample, and complete a food frequency questionnaire. At the male screening visit, he will provide consent, complete a questionnaire, provide a semen sample, if no semen analysis within the past 6 months is available, and complete a food frequency questionnaire. A total of 790 couples will be enrolled. At the first study visit the male partner will provide a semen sample and complete a dietary assessment. The male will be randomized to the placebo or antioxidant arm. Treatment will follow for 3 months. If the couple has not conceived, treatment will continue for up to an additional 3 months and the female will receive up to 3 cycles of clomid and IUI. Throughout the pre-conception window, women will use ovulation predictor kits and check a home pregnancy test with missed menses. Men will provide a semen sample after 3 months of treatment. Compliance will be assessed at 1, 3, and 6 months. An ultrasound will be performed between 7 and 9 weeks gestation and pregnancy outcomes determined.



Figure 1: Schema for the Participation Timeline

## 5.2 Study Population

#### 5.2.1 Inclusion Criteria

#### Couple

- 12 or more months of infertility (primary or secondary) for couples with female partner under 35. 6 or more months of infertility (primary or secondary) for couples with female partner 35 years of age or older.
- Heterosexual
- Cohabitating and able to have regular intercourse

#### Male:

- ≥ 18 years of age
- At least one abnormal semen parameter on a semen analysis within the past
   6 months:
  - Sperm concentration ≤15 Million/ml
  - o Total motility ≤40%
  - Normal morphology (Kruger) ≤4%
  - DNA fragmentation (SCSA, DNA fragmentation index) >25%

## Female:

- ≥18 years of age and ≤40 years of age
- For women ≥ 35 years of age, evidence of normal ovarian reserve as assessed by menstrual cycle day 3 (+/-2 days) FSH ≤10 IU/L with estradiol ≤ 70 pg/mL, AMH ≥ 1.0 ng/mL, OR antral follicle count >10 within one year prior to study initiation.
- Evidence of at least one patent fallopian tube as determined by an HSG or laparoscopy showing at least one patent fallopian tube or a saline infusion sonogram showing spillage of contrast material. OR An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or tubal disease or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
- Regular cycles defined as ≥25 days and ≤35 days in duration
- Evidence of ovulation including biphasic basal body temperatures, positive ovulation predictor kits, or progesterone level ≥3 ng/ml.

#### 5.2.2 Exclusion Criteria

## Couple:

- Previous sterilization procedures (vasectomy, tubal ligation). The prior procedure may affect study outcomes.
- Planning in vitro fertilization in the next 6 months

# Male:

- Sperm concentration < 5 million/mL on screening semen analysis</li>
- Current use of a medication or drug that would affect reproductive function or metabolism (see Appendix C for list)
- Current multivitamin or herb use (requires 1-month wash-out)
- Current serious medical illnesses, such as cancer, heart disease, or cirrhosis
- Seizure disorder
- Current use of anticoagulants
- Untreated hypothyroidism
- Uncontrolled diabetes mellitus

#### Female:

- History of radiologic or surgically confirmed moderate to severe endometriosis
- Body mass index >35 kg/m<sup>2</sup>
- Currently pregnant
- History of polycystic ovarian syndrome
- Current serious medical illnesses, such as cancer, heart disease, or cirrhosis
- History of systemic chemotherapy or pelvic radiation
- Current use of a medication or drug that would affect reproductive function or metabolism (see Appendix C for list)

## 5.2.3 Study Termination Criteria

- 1. Development or suspicion of an allergic or serious adverse reaction to any of the medications in the study
- 2. Non-compliance with study medications and/or protocol
- 3. Cessation of attempts to conceive
- 4. Assisted reproductive technology, outside of study related procedures

## 5.2.4 Rationale for Criteria

Only couples with no known female fertility problems will be eligible (\*no known endometriosis or polycystic ovarian syndrome) as this is a study of male infertility. Women must be ovulatory as this study aims to focus on male fertility. Men on anticoagulants will be excluded, as vitamin E is thought to interact with anticoagulants increasing the risk of bleeding.

We are restricting the study to couples that have been trying to conceive for at least 12 months and men with abnormal semen parameter(s) as this is a study of couples with male infertility. Abnormal semen parameters were defined by the 5<sup>th</sup> percentile lower reference limit for semen parameters from fertile men whose partners had a time-to-pregnancy of 12 months or less based on the WHO population study (53) and the SCSA time-to-pregnancy study (9). We are restricting to female partners less than 35 years of age, or between 35 and 38 years of age with normal measures of ovarian reserve, to minimize the likelihood of reduced fertility due to reproductive aging.

Our exclusion criteria include a lower limit for sperm count. Men with very low sperm counts are more likely to have hypogonadism or obstruction and would be unlikely to benefit from antioxidants. Approximately 32% of males between the ages of 31 and 50 take a daily multivitamin (54). Multivitamin use is more frequent among those with more education, higher incomes, healthier lifestyles and diets, and lower body-mass indexes (55). For this reason, exclusion of men on vitamins 1) could possibly lead to selection bias and 2) might not be feasible. Thus the inclusion criteria call for a 1-month washout period for those men taking vitamins.

#### 5.3 Recruitment

A total of 790 men will be recruited over a 2-year period (approximately 30 men per month). We will recruit subjects using methods previously proven effective in AMIGOS, which enrolled a similar study population.

## Hospital/Local Health Care Referrals

Subjects will be recruited at each site from individual practice(s) as well as faculty/resident clinics. Ongoing contact with practice and faculty members as well as with residents will be made by the investigators and coordinators, reminding them of the inclusion criteria, importance of the study, etc. In addition, the investigators will describe the study to members of other departments in the hospital, primarily family practice, medical endocrinology, urology, and gynecology who also see and treat these patients. Contact with local physicians will be made and/or grand rounds will be given to disseminate information about the study.

# Local Publicity Office

Investigators will meet with their local Public Relations offices and plan a news release about the study. They will also make themselves available for any newspaper, radio, or TV stories that may increase public awareness of the study. The full gamut of local media sources should be utilized. Often there is greater yield with more extensive coverage in smaller local outlets as opposed to brief mentions in outlets with larger circulation. News release will mention the uniqueness of the study, which may improve male fertility treatment.

#### **Local Advertisements**

Advertisements will be placed in local newspapers and will be continued on a regular basis if response is good.

## Contact with infertility support groups

Contact will be made with both national and local support groups to spread information about the study through informational brochures and/or participation in local meetings. The American Infertility Association also may be helpful in promoting awareness of this study.

## National Professional Organizations

Contact will be made with the publicity office of The American Society for Reproductive Medicine, and other potentially helpful organizations to solicit their support and potential informational releases.

#### Web sites

The study will be prominently displayed on the RMN web site. Additionally, each RMN center should have a web page devoted to this study with general as well as contact information. Information should also be available at the NICHD web site with links to each RMN center. An ad should also be placed at "Center Watch" on the web.

#### National Advertising

We would consider placing a trial ad in the health section of a select or a series of selected national publications with all of our local numbers/contacts.

#### IRB Approval

It is expressly acknowledged that all informational material that could be construed to be advertising will be approved by the appropriate IRB prior to dissemination.

#### 5.4 Screening

Couples will be screened through a 3-part process. The first step will be a review of medical records to assess for potential eligibility, when recruiting from the clinic.

Both the female and the male partner will need a screening visit; however, these can be scheduled at the same time. The screening visit will be conducted by the study coordinator and will include questionnaires and laboratory testing. The screening visit will not require physician participation, unless a physical exam is needed. Eligibility will be determined by review of responses to the questionnaire and results of the laboratory testing, and review of medical records.

## 5.5 Informed Consent

We will obtain a limited waiver of HIPAA authorization to allow us to access and use protected health information to review eligibility criteria and contact potential subjects. Female written consent including HIPAA is obtained at the screening visit for the female visit prior to any blood draws or questionnaires. A medical records release form will be obtained at the pregnancy ultrasound. Male written consent and HIPAA will be obtained at the male screening visit prior to the semen analysis and completion of questionnaires. Both males and females will be asked to sign an optional consent form for storage of de-identified residual samples (semen, blood, and data).

Randomization, Allocation, Masking: A total of 790 men will be randomized to one of two treatment groups. The randomization scheme will be generated using a computer generated random number sequence in randomly varying blocks of 4 and 6. The allocation assignments will

be managed by the data coordinating center allowing for concealment. Allocation will be 1:1 stratified by site and female age (<35 years and ≥35 years of age).

The site investigator will be provided a password protected account for a web-based secured randomization service. At the first study visit the investigator or designee will login in order to randomize a patient into the trial. The system will query the site for patient eligibility information. If the patient is eligible, the site will be provided with a patient identifier and a study kit number. The Study Coordinator at each site will be responsible for storing, dispensing, and performing pill/vial counts on the study medications.

#### 5.6 Treatment Protocols

ConceptionXR and placebo will be provided in similar packages. Package will state the study name but will not reveal the allocation assignment. The packages will be stored at room temperature (58-80° F). Each participant will be assigned 3 packages. Package 1 will contain a 30-day supply of treatment; package 2, a 60-day supply, and package 3, a 90-day supply.

## 5.6.1 *Antioxidant formulation*

The antioxidant formulation, ConceptionXR Motility Support Formula includes a combination of antioxidants: Vitamin C, Vitamin E, folic acid, selenium, L-carnitine, zinc, and lycopene, a carotenoid with antioxidant properties. The formulation also includes just one other "active" ingredient, Vitamin D. Men will take 2 pills (one in tablet form, one in capsule form) by mouth twice a day. Each antioxidant selected has been previously studied in a randomized controlled trial and found to positively impact sperm structure or function and/or pregnancy rates following assisted reproductive technology. This commercial formulation was selected based on its antioxidant formulation. Our review of the medical literature found that the above listed antioxidants have data to support their use.

Vitamin C: The total daily dosage of Vitamin C will be 500 mg. Commercial products include Vitamin C in the form of ascorbic acid at doses of 60 to 5000 mg. Randomized controlled trials (all with combination formulations) have included dosages ranging from 10 to 1000 mg (33, 34, 37, 38, 56-58). In general, Vitamin C is not used alone but in combination with vitamin E, as it appears to enhance the anti-oxidant properties of Vitamin E. The tolerable upper intake level for vitamin C is 2000 mg per day.

Vitamin E: The total daily dosage of Vitamin E in the form of d-alpha tocopheryl succinate will be 400 IU. Vitamin E has been shown to improve pregnancy rates following IVF in small randomized controlled trials (45, 46). Vitamin E also has been shown to reduce DNA fragmentation (38) and increase sperm motility at 6 months (46). Commercial formulations include a daily dosage of 150 IU to 400 IU. Randomized trials include doses ranging from 22.5 IU to 1500 IU (34, 37, 38, 45, 46, 56, 58-60). The lower doses were found in combination pills.

In general, the RCTs of Vitamin E and male fertility have tended to use higher doses than we propose. However, Vitamin E will be just one of multiple antioxidants. Second, an RCT of almost 15,000 healthy men over 50 years of age showed that 400 IU of synthetic vitamin E use was associated with a significant increased risk of hemorrhagic stroke over 8 years of treatment (61). It should be noted that the men in the MOXI trial will be, on average, younger and will take the vitamin for a short interval (at most 6 months). In another trial, the SELECT trial, of men over age 50, synthetic vitamin E at 400 IU/day for 5.5 years was found to increase the risk of prostate cancer 1.5 years after cessation of therapy. No differences in prostate cancer rates were seen during the 5.5 years of treatment (62). In addition, a meta-analysis found an increased risk of death at doses of 400 IU/day (43). Vitamin E can interact with anticoagulants increasing the risk of bleeding. Therefore, men on anticoagulants will be excluded from participation. Adverse effects of Vitamin E include fatigue, weakness, headache, nausea, diarrhea, flatulence and abdominal pain at high doses (over 1000 mg/day). However, at lower doses as prescribed in this trial, Vitamin E is generally well tolerated.

Selenium: The total daily dosage of selenium in the organic form of L-selenomethionine will be 0.20mg. Commercial products include selenium at doses between 0.05 mg and 0.133 mg. Randomized trials included doses ranging from 0.026 to 0.225mg, which the most common dose being 0.20mg (34, 56, 59, 60, 63). These trials have shown that selenium increases sperm motility at 3 and 6 months (34, 63). The tolerable upper limit intake level for selenium (from supplements and food) is 0.4 mg. Levels above this are associated with hair and nail brittleness and loss.

*L-carnitine:* The total daily dosage of L-carnitine in the form of L-carnitine-L-tartrate and L-carnitine fumerate will be 1000 mg. Commercial products include L-carnitine at doses between 50 and 1000 mg. Randomized controlled trials included doses ranging from 2000 to 3000 mg (48, 58, 64, 65). Common L-carnitine adverse effects include diarrhea, nausea, stomach cramps, and vomiting. Uncommon serious adverse effects include seizures. L-carnitine has been shown to increase pregnancy rates following IVF in small, randomized, placebo-controlled trials (36, 48).

Zinc: The total daily dosage of zinc will be 20 mg. Commercial products include zinc in the form of zinc amino acid chelate at doses of 10 to 70 mg. Randomized controlled trials have included dosages ranging from 25 to 500 mg (37, 47, 56). These small trials have shown that zinc increased pregnancy rates following ART and improved sperm motility at 3 months. The tolerable upper intake level for zinc is 40 mg per day.

Folic acid: The total daily dosage of folic acid will be 1000 mcg. Commercial products include folic acid at doses of 60 to 5000 mcg. Randomized controlled trials (including combination formulations and isolated) have included dosages ranging from 500 to 5000 mcg (56, 66, 67). These small trials have suggested that folic acid improves sperm concentration. The tolerable upper intake level for folic acid is 1000 mcg per day.

Lycopene: The total daily dosage of lycopene will be 10 mg. Commercial products include lycopene at doses of 10-100 mg. A randomized controlled trial (of an antioxidant combination) included lycopene at a dosage of 6 mg (56). Dietary lycopene intake is positively correlated with sperm morphology (68). Daily supplements containing 30mg of lycopene have been used safely.

Combination formulations: A number of small studies have examined the effect of a combination of antioxidants on pregnancy following IVF and/or semen parameters (34, 37, 38, 56-60, 63, 65, 69-73). The antioxidant formulations vary from study to study. Menevit (Lycopene, Vitamin E, Vitamin C, Zinc, Selenium, folic acid, and garlic) treatment of the male partner for 3 months prior to IVF was shown to increase subsequent pregnancy rates following IVF with ICSI compared to placebo (38.5% versus 16%) in a randomized controlled trial including 60 couples (56). This formulation is similar to ConceptionXR except that Menevit does not include Vitamin D or L-Carnitine and ConceptionXR does not include garlic. Menevit is not available in the US. Side effects in the combination anti-oxidant group occurred in 8% of males and were mild (gastroesophageal reflux and constipation).

Vitamin D: Vitamin D is included in ConceptionXR in the form of cholecalciferol at a dose of 2000IU. Cross-sectional studies suggest a positive association between serum 25-hydroxyvitamin D level and sperm motility in both fertile and infertile men (74, 75). Vitamin D supplementation has not been assessed in a clinical trial on male fertility. The tolerable upper limit of Vitamin D is 4000IU per day.

#### 5.6.2 Placebo

The placebo will weigh, smell, and look the same as the antioxidant supplement, ConceptionXR, using an inert substance. The placebo will be compounded by Theralogix.

## 5.6.3 Manufacturing of ConceptionXR and Quality Control

ConceptionXR Motility Support Formula is manufactured by Theralogix. All active components and doses along with inert components are publically available (<a href="www.theralogix.com">www.theralogix.com</a>). All Theralogix supplements are manufactured in an NSF GMP-registered facility. ConceptionXR is independently tested and certified by NSF International for content accuracy, purity, and freedom from contaminants. The average expiration date for most dry powder dietary supplements is 2 years.

## 5.6.4 Distribution

The ConceptionXR and placebo bottle will be shipped to an investigative drug service (IDS, Almac or comparable) in 3 batches. The IDS will label kits with unique blinded identifiers (randomly allocated to supplement and placebo) and distribute in a blinded fashion to the study sites.

## 5.7 Study Flow:

# 5.7.1 Screening:

## Female Screening Visit:

- 1. Obtain informed, signed consent
- 2. Complete medical history and physical exam of female study participant
  - a. Complete RMN Medical History case reporting form
  - b. Obtain Vital signs, height, weight, neck circumference
  - c. Pap smear, if necessary, per current ACOG time-frame guidelines
  - d. Standard physical exam conducted by clinician (if not done within past 12 months)
  - e. Pelvic ultrasound (or sonohysterogram) with documentation of uterine size, presence of fibroids, and ovarian dimensions within past 12 months.
- 3. Pre-conception counseling
- 4. Sonohysterogram or hysterosalpingogram to verify patency in at least one tube, and normal uterine cavity (or documentation within past 3 years). An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or tubal disease or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
- 5. Collect blood for tests to determine eligibility (if not already obtained).
- 6. Offer optional blood test for Rubella, Varicella, HIV, and genetic tests for cystic fibrosis, SMA, sickle cell, and thalassemia (based on ethnicity). The costs for these blood tests are not included in determining the patient care budget for this protocol. Patients need to be made aware that they will be responsible for paying for these tests if their insurance company does not cover the costs.

## Determine eligibility. If eligible:

- 1. Have the participant complete the following RMN questionnaires:
  - Genetic Risk Factors questionnaire
  - Female Sexual Function Index (FSFI)
  - o SF-12
  - o PHQ-9
  - o FertiQoL
  - Epworth Sleepiness
  - Stop-Bang (Sleep apnea)

- Female Sexual Distress Scale (FSDS)
- Diet History Questionnaire II (DHQ-II)
- 2. Obtain height and weight
- 3. Obtain blood and urine sample for RMN Biorepository, if consent obtained
- 4. Provide salivary collection kit and instructions, if consent obtained
- 5. Explain how to use ovulation predictor test and pregnancy tests
- 6. Advise the participant to contact us with a positive pregnancy test to schedule pregnancy ultrasound

# Male Screening Visit:

- 1. Obtain informed, signed consent
- 2. Obtain a semen sample if semen analysis has not been performed within the past 6 months.

# Determine eligibility. If eligible:

- 3. Complete the following RMN questionnaires:
  - a. Partner Genetic Risk Factors Questionnaire
  - b. SF-12
  - c. PHQ-9
  - d. FertiQoL
  - e. Epworth Sleepiness
  - f. Stop-Bang (Sleep apnea)
  - g. International Index of Erectile Function (IIEF)
  - h. Psychosexual daily questionnaire (PDQ)
  - i. Androgen Decline in the Aging Male quantitative questionnaire (qADAM)
  - j. Diet History Questionnaire II
  - k. Sun Exposure and Behaviour Inventory (SEBI)
- 4. Provide instructions for future semen collections.
- 5. Provide salivary collection kit and instructions, if consent obtained
- 6. Obtain semen sample for RMN Biorepository, if consent obtained

## 5.7.2 Study treatment visit 1 (males only):

- 1. Participant completes the ASA24.
- 2. Obtain height and weight and neck, waist and hip circumferences.
- 3. Obtain a semen sample following appropriate abstinence and evaluate by semen analysis as suggested by WHO 5 standards.
  - a. Samples will be evaluated for volume, sperm concentration, percent sperm motility, forward progressive motility, at the local site laboratory.

- b. Prepare semen slides. Incidence of normal sperm morphology will be determined using WHO 5 morphological assessment by a single technician at a central laboratory.
- c. Three aliquots of raw semen will be frozen and stored at -20° C, then shipped in batches to a central site for TUNEL analysis, SCSA, and COMET assay.
- d. If consent obtained, a fourth aliquot of raw semen will be obtained for the RMN Biorepository.

## 4. Collect blood sample

- a. Collect serum for UVA central laboratory for measurement of total testosterone, FSH, LH, vitamin D 25-OH.
- b. Collect and store serum. Randomly selected samples will be shipped to a central laboratory for analysis of antioxidant levels.
- c. If consent obtained, collect blood sample for RMN Biorepository.
- 5. Collect urine sample to be sent to a central laboratory for testing for environmental contaminants.
- 6. Randomization and assignment of study drug kit
- 7. Dispense assigned study pill kit. Instruct participant to take one capsule and one tablet twice a day. Provide 1-month supply (Package 1). Instruct participant to bring pill bottles with any remaining pills with him on day of next visit.
- 8. Dispense patient journal.
- 9. Schedule study visit 2 for ≤30 days.
- 10. Provide male with 7 ovulation strips with instructions and 2 pregnancy tests with instructions.

## 5.7.3 Study treatment visit 2 (males only):

- 1. Count remaining pills.
- 2. Assess for side effects from treatment.
- 3. Collect blood sample
  - a. Collect and store serum. Randomly selected samples will be shipped to a central laboratory for analysis of antioxidant levels.
- 4. Dispense assigned study pill kits. Instruct participant to take one capsule and one tablet twice a day. Provide 2-month supply (Package 2). Instruct participant to bring pill bottles with any remaining pills with him on day of next visit.
- 5. Dispense patient journal.
- 6. Schedule study visit 3 for ≤60 days. Provide semen collection instructions for next visit.
- 7. Provide male with 14 ovulation strips and 4 pregnancy tests.

## 5.7.4 Study treatment visit 3 (males only):

1. Participant completes the ASA24 online.

- 2. Count remaining pills.
- 3. Assess for side effects from treatment.
- 4. Collect blood sample
  - a. Collect serum for UVA central laboratory for measurement of vitamin D 25-OH.
  - b. Collect and store serum. Randomly selected samples will be shipped to a central laboratory for analysis of antioxidant levels.
- 5. Obtain a semen sample following appropriate abstinence and evaluate by semen analysis as suggested by WHO 5 standards.
  - a. Samples will be evaluated for volume, sperm concentration, percent sperm motility, forward progressive motility at the local site laboratory.
  - b. Prepare semen slides. Incidence of normal sperm morphology will be determined using Kruger Strict morphological assessment by a single technician at a central laboratory.
  - c. Three aliquots of raw semen will be frozen, stored at -20° C, and then shipped in batches to a central site for TUNEL, SCSA, and COMET assay.
- 6. Dispense assigned study pill kit. Instruct participant to take one capsule and one tablet twice a day. Provide 3-month supply (Package 3). Instruct male to have female partner call with menses to schedule baseline ultrasound for clomiphene citrate/IUI cycle.
- 7. Dispense patient journal.
- 8. Schedule study visit 4 for ≤120 days. Instruct participant to bring pill bottles with any remaining pills with him on day of next visit.

# 5.7.5 Clomid and IUI cycles (couple):

## **Baseline Ultrasound Visit**

- 1. Females will call with menses and come in Day 1-5 (Preferably day 3 for baseline monitoring) for first cycle only.
- 2. Perform comprehensive baseline ultrasound.
- 3. Dispense Infertility Treatment Medications: 10 tablets of clomiphene citrate and 10,000 IU hCG. Patient is to take clomiphene citrate 100 mg for 5 days starting on cycle days 1,2,3,4 or 5.
- 4. Dispense patient journal

# Monitoring Visit number 1: Within 3 days after completing 5-day drug cycle (Cycle Day 8-12)

- 1. Transvaginal ultrasound for endometrial and follicular monitoring
- 2. Adverse effects and concomitant medications query

## Monitoring Visit number 2 and beyond:

Visits for subjects will be conducted on an individualized basis until hCG administration. When a decision has been made to give hCG on the next day, a follow up monitoring visit on that day is unnecessary.

- Transvaginal ultrasound examination for endometrial and follicular monitoring
- Adverse effects and concomitant medications query

# hCG administration day:

- 1. 10,000 IU in 1 cc diluent delivered IM
- 2. Transvaginal ultrasound examination for endometrial and follicular monitoring is not necessary if one has been performed within 2 days.

#### Criteria for hCG administration:

- First occurrence of lead follicle reaching 20 mm (in average diameter in two dimensions), or
- First occurrence of two lead follicles greater than 18 mm diameter (in average diameter in two dimensions), or
  - The day after the lead follicle reaching 18 mm (in average diameter in two dimensions), or the day of detection of presumptive ovulation by ultrasound

## Criteria for withholding hCG:

- If a leading follicle does not reach a mean diameter of 18 mm after 18 days of treatment, or
- Endogenous LH surge happens [which can lead to premature luteinization], or
- Increased risk for OHSS and/or high-order multiple gestational pregnancy exists when more than 4 growing follicles develop (mean diameter >18 mm), or
  - \*Protocol medication adjustment:
- 1. If no ovulation or development of at least one follicle ≥ 18 mm in average diameter, then increase dosage in the subsequent cycle.
- 2. If only one follicle ≥ 18 mm in average diameter, the dosage increase for subsequent cycles will be left to physician's discretion.
- 3. If more than four follicles are ≥ 18 mm in average diameter, dosage will be reduced in the subsequent cycle.
  - \*Cancellation criteria: Cycles will be cancelled if significant adverse reactions develop in response to administered medications, if criteria for withholding hCG administration are encountered, or per patient's request.

## <u>Insemination day visit:</u>

- 1. Each site will perform its standard sperm processing and intrauterine insemination procedure.
- 2. Record parameters of semen analysis before and after sperm preparation.
- 3. Record time of insemination.
- 4. Instruct patient to check urine pregnancy test 2 weeks after insemination and call with results.
- 5. Provide clomiphene citrate for next cycle. Counsel not to take it until instructed to do so.

<u>Pregnancy test:</u> Patient is to do a home pregnancy test 2 weeks after insemination using the urine home pregnancy tests provided.

## Four possible outcomes:

- A. No pregnancy on urine pregnancy test
- B. Positive urine pregnancy test- serum βhcg level returns <5 mIU/ml- no pregnancy
- C. Positive urine pregnancy test- serum βhcg level returns >5 mIU/ml, retest for rising level in 2 days- no pregnancy
- D. Positive urine pregnancy test- serum βhcg level returns >5 mIU/ml, retest for rising level in 2 days- pregnancy

**A. Negative Urine Pregnancy Test/No pregnancy**: Repeat cycles until pregnancy occurs or male completes a total of 6 months of treatment.

Criteria to initiate Cycles 2 or 3 (Day 3 +/- 2 days):

- 1. Negative urine pregnancy test,
- 2. Male still on treatment.

Cycle 2 and 3 will be identical to Cycle 1, except that there will be no Baseline Ultrasound visit. When the subject contacts the site with the results of her urine pregnancy test or start of menses, she will be instructed by the site to start her clomiphene citrate. She will then return to the site for Monitoring Visit 1 (see above).

In women who report a positive urine pregnancy test, obtain serum βhcg level.

# B &C. Positive Urine Pregnancy Test (no pregnancy)

Patient will have a serum  $\beta$ hcg level checked. If >5 mIU/mI, return in 2 days to check for a rising level in serum  $\beta$ hCG; if the first level is <5 mIU/mI or if there is not a rising level, patient will initiate Cycles 2 or 3.

**D. Positive Urine Pregnancy Test (pregnancy)**: Biochemical pregnancy will be defined as  $\theta hCG > 5$  units/ml 2 weeks after insemination followed by a rising level two days later

- Patient will have a serum βhcg level checked. If >5 mIU/ml, patient will return in 2 days to check a rising level in serum βhcG.
- If rising βhcg level, schedule Pregnancy Ultrasound Visit. Instruct male to come to pregnancy ultrasound visit to complete study visit 4. Remind him to bring his pill bottle.

# 5.7.6 Study visit 4 (males only):

- 1. Count remaining pills.
- 2. Confirm pregnancy status (pregnant or not pregnant) of female partner.
- 3. Assess for side effects from treatment.
- 4. Obtain blood sample from those males whose female partner did not conceive.
  - a. Collect and store serum. Randomly selected samples will be shipped to a central laboratory for analysis of antioxidant levels.

# **5.7.7** *Pregnancy ultrasound(s):*

To be done between 6 and 9 weeks gestation. Clinical pregnancy rate will be defined as the identification of intrauterine sac(s) with positive fetal cardiac activity in at least one sac.

- 1. A transvaginal ultrasound will be performed between 6 and 9 weeks gestation to assess advancement of the pregnancy by locating the gestational sac(s) and to determine fetal viability by detection of fetal heart motion.
- 2. Remind participant to contact the study coordinator within 2 weeks of the end of pregnancy.
- Determine where she will be obtaining prenatal care and delivering. Obtain permission to access maternal and neonatal medical records to abstract data related to the birth of the infant.
- 4. Participation in the intervention phase of the study will end for couples that experience a pregnancy loss.
- 5. Obtain a separate consent form to enter the patient into the Pregnancy Registry.

#### 5.7.8 20-week contact:

Women who do not report an end of pregnancy prior to 20-weeks gestation, will be contacted to confirm pregnancy status and update information on site of prenatal care and planned delivery.

#### 5.7.9 Pregnancy outcome:

Subjects will be contacted to obtain pregnancy outcome information including outcome (miscarriage, ectopic, abortion, live birth) and answer follow-up questions specific to that outcome (for miscarriage: date miscarriage identified, for live birth: date of delivery, gestational number, birth weight, gender, and obstetrical complications). Medical records will also be obtained from the prenatal site, pediatrician, and hospital as needed to confirm obstetrical and neonatal outcomes.

# 6 Data Collection

**Table 1: Overview of Timing and Content of Data Collection for Primary Cohort** 

| Data Collection (multiple checks within column indicates that data acquisition is distributed over contacts and/or updates) | Semen Analysis | DNA Fragmentation<br>(TUNEL and/or SCSA) | Dietary Assessment | Compliance | Fetal development,<br>estimated date of delivery,<br>Clinical pregnancy | Pregnancy Outcomes |
|---|---|---|---|---|---|---|
| Female screening visit | | | ✓ | | | |
| Male screening visit | <b>√</b> | | ✓ | | | |
| Study visit 1 | <b>√</b> | ✓ | ✓ | ✓ | | |
| Study visit 2 | | | | ✓ | | |
| Study visit 3 | ✓ | ✓ | ✓ | ✓ | | |
| Study visit 4 | | | | ✓ | | |
| Pregnancy Ultrasound (6 wks gestation) | | | | | ✓ | |
| Pregnancy Status Update (20 to 24 wks) | | | | | | <b>✓</b> |
| Pregnancy Outcome<br>Reporting and Medical<br>Record Review | | | | | | <b>✓</b> |

# 6.1 Specimen collection, processing, and shipment

# 6.1.1 Semen Collection

Semen samples will be obtained at the screening visit (as needed), visit 1, and visit 3. Semen assessment at the screening visit and visit 1 will occur prior to treatment. Samples will be assessed using a standard semen analysis, including assessment of morphology using strict criteria, the SCSA, COMET, and TUNEL. These analyses will allow us to assess sperm motility and

DNA structure, two components frequently affected by ROS. Couples will not be informed of results until the end of the study, as this information could lead to behavior changes. Men will be asked to abstain from ejaculation 2-5 days prior to collection. Samples will be collected by masturbation at the clinical site. Samples will be allowed to liquefy for 30 minutes at 37° C prior to analyses.

# 6.1.2 Semen analysis

Subsequently the initial physical characteristics (e.g. volume, pH) will be recorded. Count and motility will be measured using 5µl of semen loaded on a sperm counting chamber (Microcell, Conception Technologies, San Diego, CA) (76). Semen smears will be made for each sample, stained by the Papanicolaou method, and shipped to a central laboratory for assessment of sperm morphology by a single technician, using strict criteria defined by WHO 5 (77). Semen analyses will be conducted at the screening visit, study visit 1 (prior to treatment), and study visit 3 (at 3 months of treatment).

## 6.1.3 DNA integrity testing

DNA integrity needs to be assessed in addition to traditional semen parameters as a significant number of men will have high levels of DNA fragmentation despite a normal semen analysis (39-41). There are three common assays of sperm DNA integrity: two of which measure actual DNA strand breaks (neutral COMET and TUNEL) and one of which measures the potential for strand breaks (SCSA) (78, 79). The SCSA assay is proposed as it is the only DNA integrity testing method that is standardized in a commercial laboratory. It is the only test in wide clinical use.

#### 6.1.4 SCSA

An aliquot of raw semen will be sent to a central laboratory. SCSA will be performed as previously described (80), generating a DNA fragmentation index (DFI) on 5000 sperm per sample. The assay is based on the color of fluorescence of acridine orange stained sperm, where red fluorescence reflects damaged DNA (single-stranded) and green fluorescence reflects native (single-stranded) DNA. The DFI is calculated as the ratio of damaged DNA (red)/total DNA (red + green). Previous studies have shown that males with sperm with a DFI greater than 25% have a longer time to natural pregnancy (9). SCSA has been shown to be highly precise and reproducible (CV 1-3%) (80). Results will be faxed to the RMN data coordinating center. SCSA will be conducted on the study visit 1 sample (prior to treatment) and study visit 3 sample.

#### 6.1.5 TUNEL

One aliquot of raw semen will be sent to a central laboratory. The TUNEL assay will be performed on fixed, permeabilized sperm as described (81, 82). End labeling of breaks will be performed using fluorescent dUTP and terminal transferase and will employ a commercial, widely used kit (TUNEL in situ cell death detection kit, Roche). All TUNEL assays will be performed at a single site will be analyzed in batches of 10–20 samples, and a minimum of 10,000 sperm will be assessed per assay. Previous ROC analysis suggests that a 20% fragmentation cutoff would yield a 96.5% sensitivity and 89.4% specificity to detect infertile males (82). TUNEL assay will be conducted on samples from study visit 1 (prior to treatment) and study visit 3 (after 3 months of treatment).

#### 6.1.6 *COMET*

One aliquot of raw semen will be sent to a central laboratory for the COMET assay. The comet assay is one of the simplest methods to measure sperm DNA damage by quantifying the single and double strand breaks. The principle of the assay is that the sperm nuclear DNA is separated in an electric field based on charge and size, which is viewed with a fluorescent DNA-specific dye. The resulting images, which resemble comets with an intact head and tail, determine the extent of DNA damage based on the intensity of staining and morphology of the comet. The COMET assay will be conducted on the study visit 1 sample (prior to treatment) and study visit 3 sample.

## 6.2 Compliance

Compliance and cross-over will be assessed via two mechanisms: 1) pill counts and 2) measurement of Vitamin E (alpha-tocopherol), L-carnitine, and zinc (and, if possible, Vitamin C and selenium) in blood. Compliance and cross-over will be assessed by these 2 mechanisms at study visits 2, 3, and 4 (corresponding to months 1, 3, and 6 of treatment). At study visit 1 (month 0 of treatment), a baseline measurement will be established.

## 6.2.1 Measurement of vitamin levels

A random sample of 10% of blood samples (as done in the SU.VI.MAX study (83)) obtained at study visits 2, 3, and 4 will be shipped to a laboratory such as the Clinical Pharmacology Analytical Services Laboratory (CPAS) in the Department of Experimental and Clinical Pharmacology in the College of Pharmacy at the University of Minnesota (<a href="http://www.pharmacy.umn.edu/cpas/services/index.htm">http://www.pharmacy.umn.edu/cpas/services/index.htm</a>). All three vitamins will be measured using a LC-MS/MS method. Internal standards are commercially available. These samples will allow us to assess for compliance. As placebos will also be samples, we will also be able to assess for cross-over.

#### 6.3 Dietary assessment

A previous observational study showed that a health-conscious diet is associated with a decrease in sperm DNA fragmentation, suggesting that natural antioxidants are beneficial to sperm (31). However, another observational study using food frequency questionnaires failed to find an association between any antioxidant measure and DNA fragmentation, perhaps because the cohort was comprised of healthy volunteers (32). Therefore, to assess for possible effect modification by baseline dietary composition and vitamin intake, we will assess these through a 24-hour recall during the 1<sup>st</sup> study visit and a food frequency questionnaire at baseline. Secondary analysis could be conducted to examine the relationship between baseline dietary composition and vitamin intake and semen parameters and couple fecundability and fertility over the study period. A second 24-hour recall will be obtained at the 3-month study visit to determine if there were differential changes in dietary composition among treatment groups.

To measure food intake, we will use the validated, self-administered, web-based, 24-hour recall questionnaire, ASA24 and Diet History Questionnaire II. The method allows for collection of detailed intake and portion sizes. It does not affect what an individual chooses to eat on a given day, due to its retrospective data collection. It is administered in close proximity to the intake

#### 6.1.6 *COMET*

One aliquot of raw semen will be sent to a central laboratory for the COMET assay. The comet assay is one of the simplest methods to measure sperm DNA damage by quantifying the single and double strand breaks. The principle of the assay is that the sperm nuclear DNA is separated in an electric field based on charge and size, which is viewed with a fluorescent DNA-specific dye. The resulting images, which resemble comets with an intact head and tail, determine the extent of DNA damage based on the intensity of staining and morphology of the comet. The COMET assay will be conducted on the study visit 1 sample (prior to treatment) and study visit 3 sample.

# 6.2 Compliance

Compliance and cross-over will be assessed via two mechanisms: 1) pill counts and 2) measurement of Vitamin E (alpha-tocopherol), L-carnitine, and zinc (and, if possible, Vitamin C and selenium) in blood. Compliance and cross-over will be assessed by these 2 mechanisms at study visits 2, 3, and 4 (corresponding to months 1, 3, and 6 of treatment). At study visit 1 (month 0 of treatment), a baseline measurement will be established.

## 6.2.1 Measurement of vitamin levels

A random sample of 10% of blood samples (as done in the SU.VI.MAX study (83)) obtained at study visits 2, 3, and 4 will be shipped to a laboratory such as the Clinical Pharmacology Analytical Services Laboratory (CPAS) in the Department of Experimental and Clinical Pharmacology in the College of Pharmacy at the University of Minnesota (<a href="http://www.pharmacy.umn.edu/cpas/services/index.htm">http://www.pharmacy.umn.edu/cpas/services/index.htm</a>). All three vitamins will be measured using a LC-MS/MS method. Internal standards are commercially available. These samples will allow us to assess for compliance. As placebos will also be samples, we will also be able to assess for cross-over.

#### 6.3 Dietary assessment

A previous observational study showed that a health-conscious diet is associated with a decrease in sperm DNA fragmentation, suggesting that natural antioxidants are beneficial to sperm (31). However, another observational study using food frequency questionnaires failed to find an association between any antioxidant measure and DNA fragmentation, perhaps because the cohort was comprised of healthy volunteers (32). Therefore, to assess for possible effect modification by baseline dietary composition and vitamin intake, we will assess these through a 24-hour recall during the 1<sup>st</sup> study visit and a food frequency questionnaire at baseline. Secondary analysis could be conducted to examine the relationship between baseline dietary composition and vitamin intake and semen parameters and couple fecundability and fertility over the study period. A second 24-hour recall will be obtained at the 3-month study visit to determine if there were differential changes in dietary composition among treatment groups.

To measure food intake, we will use the validated, self-administered, web-based, 24-hour recall questionnaire, ASA24 and Diet History Questionnaire II. The method allows for collection of detailed intake and portion sizes. It does not affect what an individual chooses to eat on a given day, due to its retrospective data collection. It is administered in close proximity to the intake

day minimizing recall issues. The ASA24 format and design is based on a modified version of the interviewer-administered Automated Multiple Pass Method (AMPM) developed by the US Department of Agriculture. The ASA24 consists of a respondent web site (<a href="https://asa24.westat.com/">https://asa24.westat.com/</a>) and a researcher website (https://asa24.westat.com/researchersite.html). The respondent website guides the participant through the completion of a 24-hour recall for the previous day from midnight to midnight using a dynamic user interface. Information and instructions on the ASA24 can be found at <a href="https://asa24.westat.com/assets-r/docs/ResearcherSite Instructions.pdf">https://asa24.westat.com/assets-r/docs/ResearcherSite Instructions.pdf</a> and a demonstration at <a href="http://asa24demo.westat.com/">https://asa24demo.westat.com/</a>. The male participants will complete the ASA24 on the day of study visit 1 and study visit 3.

The Diet History Questionnaire II (DHQ II) is a food frequency questionnaire (FFQ) developed at the Risk Factor Monitoring Branch. The DHQ II consists of a respondent website and a researcher website. The respondent website guides the participant through the completion of a questionnaire regarding portion size, usual intake, and dietary supplements over the past year. Information and instructions on the DHQ Ш can be found at http://appliedresearch.cancer.gov/dhq2/ and а demonstration at https://appliedresearch.cancer.gov/cgi-bin/dhq2.pl?module=2&method=1. In summary, the DHQ has been validated as a measure of frequency and nutrient assessment. The full and extensive list of the 176 nutrients, dietary constituents, and food groups assessed with the DHQ is available on the website. Both male and female participants will complete the DHQ II at screening.

## 6.4 Male urinary testing for environmental contaminants

Urine samples will be obtained from male participants at the visit 1 for future assessment for common environmental contaminants such as Bisphenol-A (BPA). Samples will be collected into BPA-free collection containers at the clinical site and transferred to BPA-free cryovials by study staff. Samples will be stored frozen until shipped in batches to a central laboratory for analysis.

## 6.5 Stress biomarker testing

A first morning (basal) salivary sample will be obtained from male and female participants using a salivary collection device. Participants will be told to collect the sample immediately upon awakening before eating, drinking, smoking or brushing their teeth. Samples from males will be collected around the time of study visit one and returned at the time of study visit one or by prepaid overnight shipping. Females will collect their sample shortly after their screening visit and return the sample via prepaid overnight shipping. Samples will be stored at -20°C until analysis. Samples will be analyzed for stress biomarkers such as amylase and cortisol. Participation in this part of the study will be optional.

## 6.6 Male laboratory testing (central core laboratory)

The core lab will analyze the blood samples from the males at study visit 1 (prior to treatment) for total testosterone, LH, FSH and Vitamin D25-OH. They will also analyze the blood samples from the males at study visit 3 for Vitamin D25-OH.
#### 6.7 Male sunscreen usage

There is increasing concern that benzophenone (BP)-type ultraviolet filters, used in sunscreens, are absorbed by the skin and act as endocrine disruptors (84). Sunscreen ingredients have been demonstrated in vivo2 and in vitro3 to act as endocrine disruptors: either affecting estrogen (those containing PB-2 [tetrahydroxybenzophenone] and BP-8 [hihydroxy-4-methoxybgenzophenonoe]) (85,87) while other UV filters (13 of 29 filters), disrupted progesterone's effect on sperm calcium ion channels (86). While not all UV filters have been associated with a reduction in male fertility, the SEBI (Sun Exposure and Behaviour Inventory) (88) questionnaire will be used to evaluate whether or not men using more sunscreen will experience less fecundity. Future analysis of repository blood or urine samples may be used to more accurately specify which UV filters are responsible for less fecundity.

Sunscreens with PABA block the specific sunlight spectrum responsible for cutaneous synthesis of vitamin D (89). Since the MOXI preparation contains vitamin D, the frequency and amount of both sun exposure and sunscreen usage should be documented.

#### 6.8 Quality of Life (QOL) Measures

Mood, quality of life, and sexual function will be assessed at baseline in both males and females. Quality of life will be assessed by the Medical Outcomes Survey (PHQ-9) and Short Form 12 (SF-12). Female sexual function will be assessed by the Female Sexual Function Inventory (FSFI) along with the Female Sexual Distress Scale (FSDS). This measure is considered the "gold standard" paper and pencil assessment of sexual function and has excellent psychometric properties. Male sexual response will be assessed by the International Index of Erectile Function (IIEF), a multidimensional scale for assessment of erectile dysfunction. The measure addresses the relevant domains of male sexual function (erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction). We will assess hypogonadal symptoms with the Androgen Deficiency and the Aging Male quantitative (qADAM) questionnaire and psychosexual function with the Psychosexual Daily Questionnaire (PDQ). We will assess quality of life relating to infertility and treatment with the FertiQoL survey. There may also be some impact on fertility and we will investigate this in our study. We will use two simple scales to evaluate sleep, the STOP BANG questionnaire for sleep apnea, and the Epworth Sleepiness Scale. (See Appendices)

#### 6.9 Early Pregnancy Ultrasound

A transvaginal ultrasound (standard for first trimester imaging), will be scheduled, ideally between 6 2/7 and 7 2/7 weeks of gestation; no later than 9 6/7 weeks. This ultrasound confirms estimated date of delivery, and in the case of loss, documents likely developmental stage at the time of the loss (e.g. empty gestational sac, fetal pole not heart rate, normal fetal pole). Presence and size of gestational sac, presence and size of yolk sac, presence of fetal pole and crown-rump length, and presence of cardiac motion and heart rate will be recorded. With minimal costs, ultrasounds achieve 2 study goals. They serve as an incentive to subjects for participation and compliance with study protocols and they provide estimates of miscarriage and clinical pregnancy rates.

#### 6.10 Ascertainment of Pregnancy Outcomes

Participants will be encouraged to report outcome (miscarriage, ectopic, abortion, live birth) and answer follow-up questions specific to that outcome (for miscarriage: date miscarriage identified and for live birth: date of delivery, gestational number, birth weight, gender, and obstetrical complications).

#### 6.11 Pregnancy Registry

All subjects who deliver will be encouraged to participate in our Pregnancy Registry which currently provides infant follow up till age 3. This is currently a separate protocol and we will also obtain separate informed consent for participation in this protocol.

#### 6.12 Biologic Repository

We will use the RMN biorepository as a biological specimen's bank at baseline prior to randomization in both females and males. This Biorepository will serve a two-fold purpose. First, it can serve as a repository to run additional serum assays for novel markers of infertility or treatment success that are discovered while the study is ongoing. Second, it will serve as a source of samples for further studies including proteomics, metabolomics, etc. We will collect whole blood, serum, and urine from female and male participants, if consented. We will also collect semen from male partners, if consented. Subjects will be able to opt in or opt out of these studies via separate signature on the consent form. We will also store leftover serum samples for additional post hoc studies. Study subjects will be separately consented to store and use their leftover serum samples from the study and will similarly be able to opt out. Further details of specimen processing can be found in the Manual of Operations and Procedures.

#### 6.13 Central Core Laboratory

Screening labs to determine eligibility will be run in the local RMN site labs. Given the variability of assays between labs, assays will be performed in a central lab at the Ligand Assay Core lab at the University of Virginia.

#### 7 Data Analysis

#### 7.1 Internal Pilot

We will be conducting an internal pilot study with a three-fold objective. The objective of the internal pilot is 1) to determine the distribution of various types of semen abnormalities in the study population, 2) to examine the effect of our antioxidant formulation on male semen parameters and DNA integrity at 3 months of treatment compared to controls, and 3) to determine the feasibility of the proposed recruitment paradigm.

The first 120 men enrolled in the MOXI trial will be included in the internal pilot. The 120 men will complete the entire MOXI protocol. Once the first 120 men enrolled in MOXI have completed study visit 3, the DCC will complete the data analysis for the internal pilot. After data cleaning and transformations, if needed, semen parameter measures will be analyzed using a generalized linear mixed model (including random effects for site if necessary) or generalized linear model (if fixed effects for site are used). Interaction terms will be used to determine the extent to which the change in semen parameter measures differs by type of baseline semen abnormality (oligospermia, asthenospermia, high DNA fragmentation), if there is evidence of effect modification, change estimates will be determined for type.

If we assume that 50% of the males will have low motility (<40%) after taking into account potential dropouts and that the drop-outs will be randomly distributed, we should have 30 men in each group. Based on Fedder et al. we can assume that the percentage of sperm motility at the end of treatment in antioxidant group can be increased by 32% (SD20%) from basement and that in the placebo group it will be increased by 20 % (SD12%)(83). Furthermore, Khadem et al. (38) reported that DNA fragmentation decreased from 22.1 $\pm$ 7.7% to 9.1 $\pm$ 7.2% in antioxidant group (38). Under these assumptions, or pilot phase will have 80% power to detect the differences suggested in the literature with  $\alpha$ =0.05.

Feasibility will be assessed by recruitment pace. We anticipate that the pilot enrollment will be completed by 6 months starting from when all the sites have been initiated to start the trial. Thus 120 couples will be recruited over the 6 months. The pilot goal assumes that recruitment pace will increase over the course of the entire study period.

Assuming we fail to reject the null hypothesis that motility and DNA fragmentation percentage do not differ between the two treatment groups (antioxidant and placebo), the MOXI trial will stop enrolling subjects. Enrolled couples will complete the study protocol. Data analyses will be conducted for the primary and secondary outcomes for the primary study. These results could be used to power a future study should point estimates suggest that male partner treatment with antioxidants increases live birth or pregnancy rates.

Assuming 1) we reject the null hypothesis that motility and DNA fragmentation percentage do not differ between the two treatment groups (antioxidant and placebo) and 2) we determine that the study is feasible, the MOXI trial will continue until a total of 790 couples have been enrolled. Since the primary outcome will not be analyzed for the pilot, it is not thought that adjustments in significance levels will be required for these analyses.

#### 7.2 Primary and Secondary Outcomes

The primary outcome is a live birth resulting from a pregnancy occurring within the 6 months of treatment. Live birth is defined as a delivery of a live infant after 20-weeks gestation. Secondary outcomes include pregnancy, defined by a positive home pregnancy test within the 6 months of treatment. We will conduct an intent-to-treat analysis. Cumulative incidence of live birth and pregnancy will be compared between those couples randomized to antioxidants and those couples randomized to placebo. In addition, discrete-time hazard models will be used to compare time-to-pregnancy between groups. Subsequent subgroup analyses will be conducted to assess for effect modification by type of baseline sperm abnormality. All analyses will include fixed or random effect terms as needed to account for potential site effects.

#### 7.3 Sample Size and Statistical Power

For the power analysis, we assume live birth rates of 35% in the antioxidant group and 25% in the control group, and 17% drop-out (based on drop-out rate in prior RMN trials). A 25% live birth rate was estimated, assuming 5% live birth rate in the first 3 months of timed intercourse and a 20% live birth rate in the 3 clomid/IUI cycles. The 20% live birth rate is the live birth rate in AMIGOS participants receiving up to 3 cycles of clomid/IUI and female partner under the age of 35. Under these assumptions, a sample size of 395 per group will yield 80% power using a two-sided chi square test at  $\alpha$ =0.05 (Table 2).

Table 2: Sample size estimates under a variety of assumptions

| Proportion (%)<br>of live birth in<br>placebo group | Proportion (%) of live birth in antioxidant group | Power<br>(%) | Number of patients per arm with 0% dropout | Total number of patients with 0% dropout | Total number of patients with 17% dropout |
|---|---|---|---|---|---|
| 20 | 30 | 80 | 294 | 588 | 708 |
| 20 | 30 | 90 | 392 | 784 | 944 |
| 25 | 35 | 80 | 328 | 656 | 790 |
| 25 | 35 | 90 | 440 | 880 | 1060 |
| 30 | 40 | 80 | 356 | 712 | 858 |
| 30 | 40 | 90 | 477 | 954 | 1150 |
| 20 | 35 | 80 | 138 | 276 | 332 |
| 20 | 35 | 90 | 185 | 370 | 446 |
| 25 | 40 | 80 | 152 | 304 | 366 |
| 25 | 40 | 90 | 203 | 406 | 490 |

For subgroup analyses, power is dependent on the distribution of the sperm abnormalities, the control live birth rate and the treatment effect difference (see Table 3).

**Table 3: Power for subgroup analyses** 

| Proportion affected (%) | Total N for subgroup | Control Group<br>Pregnancy<br>Proportion (%) | Treatment Effect Difference (%) | Alpha | Power (%) |
|---|---|---|---|---|---|
| 70 | 552 | 20 | 10 | 0.05 | 78 |
| 60 | 474 | 20 | 10 | 0.05 | 71 |
| 50 | 394 | 20 | 10 | 0.05 | 63 |
| 40 | 316 | 20 | 10 | 0.05 | 54 |
| 30 | 236 | 20 | 10 | 0.05 | 43 |
| 70 | 553 | 20 | 15 | 0.05 | 98 |
| 60 | 474 | 20 | 15 | 0.05 | 96 |
| 50 | 395 | 20 | 15 | 0.05 | 92 |
| 40 | 316 | 20 | 15 | 0.05 | 85 |
| 30 | 237 | 20 | 15 | 0.05 | 74 |
| 70 | 553 | 25 | 15 | 0.05 | 97 |

#### 2016.10.12

| 60 | 474 | 25 | 15 | 0.05 | 94 |
|----|-----|----|----|------|----|
| 50 | 395 | 25 | 15 | 0.05 | 89 |
| 40 | 316 | 25 | 15 | 0.05 | 82 |
| 30 | 237 | 25 | 15 | 0.05 | 69 |

#### 8 Technical Aspects

#### 8.1 Reporting Adverse Events

All serious adverse events (SAEs) that occur from the start of study drug through thirty days after the last dose of study medication must be reported or if the patient is pregnant, 6 weeks following delivery. A serious adverse event is defined as: fatal or immediately life-threatening; severely or permanently disabling; requiring or prolonging inpatient hospitalization; overdose (intentional or accidental); congenital anomaly; pregnancy loss after 20-weeks gestation; neonatal death up to 6 weeks after delivery; or, any event adversely affecting the study's risk/benefit ratio. Additionally, any event that, based on appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the outcomes listed above is considered an SAE.

If an SAE occurs and is thought to be related to the study medication, the study medication will be discontinued. Twenty-four hour unblinding will be available through the web-based randomization system to break the randomization code for the individual patient if this is required by the PI for proper treatment of the patient.

The site PI will report the SAE by completing and signing the Serious Adverse Event Report Form [available in the "Study Forms" section of the RMN members-only website], and then emailing the document in PDF format to <a href="mailto:rmn.dcc@mailman.yale.edu">rmn.dcc@mailman.yale.edu</a>. Subjects will be identified by study number only. No other identifying information will be included on the form. The site PI must determine and record on the SAE form whether the SAE is unanticipated or anticipated, and if it is related, possibly related, or unrelated to participation in the research.

DCC staff will enter the SAE information in the central database. The Safety Surveillance team, consisting of the DCC, NICHD research scientist and lead PI of the protocol, will analyze the SAE to determine if it meets the criteria listed in the OHRP 45CFR46 and/or FDA 21CFR312.32 & 3.14.80.

These determinations will dictate timeframes for sites' submission to the DCC, and the DCC's submission to the DSMB:

Upon receiving notification of an SAE, the DSMB will review it via a closed-session email or conference-call discussion arranged by the NICHD RMN Committee Coordinator (RMN CC). The DSMB will send a report to the RMN CC within two weeks; reports for life-threatening SAEs will be submitted in one week. The DSMB report will include: statement indicating what related information the DSMB reviewed; the review date; the DSMB's assessment of the information reviewed; and the DSMB's recommendation, if any, for the DCC.

Table 4: Types of Serious Adverse Events and Their Reporting Requirements

| ТҮРЕ | SITE | DCC |
|---|---|---|
| Unanticipated and | Report to DCC within 1 business | Notify DSMB by end of next |
| related/possibly related SAE, | day of discovery | business day of receiving site |
| fatal or life-threatening | | report |
| Other unanticipated and | Report to DCC within 1 business | Notify DSMB 5 business days of |
| related/possibly related SAE | day of discovery | receiving site report |
| Anticipated and related/possibly | Report to DCC within 5 business | Notify DSMB 5 business days of |
| related SAE | days of discovery | receiving site report |
| Unrelated SAE (anticipated or | Report to DCC within 10 | Notify DSMB within 10 business |
| unanticipated | business days (no more than 3 | days (no more than 3 weeks) of |
| | weeks) of discovery | receiving site report |

The RMN CC will then forward the DSMB report to the DCC for the record and appropriate distribution. The DCC will forward reportable events to all RMN investigators, NICHD, and the FDA on behalf of the NICHD if the protocol is under IND. The NICHD Project Scientist will review, sign, and return the IND safety report to the DCC within 2 business days, and will follow up with the site PI and DCC on the SAE until it is resolved. The Protocol PI will evaluate the frequency and severity of the SAEs and determine if modifications to the protocol and consent form are required. Site PIs will report the SAE to their site IRB according to local IRB requirements. For more information, please see the RMN/DSMB Communication Procedure.

Adverse events deemed non-serious will also be recorded throughout study participation from the start of study drug through one week after the last dose of study medication, and reported to the DCC. If an anticipated serious adverse event occurs at a frequency greater than expected, the DCC will notify the DSMB by the end of the next business day of discovery and follow the procedures for reporting serious and unanticipated and related adverse events. The DCC will forward relevant safety information to the DSMB. If an adverse event not initially determined to be reportable to the FDA under 21CFR312.32 is so reportable, the DCC will report the adverse event to the FDA within 15 calendar days after the determination is made. A flow chart for SAEs follows:

Figure 2: SAE flowchart



CFR= Code of Federal Regulations

#### 8.2 Data Collection and Management (including quality assurance/compliance measures)

#### 8.2.1 Data Entry and Forms

Case Report Forms (CRFs) will be developed as the protocol is developed. They will also be implemented in a Web-based Oracle data management system. The Web data entry forms will be similar to the paper forms with the same questions. However, the Web forms usually have more flexibility than the paper forms, such as pull-down menus.

#### 8.2.2 Features of Data Management System

Features of the data management system include study definition; different types of data entry (including double entries and complete audit trail); forms control; query capture, reporting, and resolution; dictionary coding of Adverse Events (AEs) and medical terms; and clinical data review Tools; and prepares data and CRF images to FDA e-Submission Standards. The enduser/reporting/ad hoc query front-end uses a standard Web browser, so that data entry and browsing can be done from any machine with Internet access, without purchase of special software. Login to this system will be through a secured Web server with the security under the protection of Yale Center for Clinical Investigations.

#### 8.2.3 Data Security

A data server and Web server will be used. The data server will be managed by YNHH IT center and the website two servers will be separated and managed by Forte Research Systems. The web server will be accessible through a secured login, but the data server can only be accessed through the web server. For security purposes, no login to the data server will be permitted, and access to the back end is limited to authorized individuals. PHI, including patient names and addresses, will be locked and secured at the participating sites, and data will be linked through a unique identification number, which will be assigned after a patient is screened or enrolled. Access will be limited to authorized individuals (21 CFR 11.10(d)). Each user of the system will have an individual account. The user will log into the account at the beginning of a data entry session, input information (include changes) on the electronic record, and log out at the completion of the data entry session. The system will be designed to limit the number of log-in attempts and record unauthorized access log-in attempts. Individuals will work only under their own access key, and not share these with others. The system will not allow an individual to log onto the system to provide another person access to the system. Access key Users will be asked to change their passwords at established intervals commensurate with a documented risk assessment. This plan has been adapted from the guidelines for computerized systems used in clinical investigations established by the U.S. Department of Health and Human Services Food and Drug Administration.

#### 8.2.4 Data Quality Control

#### Competency to perform procedure/tests in the protocol

The site PI will be responsible for ensuring that study related tests are performed by competent personnel. The criteria for determination of competency may vary between sites in the study.

Attempts will be made to standardize operating procedures whenever possible to minimize intersite variation.

#### **Quality Control Steps**

Quality control of data will be handled on three different levels. The first level is the real-time logical and range checking built into the web-based data entry system. The research coordinators and data entry clerks at the participating sites are required to ensure the data accuracy as the first defense. The second is the remote data monitoring and validation that is the primary responsibility of the data manager and programmer at the DCC. The data manager will conduct monthly comprehensive data checks (SAS programs run on a regular basis as a systematic search for common errors and omissions), as well as regular manual checks (within the database system). Manual checks will identify more complicated and less common errors. The data manager will query sites until each irregularity is resolved. The third level of quality control will be the site visits, where data in our database will be compared against source documents. Identified errors will be resolved between our center and clinical sites. The visits will assure data quality and patient protection.

An audit trail will be added as another security measure. This will ensure that only authorized additions, deletions, or alterations of information in the electronic record have occurred and allows a means to reconstruct significant details about study conduct and source data collection necessary to verify the quality and integrity of data. Computer generated, time-stamped audit trails will be implemented for tracking changes to electronic source documentation.

Controls will be established to ensure that the system's date and time are correct. This is a multicenter clinical trial and will be located in different time zones. System documentation will explain time zone references as well as zone acronyms. Dates and times will include the year, month, day, hour, and minute to the date provided by international standard-setting agencies (e.g. US National Institute of Standards and Technology). The ability to change the date or time will be limited to authorized personnel, and such personnel will be notified if a system date or time discrepancy is detected.

In addition to internal safeguards built into the computerized system, external safeguards will be implemented. Data will be stored at the Data Coordination Center. Records will be regularly backed up, and record logs maintained to prevent a catastrophic loss and ensure the quality and integrity of the data. This plan has been adapted from the guidelines for computerized systems used in clinical investigations established by the U.S Department of Health and Human Services Food and Drug Administration.

#### 8.3 Study Monitoring

A monitoring plan that satisfies ICH/GCP guidelines for monitoring clinical trials will be used. A Project Manager from the DCC will lead this effort, and report findings to the DCC PI. The Project Manager will have full knowledge of the study protocol, Manuals of Procedures, and is familiar with the database system and is trained to review patient charts. The Project Manager will be responsible for training and supervising other personnel.

Once personnel at participating site are trained to recruit patients, the Project Manager will be sent to the site to help initiate the study according to the study protocol, and to ensure that the clinical site meets the scientific, clinical, and regulatory requirements. For example, the Project Manager will review all signed and dated forms required by the FDA (such as financial disclosure forms), the curriculum vitae and certifications of the investigators and personnel, CRF training, and the written IRB approval of the protocol and consent form.

The on-site monitor will return to the clinical site after a defined number of patients are recruited (can be as early as the recruitment of the 2<sup>nd</sup> patient) or a certain time period has passed, depending on the duration of the protocol execution. The schedule of visits will be discussed and agreed in the Steering Committee and we anticipate that the Project Manager will visit each participating site at least once.

During the site visit, the clinical sites should provide to the monitor a space and access to all relevant records including medical records and regulatory binders, and there would be immediate verbal feedback provided to the site after original source documents are compared to entries in the CRF. The clinical sites must agree to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits are resolved. The on-site monitor will conduct an audit of a random sample of entered information against the source documents, a review of all regulatory documents, a review of all informed consents, and a review of all pharmacy logs. The clinical site PI and coordinator should be available to meet the monitor during the visit. The monitor will review electronic data from all sites, providing a method for identifying systematic errors or problems.

To assure Good Clinical/Laboratory Practice, the monitor will control adherence to the protocol at the clinical sites and evaluate the competence of the personnel at the clinical sites including the ability to obtain written informed consents and record data correctly. The monitor will inform the DCC PI, the Steering Committee, and NICHD regarding problems relating to facilities, technical equipment, or medical staff. A thorough written report will follow each site-visit and will include a detailed itemization of discrepancies and items requiring follow-up or reconciliation. This report will also be forwarded to the NICHD Research Scientist for review. The monitor will be responsible for maintaining regular contacts between the investigators in the clinical sites and the RMN. When the study ends, the monitor will also visit the clinical site to provide assistance for close-out.

#### 8.4 Data and Safety Monitoring Board

The NICHD has established an independent DSMB to review and interpret data generated from RMN studies and to review protocols prior to their implementation. Its primary objectives are to ensure the safety of study subjects, the integrity of the research data and to provide NICHD with advice on the ethical and safe progression of studies conducted in the RMN. The DSMB advises on research design issues, data quality and analysis, and research participant protections for each prospective and on-going study. A copy of the DSMB Charter can be found in the appendix.

The DSMB members are appointed by the Director of NICHD in accordance with established NIH and NICHD policies. DSMB members are experts in and represent the following fields:

biostatistics, epidemiology, infertility, gynecology, andrology and ethics. The NICHD Committee Coordinator is responsible for scheduling regular committee meetings, recording all meeting minutes and summarizing the committee recommendations for the Steering Committee and NICHD. Steering Committee members are prohibited from attending closed sessions of the DSMB. Open sessions may be attended by Steering Committee members or Chairperson when requested by NICHD and the DSMB.

The DSMB has quarterly teleconferences to review Network randomized trial protocols with respect to ethical and safety standards, monitors the safety of on-going clinical trials, monitors the integrity of the data with respect to original study design, and provides advice on study conduct. The DSMB periodically monitors data quality, including protocol adherence and adverse events. As outlined in the protocols, the DSMB will conduct interim evaluations of the data. It may recommend protocol modifications based on concern for subject welfare and scientific integrity.

#### 8.5 Reporting

Administrative Reports will be prepared by the DCC - which include monthly and quarterly reports on accrual, data quality and study compliance - and presented to the Steering Committee and DSMB. Statistical reports include reports to the SC, DSMB and AB from the data analysis, and special reports for scientific manuscripts.

Statistical Reports will be generated in SAS. Reports are provided for DSMB reviews, and for final analysis of study results in preparation for scientific publications. The content of the interim reports will be very complete, and will serve as the template for the final report of each study, which in turn will form the basis of the publication of the results. Our proposed reports to the DSMB would include the following: a protocol description and history; accrual rates; site performance in terms of accrual; eligibility; protocol violations; data accuracy and minority representation; patient characteristics by treatment and site; and the rate of adverse experiences.

#### 8.6 Obligation of the Investigator

#### 8.6.1 IRB Review

The site PI is responsible for submitting the approved protocol and consent form to the IRB for review. The IRB must approve all aspects of the study as detailed in the protocol, including the patient informed consent form. It is anticipated that there will be minor site-specific changes in the consent form. The IRB must periodically review the status of the study at appropriate intervals not exceeding one year. The site PI will also be responsible for submitting revisions to the protocol to the IRB, as directed by the DCC, and promptly communicating serious adverse events that result during the study, to both the local IRB and the DCC. After the approval, the informed consent and IRB approval (or amendment) letters must be forwarded to the DCC.

#### 8.6.2 *Maintenance/Retention of site records*

In order to comply with Good Clinical Practice (GCP) requirements, the investigators must maintain the master patient log that identifies all patients entered into the study for a period of two years after the study ends so that the subjects can be identified by audit. The PI must maintain adequate records pertaining to subjects' files and other source data for a minimum of 5 years after completion of the study.

#### 8.7 Regulatory Requirements

The DCC will work with NICHD staff by providing them with clinical study data, reports, and other support as required for AE Reporting and IND submissions. The Project Managers will work with NICHD colleagues in meeting all regulatory requirements including compliance with ICH and HIPAA requirements, FDA code for federal regulations (Title 21), and IND applications. For example, the DCC Project Managers will register this clinical trial in a timely manner with <a href="ClinicalTrials.gov">ClinicalTrials.gov</a> via a web based data entry system called the Protocol Registration System (PRS).

#### 8.8 Protocol Amendments

Once the protocol is approved by the Steering Committee, it is then reviewed by an Advisory Board and a DSMB. After all approvals, the DCC will finalize the protocol document that serves as the agreement among all members of the Network. In the meantime, because the DCC administers all patient care costs for the RMN, the DCC will promptly issue subcontracts to the participating sites based on the cost agreements made by the Steering Committee and NICHD.

After the protocols are approved by the RMN and the Steering Committee decides that changes are necessary for scientific or clinical reasons, the DCC will facilitate the procedure in a timely and diligent fashion. The RMN investigators and key personnel will participate in teleconferences and meetings, discuss, vote, and document circumstance and rationales for the changes as well as the implementation procedure for the changes. These include revising study hypotheses, designs, sample sizes, data entry forms, and appropriate statistical analyses. Once the amendments are finalized and agreed to by the RMN, they will be submitted to the IRB and DSMB for review and approval.

# 8.9 Timeline

#### **Table 5: Timeline for MOXI**

| Study Activities | | Year 1 | | Year 2 | | | Year 3 | | | Year 4 | | | Year 5 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Activities | J-M | A-J | J-S | 0-D | J-M | A-J | J-S | 0-D | J-M | A-J | J-S | 0-D | J-M | A-J | J-S | 0-D | J-M | A-J | J-S 0-D |
| IND exemption | | | | | | | | | | | | | | | | | | | |
| Formulate, test, package antioxidant and placebo | | | | | | | | | | | | | | | | | | | |
| Finalize protocol, IRB revisions, interview modifications | | | | | | | | | | | | | | | | | | | |
| Active enrollment of participants | | | | | | | | | | | | | | | | | | | |
| Treatment of participants | | | | | | | | | | | | | | | | | | | |
| Pregnancy Ultrasound | | | | | | | | | | | | | | | | | | | |
| Determination of Pregnancy Outcome | | | | | | | | | | | | | | | | | | | |
| Medical Record Abstraction | | | | | | | | | | | | | | | | | | | |
| Clean and compile data | | | | | | | | | | | | | | | | | | | |
| Analyze data (begin with clinical fecundability) | | | | | | | | | | | | | | | | | | | |
| Prepare and disseminate results | | • | | | | • | | | | • | • | | | • | • | | | | |

#### 9 RMN Publications Policy

The publications policy proposes guidelines for publications that originate from our collaborative Reproductive Medicine Network. Decisions concerning publications shall be determined by consensus (majority vote) of the collaborating Principal Investigators (or designees) noted below as the "Network." This policy is designed to promote prompt, exact, quality publications and presentations of Network studies with appropriate academic recognition of those with significant contributions. Protocols are classified into three types: 'Main Study' (which may include major and minor publications), "Ancillary Study', and 'Pilot Study'. Additionally, there may be publications from concepts or ideas generated by the RMN ("Related Publications") or from other groups utilizing RMN data and/or specimens, known as "Outside Studies" (those utilizing data and/or specimens from the RMN studies). Abstract submissions to national meetings will also follow the publications policy below. The progress of publications (including presentations) will be a standing agenda note on all teleconferences and meetings. The Steering Committee will make the final decision regarding disputes with respect to analysis request approval, prioritization, presentation, authorship and/or manuscript submission.

#### 9.1 Main Study

A Main Study is a Network study designed prospectively by an investigator independent of other studies. Generally, that investigator becomes Lead Investigator of the protocol and Chair of the Protocol Subcommittee. At the end of each Main Study, a primary analysis resulting in the primary manuscript and a number of secondary analyses is produced based on the research questions stated in the protocol. The Protocol Subcommittee Chair is the primary author of the primary analysis. A Main Study can generate major (related to the major hypotheses) and minor publications (relating to secondary hypotheses).

#### 9.1.1 Major Publications

A major publication is defined as one reporting results of the major hypotheses tested. (For example: Does hMG/IUI increase cyclic fecundity in couples with unexplained or male factor infertility?)

#### a. Authorship

Publications will include the names of investigators from each RMU and the DCC rather than merely identify the "Reproductive Medicine Network". Each RMU and the DCC will have up to two authors per publication, ordinarily the PI and the Co-PI, but this may at times involve another investigator who has contributed to the study at his/her site, in lieu of the PI or Co-PI. The Principal Investigator at each RMU will be responsible for submitting the names of the two authors from that unit and designating them as either the primary and secondary authors of the unit. No more than 2 authors may represent a RMN site. An ancillary site (such as a SCCPIR) may only have 1 investigator. The Steering Committee Chair and NICHD Project Scientist will be authors. Occasionally, additional authors, both within and outside the RMN

may be appropriate. In these cases, the final decision will be by Network consensus (majority vote of the Steering Committee required).

For the purpose of authorship, only one person from each site owns the primary PI status. This "PI" status is determined by the duration of the time from the start to end date of the site award. It is determined by whoever has served longer. There is NO automatic authorship for other PIs (new or old). They will be treated as any other RMN investigators, and their authorship would be resolved on a case-by-case basis per the current policy (i.e. based on the contribution to specific manuscripts and recommended by the first author and/or writing group). The general order of the authorship is as follows: Group A (the protocol lead PI and site PIs), Group B (important and long term contributors such as some additional site PIs, CREST PIs, DCC second author, core lab author, some co-Investigators), Group C (nominated ad hoc co-authors such as some additional site PIs, DCC third author, and others), Group D (SC Chair, NICHD Project Scientist, and DCC PI), and finally the RMN.

#### **b.** First Author

The lead investigator initiating the protocol, chairing the Protocol Subcommittee will be the first author. The first author will always be expected to prepare the initial draft of the manuscript, after receiving approval from the Network to proceed. The author will prepare the first draft of the manuscript in a timely fashion after receiving all the relevant data analyses from the DCC. The primary author will circulate the final draft to all authors prior to submission, with a timely turnaround of comments from other authors expected. Final decision of the manuscript content will be determined by the Protocol Subcommittee. In the event that the initiating protocol investigator declines first authorship or fails to meet the timeline determined by the Steering Committee (as determined by majority vote) and monitored monthly, the next RMU investigator in the rank order of authors (described below) will be the first author.

#### **c.** Authorship Order

All authorships are expected to meet reasonable criteria as set forth by the International Committee of Medical Journal Editors. (Uniform requirements for manuscripts submitted to biomedical journals: <a href="http://www.icmje.org">http://www.icmje.org</a>. Updated February 2006. Accessed April 4, 2007.) The overall authorship order will be 1) the primary author, 2) RMU investigators, additional outside investigators with a limit of one author per site (e.g. SCCPIR investigators if applicable), followed by the Steering Committee Chair, NIH Project Scientist, and then the authors of the DCC.

**Table 6: RMN Publication Authorship** 

| Authorship Order<br>Category | Description |
|---|---|
| 1 | Lead Investigator of the Protocol (N = 1) |
| 2 | Primary RMN Investigators of the Protocol (N = 6);<br>DCC Investigator (N = 1) |
| 3 | Outside Investigators (i.e. Primary Investigator of SCCPIR sites) (N = to be determined) |
| 4 | Additional Investigators (by Steering Committee vote) (N = to be determined) |
| 5 | Secondary RMN Investigators (N = 7) |
| 6 | Steering Committee Chair (N = 1) |
| 7 | NIH Project Scientist (N = 1) |
| 8 | DCC PI (N = 1) |
| 9 | "for the NICHD Reproductive Medicine Network" |

Table 7: Authorship Order of the RMUs and Outside Sites

| Investigative<br>Sites | # Subjects<br>Rank | Accuracy<br>Rank | Total Rank | Authorship<br>Order |
|---|---|---|---|---|
| А | 1 | 4 | 5 | 3 |
| В | 2 | 7 | 9 | 6 |
| С | 3 | 1 | 4 | 2 |
| D | 4 | 2 | 6 | 4 |
| Е | 5 | 3 | 8 | 5 |
| F | 6 | 5 | 11 | 7 |

It is anticipated that there will be up to 18-25 authors per major manuscript. The authorship order of the RMUs and outside sites will be based upon subject recruitment, data accuracy and promptness of data report according to the chart below:

Data accuracy will be ranked according to the rate of missing or false data entries/randomized subjects at each site. Inquiries that show data was accurately entered will not count against this rate of data inaccuracy. Each site's PI will be responsible for documenting the contributions to the study of that site's authors. In the event the journal editor requires fewer authors even after written documentation of the authors' contribution has been provided, the Steering Committee will vote on the authorship order which will include at a minimum the Lead Investigator and PI of the DCC (or his/her designee) in the positions listed above with the authorship order ending with the footnoted statement "for the Reproductive Medicine Network". The other authors will be referenced in the footnote and listed in the title page.

#### d. Acknowledgement Section

The acknowledgement section will include other investigators and study personnel who contributed substantially to the study by site, as well as members of the Advisory Board and the Data and Safety Monitoring Board. The designation will list the initials of the individuals followed by their highest degree (e.g. C. L. Gnatuk, J.A. Ober, R.N., etc.).

Significant contributions include but are not limited to protocol review, initiation and participation at each site, subject recruitment and enrollment, study conduct, data analysis, and preparation of the manuscript.

#### 9.1.2 Minor Publications

Minor studies are defined as those in which the hypotheses would not be the main elements of Network studies, but in which the study data base would be utilized to test secondary hypotheses. (One example would be testing whether metformin use spares the dose of clomiphene resulting in lower dose needs.) Ideas for "minor studies" will, in general, be proposed by a single individual, who would direct all efforts leading to publication and representation. The results from minor studies would be handled similarly to those from major studies. The "Protocol" is defined as the Concept Protocol/study design of the hypothesis resulting in the publication.

Authorship will follow the Major Publications guidelines above with the exception that the individual leading the minor study would be the first author, followed by the ranked primary RMN investigators involved in developing the Concept Protocol. The Lead Investigator of the minor publication can propose additional investigators who contributed to the study, whose inclusion in the authorship will be voted on by the Steering Committee (majority vote of SC required for inclusion in authorship). Centers may wish to withdraw inclusion from authorship of publications

of minor studies in which only data are contributed, and this will be the decision of the individual site (RMU) PI.

#### 9.2 Ancillary Study

An Ancillary Study is an observational study, conducted as a supplement to a Main Study. By definition, an Ancillary Study involves all or a subset of patients enrolled in a Main Study. An Ancillary Study does not involve any additional participants. To be defined as an Ancillary Study, there must be a need for collection of additional data not already collected in the Main Study. An Ancillary Study may also be designed by another Network investigator, who would serve as the lead investigator and primary author of the paper. Ancillary Studies may be a "single-center" or "multi-center".

A "single-center" Ancillary Study is a study in which all data are collected, stored and analyzed at a single center. The center bears the additional cost of such a study. The study requires approval of the Main Study Protocol Subcommittee and the Steering Committee. The center conducting the study is responsible for the analysis and reporting of the results. Abstracts and manuscripts resulting from data from the single-center Ancillary Study are not subject to the RMN Publications Policies.

A "multi-center" Ancillary Study is defined as one for which data or material (such as specimens) are collected at more than one center, or additional funds for conduct of the study are provided by the NICHD RMN and the DCC provides data analysis. Multi-center Ancillary Studies require the approval of the Main Study Protocol Subcommittee and the Steering Committee.

Authorship will be as per Major Publications above with the exception that the individual leading the Ancillary Study and writing the paper would be the first author, followed by ranked RMN primary investigators, etc. A center not participating in the Ancillary Study would not receive authorship unless by majority vote of the Steering Committee.

#### 9.2.1 Publication Policy on Ancillary Papers

#### <u>Authorship</u>

- 1. RMN will be included as the group author and the acknowledgement will define the entire RMN roster as provided by all PIs.
- 2. The SC Chair, the NICHD Project Scientist, and all PIs will be co-authors upfront. The order will be recommended by the lead author(s).
- 3. Based on the ICJME statement for authorship (http://www.icmje.org/ethical\_1author.html), anyone who makes additional contributions that are documented and substantive will be co-authors. Correcting typos and making grammar suggestions may be below the threshold.
- 4. The responsibilities of the lead authors and the DCC:

- a) If the first and corresponding authorships are offered to a fellow and the PI at a site, this team will recommend the order of the others. The DCC prepares the data for a specific manuscript with a note from the SC that the data should not be used for 'mining' other than answering the predefined questions. The site PI is responsible for the appropriate conduct of the analysis.
- b) The lead author or shared lead authors (at most two) from an RMN or CREST site is given the first choice of one authorship position and the DCC PI makes the second choice. These authors recommend the order of the others. The DCC will assist in the concepts, data preparation, data analysis, and manuscript section writing. If the lead author is not a site PI, the PI plays an administrative and logistic role to ensure that the lead author, whether within the institution, an affiliated CREST site or any other collaborating center, meets the timelines and expectations expressed below, and in return will be offered the second author, or the one preceding the DCC senior author position.

#### **Timeline and expectations**

- 1. The DCC prepares the data set within one month upon receiving the proper specification of the variables and cohort(s), assuming that the data exist in the database.
- 2. Time from receipt of primary data to first draft is not expected to exceed 3 months. Time from first draft to submitted manuscript is not expected to exceed 3 months.
- Co-authors are expected to return comments and edits on manuscript drafts within two
  weeks of the request unless otherwise stated. Failure to respond within this time frame
  will lead to the assumption that the co-author fully approves the draft and has no
  comments or corrections.
- 4. The lead author(s) will be responsible for updating the progress of manuscripts at his/her site (and any CREST sites affiliated with that RMN site) on the Publication Subcommittee conference calls (which will replace Recruitment Subcommittee conference calls) to ensure that reasonable progress is occurring. The Publication Subcommittee can vote to change the authorship if the progress remains slow (e.g., exceeding the timeline expressed above) after two warnings.

#### 9.3 Pilot Study

A Pilot Study is a preliminary study that generates data to help in the design of a Main Study and is the responsibility of the Main Study Protocol Subcommittee. The DCC collaborates with the Protocol Committee to complete the analysis, which may or may not generate an abstract for presentation and/or a manuscript for publication. The DCC writes a Final Report if there is sufficient data to justify one. It is not expected that there will be any secondary analyses resulting from a Pilot Study.

#### 9.4 Related Publications

A related publication is one that has had significant input from members of the RMN Steering Committee at formal meetings in terms of study significance and design. It is distinct from an ancillary publication in that a related publication reports on a study, concept or new methodology that has not been subjected to formal DSMB review and approval. Generally, "Related Publications" will arise from ideas and studies discussed with the Steering Committee, but not voted upon to become formal protocols.

The investigator who initiates, conducts and writes the study, and those whom he/she names will be the sole authors. The authors should acknowledge the contribution of the NICHD Reproductive Medicine Network in the author line of the publication according to the format of the journal.

#### 9.5 Outside Studies

Outside studies will result from the sharing of intellectual property, data and/or specimens with investigators whose protocols have been approved by the Steering Committee, and who comply with all components of those policies. All publications will acknowledge the assistance of the NICHD, the RMN, and the Protocol Subcommittee in making the database available on behalf of the project. In addition, however, a disclaimer will need to be included stating, "The contents of this report represent the views of the authors and do not represent the views of the NICHD Reproductive Medicine Network." The authors will be requested to cc the submitted manuscript to the NICHD program official to ensure compliance. These policies apply to both Network centers and outside centers.

#### 9.6 Presentations

Network data should be presented before national organizations by the Lead Investigators of Main Studies, Ancillary, and Pilot studies. Organizations that might be appropriate include the American Fertility Society, the Society for Gynecologic Investigation, the American College of Obstetricians and Gynecologists, the American Urology Society and other urology or andrology societies. All presentations will be approved by the Publications and Presentations Committee. Once data are published in at least abstract form, all members of the Network can cite them publicly in lectures.

However, investigators should avoid citing specific numbers in review articles and chapters, for this could jeopardize peer review publication. Authorship, First Author, and Author Order are as described for Major Publications, and if there is an authorship limit to the abstract, we will follow the plan above under Major Publications. Oral and poster presentations, including those resulting from secondary analyses at professional societies, must list all authors and participating institutions. In addition, they must include both the NICHD RMN logo and NIH Department of Health and Human Services logos that can be found on the Network web site.

#### 9.7 Timelines

After conclusion of each protocol, the initiating investigator, designated as first author, will consult with the DCC for data analysis and conclusions. The investigator will draft an abstract for distribution to the Network and discussion at the next teleconference or Steering Committee meeting. This should be completed within two months of study completion. Presentation of such abstract may be discussed at this time.

The first author will prepare a draft manuscript within 3 months of data analysis for Network distribution. After incorporating network comments, discussion at the next Steering Committee meeting should allow preparation for publication to ensue in the following 3 months, such that submission will be possible 6 months after data analysis is complete.

#### 9.8 NICHD Clearance

Prior to submitting an abstract for presentation or publication for journal review, the document should be sent to the Project Scientist for submission for NICHD Clearance.

#### 10 References

- 1. Wang A, Fanning L, Anderson DJ, Loughlin KR. Generation of reactive oxygen species by leukocytes and sperm following exposure to urogenital tract infection. Arch Androl 1997;39:11-7.
- 2. Agarwal A, Prabakaran S, Allamaneni SS. Relationship between oxidative stress, varicocele and infertility: a meta-analysis. Reprod Biomed Online 2006;12:630-3.
- 3. O'Flaherty C, Vaisheva F, Hales BF, Chan P, Robaire B. Characterization of sperm chromatin quality in testicular cancer and Hodgkin's lymphoma patients prior to chemotherapy. Hum Reprod 2008;23:1044-52.
- 4. Anderson D, Schmid TE, Baumgartner A, Cemeli-Carratala E, Brinkworth MH, Wood JM. Oestrogenic compounds and oxidative stress (in human sperm and lymphocytes in the Comet assay). Mutation Research/Reviews in Mutation Research 2003;544:173-8.
- 5. Saleh RA, Agarwal A, Sharma RK, Nelson DR, Thomas AJ, Jr. Effect of cigarette smoking on levels of seminal oxidative stress in infertile men: a prospective study. Fertil Steril 2002;78:491-9.
- 6. Jones R, Mann T, Sherins R. Peroxidative breakdown of phospholipids in human spermatozoa, spermicidal properties of fatty acid peroxides, and protective action of seminal plasma. Fertil Steril 1979;31:531-7.
- 7. Aitken RJ. Generation of reactive oxygen species, lipid peroxidation, and human sperm function. Biology of reproduction 1989;41:183-97.
- 8. Gharagozloo P, Aitken RJ. The role of sperm oxidative stress in male infertility and the significance of oral antioxidant therapy. Human Reproduction;26:1628-40.
- 9. Evenson DP, Jost LK, Marshall D, Zinaman MJ, Clegg E, Purvis K *et al.* Utility of the sperm chromatin structure assay as a diagnostic and prognostic tool in the human fertility clinic. Hum Reprod 1999;14:1039-49.
- 10. Guzick DS, Overstreet JW, Factor-Litvak P, Brazil CK, Nakajima ST, Coutifaris C *et al.* Sperm morphology, motility, and concentration in fertile and infertile men. N Engl J Med 2001;345:1388-93.
- 11. Thomson LK. Oxidative deoxyribonucleic acid damage in sperm has a negative impact on clinical pregnancy rate in intrauterine insemination but not intracytoplasmic sperm injection cycles. Fertility and sterility 2011;96:843-7.
- 12. Hu J, Zhu W, Liu W, Fan L. Factors affecting fecundity among sperm donors: a multivariate analysis. Andrologia 2011;43:155-62.
- 13. Bungum M, Humaidan P, Spano M, Jepson K, Bungum L, Giwercman A. The predictive value of sperm chromatin structure assay (SCSA) parameters for the outcome of intrauterine insemination, IVF and ICSI. Human Reproduction 2004;19:1401-8.
- 14. Chi H-J, Chung D-Y, Choi S-Y, Kim J-H, Kim G-Y, Lee J-S *et al.* Integrity of human sperm DNA assessed by the neutral comet assay and its relationship to semen parameters and clinical outcomes for the IVF-ET program. Clin Exp Reprod Med 2011;38:10-7.
- 15. Simon L, Lutton D, McManus J, Lewis SEM. Sperm DNA damage measured by the alkaline Comet assay as an independent predictor of male infertility and in vitro fertilization success. Fertility and sterility 2011;95:652-7.

- 16. Jiang H, He RB, Wang CL, Zhu J. The relationship of sperm DNA fragmentation index with the outcomes of in-vitro fertilisation-embryo transfer and intracytoplasmic sperm injection. Journal of Obstetrics & Gynaecology 2011;31:636-9.
- 17. Meseguer M, Santiso R, Garrido N, GarcÃa-Herrero S, Remohà J, Fernandez JL. Effect of sperm DNA fragmentation on pregnancy outcome depends on oocyte quality. Fertility and sterility 2011;95:124-8.
- 18. Speyer BE, Pizzey AR, Ranieri M, Joshi R, Delhanty JDA, Serhal P. Fall in implantation rates following ICSI with sperm with high DNA fragmentation. Human Reproduction 2010;25:1609-18.
- 19. Henkel R, Hajimohammad M, Stalf T, Hoogendijk C, Mehnert C, Menkveld R *et al.* Influence of deoxyribonucleic acid damage on fertilization and pregnancy. Fertility and sterility 2004;81:965-72.
- 20. Larson-Cook KL, Brannian JD, Hansen KA, Kasperson KM, Aamold ET, Evenson DP. Relationship between the outcomes of assisted reproductive techniques and sperm DNA fragmentation as measured by the sperm chromatin structure assay. Fertility and sterility 2003;80:895-902.
- 21. Sharbatoghli M, Valojerdi M, Amanlou M, Khosravi F, Jafar-abadi M. Relationship of sperm DNA fragmentation, apoptosis and dysfunction of mitochondrial membrane potential with semen parameters and ART outcome after intracytoplasmic sperm injection. Archives of Gynecology and Obstetrics 2012:1-8.
- 22. Esbert M, Pacheco A, Vidal F, Florensa M, Riqueros M, Ballesteros A *et al.* Impact of sperm DNA fragmentation on the outcome of IVF with own or donated oocytes. Reproductive BioMedicine Online 2011;23:704-10.
- 23. Simon L, Brunborg G, Stevenson M, Lutton D, McManus J, Lewis SEM. Clinical significance of sperm DNA damage in assisted reproduction outcome. Human Reproduction 2010;25:1594-608.
- 24. Nijs M, Creemers E, Cox A, Franssen K, Janssen M, Vanheusden E *et al.* Chromomycin A3 staining, sperm chromatin structure assay and hyaluronic acid binding assay as predictors for assisted reproductive outcome. Reproductive BioMedicine Online (Reproductive Healthcare Limited) 2009;19:671-84.
- 25. Avendaño C, Franchi A, Duran H, Oehninger S. DNA fragmentation of normal spermatozoa negatively impacts embryo quality and intracytoplasmic sperm injection outcome. Fertility and sterility 2010;94:549-57.
- 26. Spano M, Cordelli E, Leter G, Lombardo F, Lenzi A, Gandini L. Nuclear chromatin variations in human spermatozoa undergoing swim-up and cryopreservation evaluated by the flow cytometric sperm chromatin structure assay. Mol Hum Reprod 1999;5:29-37.
- 27. Song GJ, Norkus EP, Lewis V. Relationship between seminal ascorbic acid and sperm DNA integrity in infertile men. Int J Androl 2006;29:569-75.
- 28. Lewis SE, Sterling ES, Young IS, Thompson W. Comparison of individual antioxidants of sperm and seminal plasma in fertile and infertile men. Fertil Steril 1997;67:142-7.
- 29. Fraga CG, Motchnik PA, Shigenaga MK, Helbock HJ, Jacob RA, Ames BN. Ascorbic acid protects against endogenous oxidative DNA damage in human sperm. Proc Natl Acad Sci U S A 1991;88:11003-6.

- 30. Balercia G, Armeni T, Mantero F, Principato G, Regoli F. Total oxyradical scavenging capacity toward different reactive oxygen species in seminal plasma and sperm cells. Clin Chem Lab Med 2003;41:13-9.
- 31. Vujkovic M, de Vries JH, Dohle GR, Bonsel GJ, Lindemans J, Macklon NS *et al.* Associations between dietary patterns and semen quality in men undergoing IVF/ICSI treatment. Human Reproduction 2009;24:1304-12.
- 32. Silver EW. Effect of antioxidant intake on sperm chromatin stability in healthy nonsmoking men. Journal of andrology 2005;26:550-6.
- 33. Dawson EB, Harris WA, Powell LC. Relationship between ascorbic acid and male fertility. World Rev Nutr Diet 1990;62:1-26.
- 34. Scott R, MacPherson A, Yates RW, Hussain B, Dixon J. The effect of oral selenium supplementation on human sperm motility. Br J Urol 1998;82:76-80.
- 35. Ciftci H, Verit A, Savas M, Yeni E, Erel O. Effects of N-acetylcysteine on semen parameters and oxidative/antioxidant status. Urology 2009;74:73-6.
- 36. Peivandi S, Abasali K, Narges M. Effects of L-carnitine on infertile men's spermogram; a randomised clinical trial. Journal of Reproduction and Infertility 2010;10:331.
- 37. Omu AE, Al-Azemi MK, Kehinde EO, Anim JT, Oriowo MA, Mathew TC. Indications of the mechanisms involved in improved sperm parameters by zinc therapy. Med Princ Pract 2008;17:108-16.
- 38. Greco E. Reduction of the incidence of sperm DNA fragmentation by oral antioxidant treatment. Journal of andrology 2005;26:349-53.
- 39. Spano M, Bonde JP, Hjollund HI, Kolstad HA, Cordelli E, Leter G. Sperm chromatin damage impairs human fertility. The Danish First Pregnancy Planner Study Team. Fertil Steril 2000;73:43-50.
- 40. Kodama H, Yamaguchi R, Fukuda J, Kasai H, Tanaka T. Increased oxidative deoxyribonucleic acid damage in the spermatozoa of infertile male patients. Fertility and sterility 1997;68:519-24.
- 41. Zini A. Reactive oxygen species in semen of infertile patients: levels of superoxide dismutase- and catalase-like activities in seminal plasma and spermatozoa. International Journal of Andrology 1993;16:183-8.
- 42. Tesarik J, Greco E, Mendoza C. Late, but not early, paternal effect on human embryo development is related to sperm DNA fragmentation. Human Reproduction 2004;19:611-5.
- 43. Robinson L, Gallos ID, Conner SJ, Rajkhowa M, Miller D, Lewis S *et al.* The effect of sperm DNA fragmentation on miscarriage rates: a systematic review and meta-analysis. Human Reproduction;27:2908-17.
- 44. Showell MG, Brown J, Yazdani A, Stankiewicz MT, Hart RJ. Antioxidants for male subfertility. Cochrane Database Syst Rev:CD007411.
- 45. Kessopoulou E, Powers HJ, Sharma KK, Pearson MJ, Russell JM, Cooke ID *et al.* A double-blind randomized placebo cross-over controlled trial using the antioxidant vitamin E to treat reactive oxygen species associated male infertility. Fertil Steril 1995;64:825-31.
- 46. Suleiman SA, Ali ME, Zaki ZM, el-Malik EM, Nasr MA. Lipid peroxidation and human sperm motility: protective role of vitamin E. J Androl 1996;17:530-7.

- 47. Omu AE, Dashti H, Al-Othman S. Treatment of asthenozoospermia with zinc sulphate: andrological, immunological and obstetric outcome. Eur J Obstet Gynecol Reprod Biol 1998;79:179-84.
- 48. Lenzi A, Lombardo F, Sgro P, Salacone P, Caponecchia L, Dondero F *et al.* Use of carnitine therapy in selected cases of male factor infertility: a double-blind crossover trial. Fertil Steril 2003;79:292-300.
- 49. Reichenberg A, Gross R, Weiser M, Bresnahan M, Silverman J, Harlap S *et al.* Advancing paternal age and autism. Arch Gen Psychiatry 2006;63:1026-32.
- 50. Sipos A, Rasmussen F, Harrison G, Tynelius P, Lewis G, Leon DA *et al.* Paternal age and schizophrenia: a population based cohort study. BMJ 2004;329:1070.
- 51. Zhu JL, Madsen KM, Vestergaard M, Olesen AV, Basso O, Olsen J. Paternal age and congenital malformations. Hum Reprod 2005;20:3173-7.
- 52. Hammiche F, Laven JSE, Boxmeer JC, Dohle GR, Steegers EAP, Steegers-Theunissen RPM. Sperm Quality Decline Among Men Below 60 Years of Age Undergoing IVF or ICSI Treatment. J Androl 2011;32:70-6.
- 53. Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HWG, Behre HM *et al.* World Health Organization reference values for human semen characteristics. Human Reproduction Update 2010;16:231-45.
- 54. Bailey RL, Gahche JJ, Lentino CV, Dwyer JT, Engel JS, Thomas PR *et al.* Dietary supplement use in the United States, 2003-2006. J Nutr 2011;141:261-6.
- 55. Panel NS-o-t-S. National Institutes of Health state-of-the-science conference statement: multivitamin/mineral supplements and chronic disease prevention. Am J Clin Nutr 2007;85:257S-64S.
- 56. Tremellen K, Miari G, Froiland D, Thompson J. A randomised control trial examining the effect of an antioxidant (Menevit) on pregnancy outcome during IVF-ICSI treatment. Aust N Z J Obstet Gynaecol 2007;47:216-21.
- 57. Galatioto GP, G.L. G, Angelozzi G, Sacchetti A, Innominato PF, Pace Gea. May antioxidant therapy improve sperm parameters of men with persistent oligospermia after retrograde embolization for varicocele? World Journal of Urology 2008;26:97-102.
- 58. Li Z, Chen GW, Shang XJ, Bai WJ, Han YF, Chen B *et al.* [A controlled randomized trial of the use of combined L-carnitine and acetyl-L-carnitine treatment in men with oligoasthenozoospermia]. Zhonghua Nan Ke Xue 2005;11:761-4.
- 59. Keskes-Ammar L, Feki-Chakroun N, Rebai T, Sahnoun Z, Ghozzi H, Hammami S *et al.* Sperm oxidative stress and the effect of an oral vitamin E and selenium supplement on semen quality in infertile men. Arch Androl 2003;49:83-94.
- 60. Nozha CF, Leila AK, Zouhir S, Hanen G, Z. K, Tarek R. Oxidateive stress and male infertility:comparative study of combined vitamin E/selenium treatment versus vitamin B. Hum Reprod 2001;17:111-2.
- 61. Sesso HD, Buring JE, Christen WG, Kurth T, Belanger C, MacFadyen J *et al.* Vitamins E and C in the prevention of cardiovascular disease in men: the Physicians' Health Study II randomized controlled trial. JAMA 2008;300:2123-33.
- 62. Klein EA, Thompson IM, Jr., Tangen CM, Crowley JJ, Lucia MS, Goodman PJ *et al.* Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA;306:1549-56.

- 63. Safarinejad MR, Safarinejad S. Efficacy of selenium and/or N-acetyl-cysteine for improving semen parameters in infertile men: a double-blind, placebo controlled, randomized study. J Urol 2009;181:741-51.
- 64. Lombardo F, Gandini L, Agarwal A, Sgro P, Dondero F, Lenzi A. A prospective double blind placebo controlled cross over trial of carnitine therapy in selected cases of male infertility. Fertil Steril 2002;78 Suppl 1:68-9.
- 65. Sigman M, Glass S, Campagnone J, Pryor JL. Carnitine for the treatment of idiopathic asthenospermia: a randomized, double-blind, placebo-controlled trial. Fertil Steril 2006;85:1409-14.
- 66. Raigani M, Yaghmaei B, Amirjannti N, Lakpour N, Akhondi MM, Zeraati H *et al.* The micronutrient supplements, zinc sulphate and folic acid, did not ameliorate sperm functional parameters in oligoasthenoteratozoospermic men. Andrologia.
- 67. Azizollahi G, Azizollahi S, Babaei H, Kianinejad M, Baneshi MR, Nematollahi-mahani SN. Effects of supplement therapy on sperm parameters, protamine content and acrosomal integrity of varicocelectomized subjects. J Assist Reprod Genet;30:593-9.
- 68. Zareba P, Colaci DS, Afeiche M, Gaskins AJ, Jorgensen N, Mendiola J *et al.* Semen quality in relation to antioxidant intake in a healthy male population. Fertil Steril;100:1572-9.
- 69. Balercia G. Placebo-controlled double-blind randomized trial on the use of L-carnitine, L-acetylcarnitine, or combined L-carnitine and L-acetylcarnitine in men with idiopathic asthenozoospermia. Fertility and sterility 2005;84:662-71.
- 70. Biagiotti G, Cavallini G, Modenini F, Vitali G, Magli C, Ferraretti A. Prostaglandins pulsed down-regulation enhances carnitine therapy performance in severe idiopathic oligoasthenospermia. Hum Reprod 2003;18 Suppl 1:202.
- 71. Cavallini G, Ferraretti AP, Gianaroli L, Biagiotti G, Vitali G. Cinnoxicam and L-carnitine/acetyl-L-carnitine treatment for idiopathic and varicocele-associated oligoasthenospermia. J Androl 2004;25:761-70; discussion 71-2.
- 72. Lenzi A, Sgro P, Salacone P, Paoli D, Gilio B, Lombardo F *et al.* A placebo-controlled double-blind randomized trial of the use of combined l-carnitine and l-acetyl-carnitine treatment in men with asthenozoospermia. Fertil Steril 2004;81:1578-84.
- 73. Zalata A, Christophe A, Horrobin D, Dhooge W, F. C. Effect of essential fatty acids adn antioxidants dietary supplementation on the oxidative DNA damage of the human spermatozoa. ESHRE 14th annual meeting Goteborg 1998:270-1.
- 74. Blomberg Jensen M, Jorgensen A, Nielsen JE, Bjerrum PJ, Skalkam M, Petersen JH *et al.* Expression of the vitamin D metabolizing enzyme CYP24A1 at the annulus of human spermatozoa may serve as a novel marker of semen quality. Int J Androl;35:499-510.
- 75. Yang B, Sun H, Wan Y, Wang H, Qin W, Yang L *et al.* Associations between testosterone, bone mineral density, vitamin D and semen quality in fertile and infertile Chinese men. Int J Androl;35:783-92.
- 76. Overstreet JW, Brazil CK. Semen analysis. In: L.I. L, Howards SS, eds. Infertility in the male. St. Louis: Mosby-Year Book, 1997:497-90.
- 77. Idem. WHO laboratory manual for the examination of human semen and sperm-cervical mucus interaction. 4th ed. Cambridge, England: Cambridge University Press, 1999.
- 78. Sakkas D, Alvarez JG. Sperm DNA fragmentation: mechanisms of origin, impact on reproductive outcome, and analysis. Fertil Steril 2010;93:1027-36.

- 79. Henkel R, Hoogendijk CF, Bouic PJD, Kruger TF. TUNEL assay and SCSA determine different aspects of sperm DNA damage. Andrologia 2010;42:305-13.
- 80. Evenson DP, Larson KL, Jost LK. Sperm chromatin structure assay: its clinical use for detecting sperm DNA fragmentation in male infertility and comparisons with other techniques. J Androl 2002;23:25-43.
- 81. Sharma RK, Sabanegh E, Mahfouz R, Gupta S, Thiyagarajan A, Agarwal A. TUNEL as a Test for Sperm DNA Damage in the Evaluation of Male Infertility. Urology 2010;76:1380-6.
- 82. Sergerie M, Laforest G, Bujan L, Bissonnette F, Bleau G. Sperm DNA fragmentation: threshold value in male fertility. Hum Reprod 2005;20:3446-51.
- 83. Fedder MD, Jakobsen HB, Giversen I, Christensen LP, Parner ET, Fedder J. An extract of pomegranate fruit and galangal rhizome increases the numbers of motile sperm: a prospective, randomised, controlled, double-blinded trial. PLoS One 2014;9:e108532.
- 84. Louis GMB, Kannan K, Sapra KJ, Maisog J, Sundaram R. Urinary concentrations of Benzophenone-Type Ultraviolet Radiation Filters and Couples' Fecundity. Am J Epidem 2014;180(12) 1168-1175.
- 85. Louis GMB, Chen Z, Kim S, Sapra KJ, Bae J, Kannan K. Urinary concentrations of benzophenone-type ultraviolet light filters and semen quality. Fertil Steril 2015;104:989-996.
- 86. The Endocrine Society. Some sunscreen ingredients may disrupt sperm cell function. ScienceDaily April 1, 2016. www.sciencedialy.com/releases/2016/04/160401111847.htm
- 87. Niederberger C. Editorial. Re: Urinary concentrations of benzophenone-type ultraviolet light filters and semen quality. J Urology 2015;194(6):1711-1712.
- 88. Jennings L, Karia PS, Jambusaria-Pahlajani A, Whalen FM, Schmults CD. The Sun Exposure and Behaviour Inventory (SEBI): validation of an instrument to assess sun exposure and sun protective practices. J Eur Acad Dermatol Venereol 2013;27(6):706-15.
- 89. Matsouka LY, Wortsman J, Hanifan N, Holick MF. Chronic sunscreen use decreases circulating concentrations of 25-hydroxyvitamin D. A preliminary study. Arch Dermatol 1988;124(12):1802-4.

#### 11 Informed Consent

#### 11.1 Informed Consent Template – Male Partners

# University of North Carolina Research Subject Combined Informed Consent and HIPAA Authorization Form

Protocol Title: Males, Antioxidants, and Infertility (MOXI) Trial

Principal Anne Steiner, MD, MPH

Investigator: 4007 Old Clinic Bldg, CB 7570

Chapel Hill, NC 27599

919-966-5283

Emergency 919-966-5283 Monday to Friday, 9AM to 5PM Contact:

919-966-4131 During non-business hours (Ask for

the Reproductive Endocrinologist on call)

# Why am I being asked to volunteer?

You are being invited to participate in a research study. Your participation is voluntary which means you can choose whether or not you want to participate. If you choose not to participate, there will be no loss of benefits to which you are otherwise entitled. Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. The research team is going to talk to you about the research study, and they will give you this consent form to read. You may also decide to discuss it with your family, friends, or family doctor. You may find some of the medical language difficult to understand. Please ask the study doctor and/or the research team about this form. If you decide to participate, you will be asked to sign this form.

# What is the purpose of this research study?

The purpose of this research study is to learn if taking antioxidants can improve male fertility. After 1 year of trying, some couples will not become pregnant. This is called infertility. Male infertility can be caused by DNA damage in sperm. The DNA damage affects the sperm's ability to move or fuse with the egg. Earlier studies have shown that taking antioxidants such as vitamin C, vitamin E, selenium, N-acetylcysteine, L-carnitine, and Zinc might improve this DNA damage. While we know that taking antioxidants might improve DNA damage, we don't know if taking antioxidants can help couples get pregnant. This study will try to determine if taking antioxidants can help infertile couples achieve pregnancy.

You are being invited to participate in this research study because you are an adult male and you and your partner are currently experiencing infertility. To participate in this study you must be trying to get pregnant and living with your female partner.

## How many people will take part in this study?

A total of approximately 790 couples at six institutions will take part in this study, including approximately 50 people from this institution.

# How long will I be in the study?

You will be enrolled in the study for a minimum of 3 months or a maximum of 6 months.

# What am I being asked to do?

If you decide to take part in this study, you and your partner will be asked to complete a brief eligibility questionnaire by phone or in person. If you and your partner qualify to take part in research, you and your partner will be scheduled to come into one of the study centers for a screening visit. This consent form will be reviewed by you and the study coordinator. The purpose of the study, all procedures involved, the risks, and the time commitment related to this study will be discussed. Once all questions have been answered, you will sign this consent form. A copy of this signed consent form will be given to you for your records. Your partner will also sign a separate consent form for participation in this study.

Your <u>screening visit</u> will include the following tests and assessments:

• Complete a questionnaire about your medical history, current medications, infertility history, demographic information, and family history.

 You will be asked to provide a semen sample if you have not had a semen analysis within the past 6 months, which will be used to determine if you are eligible for the study. If you have previously had a semen analysis test done within the past 6 months, we will ask you to sign a medical release form so we can obtain those results.

If you are considered eligible, you will be given 8 questionnaires to complete. A Medical Outcomes Survey (PHQ-9) and the Short Form 12 (SF 12 will assess your daily activities. A Risk Factor for Genetic Disorders questionnaire is completed to determine if you have an increased risk of fathering a child with a genetic disorder. FertiQOL will assess how your infertility affects your thoughts and feelings. The Stop Bang Questionnaire and Epworth Sleepiness Scale (ESS) will assess your sleep habits. The Diet History Questionnaire will be completed to assess your food choices over the past year. The International Index of Erectile Function Survey (IIEF), Psychosexual Daily Questionnaire (PDQ) and qADAM questionnaire will assess your sexual function. The Sun Exposure and Behaviour Inventory (SEBI) will assess your sunscreen usage. You will be free to skip any questions that you would prefer not to answer. If both you and your partner are considered eligible for the study, you will return to the study center to begin study treatment. You will be randomized by a computer system to receive either an antioxidant formulation or placebo. A placebo is a pill that looks just like the antioxidant tablets but does not contain any active medication.

Neither you nor your study team will know which treatment you will receive. Half of participants are expected to receive placebo. You will take the study drug for at least three and up to six months. You will be asked to provide a semen sample at study visit 1 and 90 days later, at study visit 3. We will also obtain approximately 15mL of blood (2 teaspoons) from your vein at study visits 1, 2, 3 and 4. If you and your partner have not become pregnant by the end of three months of study treatment, your partner will receive up to three cycles of infertility treatment in the form of clomiphene citrate and intrauterine insemination (IUI). You will be given an additional 3 months of study medication to take during this time.

This study will include the following tests and assessments:

#### Questionnaires

You will be required to complete the questionnaires described above at your screening visit. In addition, you will also complete the ASA24, which asks you questions about the food you have eaten over the past 24 hours. You will be asked to complete the ASA24 twice throughout this study, at study visit 1 and study visit 3.

#### **Blood Draws**

We will collect approximately 15mL of blood (2 teaspoons) from your vein at four different times throughout the study. These blood draws will be used to look at certain reproductive hormones and vitamin levels in your blood. You will not be given these results.

#### Urine sample

You will provide a urine sample at the first study visit. The urine sample will be used to test for common environmental pollutants. You will not be given these results.

#### Semen Collection

You will be asked to provide a semen sample at screening (if necessary), study visit 1, study visit 3, and for each insemination cycle up to 3 cycles. For this semen analysis test, it is important to not have sex or masturbate for 48 hours prior to collecting your samples.

The following are the instructions you will follow to collect your sample. There is a private room near the lab where specimens can be collected.

- 1. Wash your hands and genitals in the normal way and dry thoroughly.
- 2. Use the cup provided by the study coordinator or the lab. Do not open the container until you are ready to produce the sample.
- 3. Collect the sample by masturbation, putting the entire specimen directly into the cup.
- 4. Do not use lubricants or condoms, as these are harmful to sperm.
- 5. Seal the cup immediately with the lid.

Once you have completed your collection, a semen analysis will be performed to determine the concentration of sperm, motility (moving) and morphology (appearance). You will be given your results.

#### Repository Semen and Blood Specimen Collection

If you consent to the optional part of the study, an additional 2 tablespoons of blood will be drawn for future testing. A portion of your semen will also be collected and stored as part of the repository. These will only be collected if you have consented to the optional part of the study.

#### Study Timeline

#### Study visit 1

Complete a food intake questionnaire (ASA24) online

- Height / Weight
- Measurement of neck, waist and hip circumference
- Provide a semen sample
- Provide a urine sample
- Provide a blood sample
- Randomization
- Pick up one month's supply of study medication

#### Study visit 2 (approximately 30 days after visit 1)

- Provide a blood sample
- · Give old study pill packages, including any leftover pills to study staff
- Pick up 2 month's supply of study medication
- Pick up ovulation strips and pregnancy tests
- Schedule next study visit

#### Study visit 3 (approximately 60 days after visit 2)

- Complete a food intake questionnaire (ASA24) online
- · Give old study pill packages, including any leftover pills to study staff
- Provide a semen sample
- Provide a blood sample
- Pick up 3 month's supply of study medication

#### If you and your partner have not become pregnant:

#### Clomiphene Citrate + Intrauterine Insemination Cycles (up to 3)

- Assist your partner with the injection of hCG trigger medication
- Provide semen for IUI

#### Study visit 4 (approximately 90 days following visit 3)

- Provide a blood sample
- Give old study pill packages to study staff, including any leftover pills

# The following study procedures will be performed once you and your partner have become pregnant:

Pregnancy Ultrasound (between 6 to 9 weeks gestation)

- Pregnancy Status Update: Women will be contacted by study staff (usually between 20 and 22 weeks gestation) to get an update on where she is receiving prenatal care and where she expects to deliver her baby.
- Pregnancy Outcome: Study staff will contact you or your partner after the planned delivery date to obtain pregnancy outcome information such as birth weight, date of delivery, or delivery complications.

# What will happen to the blood sample that I donate to the study?

The sample of blood you donate to the study will not have your name on it and will be stored in a freezer with other samples. The samples will be stored until they are used by the investigators at The University of North Carolina, or their collaborators. The blood will be tested for certain reproductive hormones and vitamin levels in your blood. You will not be able to remove your sample once it is donated.

### What are the possible risks or discomforts?

You may experience minimal discomfort, bruising, and a low risk of infection with the blood draw. We understand that you may not want others to know that you and your partner are trying to get pregnant. We will do our best to protect your confidentiality. In addition, there may be uncommon or previously unknown risks related to the study medication or study procedures. You should report any problems to the researcher. The doses of antioxidants in the supplement have been shown to be safe. Do not take any vitamins in addition to the supplement you are provided as you may then exceed the safe dosage of each vitamin.

#### Risks of Genetic Testing:

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information.

This law generally will protect you in the following ways:

Health insurance companies and group health plans may not request your genetic information that we get from this research.

Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.

Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this Federal law does not protect you or your family against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Also, GINA does not prohibit discrimination of individuals with a genetic disorder that has been diagnosed. However, in order to do everything possible to keep this from happening, the results of this test will NOT be given to anyone outside the study staff. This means that it will not be made available to you, your family members, your private physician, your employer, your insurance company or any other party as allowed by law.

# What if new information becomes available about the study?

During the course of this study, we may find more information that could be important to you. This includes information that, once learned, might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

# What are the possible benefits of the study?

You will not benefit personally from being in this research study. Research is designed to benefit society by gaining new knowledge.

# What other choices do I have if I do not participate?

You do not have to participate in this study to receive treatment for your infertility. Choosing not to participate will not have any effect on your clinical care.

# Will I be paid for being in this study?

You will not be paid to be in the study but you will receive study medications (antioxidant pills or placebo) free of charge. You and your partner will receive six free pregnancy tests and 21 ovulation strips while participating in this study. If you and your partner do not become pregnant following 3 months of study treatment, your partner will receive infertility treatment in the form of clomiphene citrate and intrauterine insemination. If your partner becomes pregnant during the study, you will receive an ultrasound of your baby. You will not have to pay for the antioxidant, placebo, clomiphene citrate, the IUI procedures, or the pregnancy ultrasound.
## Will I have to pay for anything?

For costs of tests and procedures that are only being done for the research study:

- The semen analysis will be provided by the Reproductive Medicine Network at no cost to you.
- You and/or your insurance company will not be charged for the cost of any tests or procedures that are required as part of the research.
- The research-related tests and procedures that will be provided at no cost to you include: semen analysis and research-related blood work and urine collection.

For costs of medical services for care you would receive even if you were not in this research study:

- You and/or your insurance company will be responsible for the cost of routine medications, tests and procedures that you would receive even if you were not in this research.
- You and/or your insurance company will be billed for the costs of these routine tests and procedures in the usual manner.
- You will be responsible for any co-payments, co-insurance and deductibles that are standard for your insurance coverage.
- You will be responsible for any charges not reimbursed by your insurance company.
- Some insurance companies will not pay for routine costs for people taking part in research studies. Before deciding to be in this research you should check with your insurance company to find out what they will pay for.

If you have any questions about costs and insurance, ask the research study doctor or a member of the research team about putting you in touch with a financial counselor to determine exactly what the deductible and co-pay will be for you; this is highly variable depending on your type of insurance."

# What happens if I am injured from being in the study?

All research involves a chance that something bad might happen to you. This may include the risk of personal injury. In spite of all safety measures, you might develop a reaction or injury from being in this study.

We will offer you the care needed to treat injuries directly resulting from taking part in this research. We may bill your insurance company or other third parties, if appropriate,

for the costs of the care you get for the injury, but you may also be responsible for some of them.

There are no plans for the University of North Carolina to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

If you think you have been injured as a result of taking part in this research study, tell the person in charge of the research study as soon as possible. The researcher's name and phone number are listed in the consent form.

#### When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed all visits, and all information has been collected. This study may also be stopped at any time by your physician, the study Sponsor, or the Food and Drug Administration (FDA) without your consent because:

- The Primary Investigator feels it is necessary for your health or safety.
   Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision.
- You have not followed study instructions.
- The Sponsor, the study Principal Investigator, or the Food and Drug Administration (FDA) has decided to stop the study.

If you decide to participate, you are free to leave the study at any time. Withdrawal will not interfere with your future care.

# What information about me may be collected, used or shared with others?

The following information may be used or disclosed for this research project:

- Name, address, telephone number, email address, date of birth
- Medical record number
- Information from your medical records pertaining to your medical history, pregnancy outcome, and information related to all assessments and treatments for this pregnancy

# Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

do the research

- oversee the research
- see if the research was done right.

## Who may use and share information about me?

The following individuals may use or share your information for this research study:

Representatives of the following people/groups <u>within</u> The University of North Carolina may use your health information and share it with other specific groups in connection with this research study.

- The principal investigator, Anne Steiner, MD, MPH
- The University of North Carolina-Chapel Hill Institutional Review Board
- The University of North Carolina-Chapel Hill Human Subjects Protection Office
- The members of the research team working with Anne Steiner
- Other authorized personnel at The University of North Carolina who may have access to your information to perform their daily duties (laboratory personnel, financial personnel, etc.).

# Who, outside of the School of Medicine, might receive my information?

The above people/groups may share your health information with the following people/groups <u>outside</u> The University of North Carolina for their use in connection with this research study. These groups, while monitoring the research study, may also review and/or copy your original The University of North Carolina records.

- The Office of Human Research Protections in the U.S. Department of Health and Human Services
- Food and Drug Administration
- Data Coordination Center at Yale University
- Reproductive Medicine Network of the Eunice Kennedy Shriver National Institute of Child Health and Human Development
- National Institute of Health
- The University of Pennsylvania Institutional Review Board
- The University of Pennsylvania Human Subjects Protection Office

Once your personal health information is disclosed to others outside the School of Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to The University of North Carolina procedures developed to protect your privacy.

# How long may the School of Medicine use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire.

Your information may be held in a research database. However, the School of Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- The University of North Carolina's Institutional Review Board grants permission
- As permitted by law
- As permitted by law

#### Who is sponsoring this study?

This research is funded by the Eunice Kennedy Shriver National Institute of Child Health and Human Development. This means that the research team is being paid by the sponsor for doing the study. The researchers do not, however, have a direct financial interest with the sponsor or in the final results of the study.

# Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigator for the study. If you withdraw your permission, you will not be able to stay in this study.

# Who can see or use my information? How will my personal information be protected?

The investigators and the research team will be able to see your medical records as authorized by you. Results of laboratory tests and clinical procedures done for the monitoring or treatment of your infertility will be placed in your medical record and will be accessible to employees of the health system that are not part of the research team. This information may also be viewed by your insurance company during routine audits.

#### Privacy and confidentiality measures:

Your records that are used in the research at The University of North Carolina will include your study identification number, your initials, and visit date and will be kept in a secured area in a locked file cabinet. Your samples collected for research purposes will be labeled with your study identification number, initials, and visit date and will be stored in a -80 degree freezer.

For research records sent to the Data Coordination Center at Yale University, you will be identified by your study identification number and study visit date. Your blood specimens will not identify you and you cannot be linked to your specimen. The list that matches your name with your code number will be kept in a secured area in a locked file cabinet or in a password-protected electronic document at University of North Carolina.

To help protect your privacy, a Certificate of Confidentiality will be obtained from the federal government. This Certificate means that the researchers cannot be forced (for example by court subpoena) to share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the U.S. government that is used for checking or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate, however, does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information. This means that you and your family should actively protect your own privacy.

The Certificate of Confidentiality does not prevent researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under the following circumstances: child abuse, intent to harm yourself or others, or if you have reportable communicable disease that state or federal law requires us to report such as Tuberculosis, HIV infection, or Syphilis.

In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared. Your de-identified information may be used in the future for other research. Your de-identified data will be shared with the National Institute of Child Health and Human Development on the Data and Specimen Hub which is a resource for investigators to share de-identified research data from studies.

A copy of this consent form will go in to your medical record. This will allow the doctors caring for you to know what study medications or tests you may be receiving as a part of the study and know how to take care of you if you have other health problems or needs during the study.

We will do our best to make sure that the personal information obtained during the course of this research study will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. If this study is being overseen by the Food and Drug Administration (FDA), they may review your research records.

If you test positive for reportable infectious diseases, by law we have to report the infection to the City of Philadelphia Health Department/PA Department of Health. We would report your name, gender, racial/ethnic background, and the month and year you were born.

#### Electronic Medical Records and Research Results

#### What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of the record of your care within a health system. An EMR is simply a computerized version of a paper medical record.

If you are receiving care or have received care within the University of North Carolina Health System (outpatient or inpatient) and are participating in a University of North Carolina research study, results of research-related procedures (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in your existing EMR maintained by UNC.

If you have never received care within UPHS and are participating in a University of North Carolina research study that uses UNC services, an EMR will be created for you for the purpose of maintaining any results of procedures performed as part of this research study. The creation of this EMR is required for your participation in this study. In order to create your EMR, the study team will need to obtain basic information about you that would be similar to the information you would provide the first time you visit a

hospital or medical facility (i.e. your name, the name of your primary doctor, the type of insurance you have). Results of research procedures performed as part of your participation in the study (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in this EMR.

Once placed in your EMR, these results are accessible to appropriate UNC workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by UNC to be appropriate to have access to your EMR (e.g. health insurance company, disability provider, etc.).

# Who can I call with questions, complaints or if I'm concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigator listed on page one of this form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the Institutional Review Board with any question, concerns or complaints at the University of North Carolina by calling 919-966-3113 or by email to IRB subjects@unc.edu.

When you sign this form, you are agreeing to take part in this research study. This means that you have read the consent form, your questions have been answered, and you have decided to volunteer. Your signature also means that you are permitting the University of North Carolina to use your personal health information collected about you for research purposes within our institution. You are also allowing the University of North Carolina to disclose that personal health information to outside organizations or people involved with the operations of this study.

| A copy of this consent form will | be given to you. | |
|---|---|---|
| Name of Subject (Please Prin | t) Signature of Subject | Date |
| Name of Person Obtaining<br>Consent (Please Print) | Signature | Date |

## Optional part(s) of the study

In addition to the main part of the research study, there is another part of the research. You can be in the main part of the research without agreeing to be in this optional part.

### Optional Collection of Saliva for Biomarkers of Stress

As part of an optional part of the study, you will provide us with a sample of saliva. This saliva sample will be tested for biomarkers of stress such as amylase and cortisol. You will be asked to collect the sample upon wakening using a kit provided to you. There are no risks or pain associated with the collection. The sample can be returned in person or via prepaid overnight shipping. Neither you nor your doctor will receive the

results of these tests. There is no cost to you to participate in this optional portion of the study.

You should initial below to indicate your preference for the collection of your saliva for testing:

\_\_\_\_\_ I give my permission for my saliva to be collected and tested for stress biomarkers.

\_\_\_\_ I decline my permission for my saliva to be collected and tested for stress biomarkers.

#### Optional Storage of Blood for RMN Biologic Repository

As part of an optional study, we are obtaining a sample of your blood to be stored in a Biologic Repository by the Reproductive Medicine Network for future use. If you agree, approximately 2 tablespoons of your blood will be collected at the randomization visit and shipped to the RMN Biologic Repository (a central location) and stored for a minimum of 5 years, and perhaps into the future. Your sample will be tested for DNA and to measure other substances in your blood. If you agree to allow us to collect and store a blood sample from you for future use in the repository, your sample will be labeled with a bar code label and unique identifier. These samples will be stored in a locked laboratory at The University of North Carolina, until shipment to the repository. If you consent to the collection of your blood for the repository, it will be kept indefinitely or until the sample is exhausted by the Reproductive Medicine Network. Once your blood has left The University of North Carolina, there is no way to have it returned or withdrawn for testing. You will not be able to withdraw your permission for the use of your blood sample for future use at this time.

We are also collecting blood and urine as a part of this study. If you agree, we would like to retain any leftovers after their use in the study for future use, including measuring other substances from your blood and urine. If you agree to let us retain these samples they will be stored in a locked laboratory at The University of North Carolina, until shipment to the repository. If you consent to the retention of these samples blood and urine for the repository, they will be kept indefinitely or until the sample is exhausted by the Reproductive Medicine Network. Once your blood and urine has left the University of North Carolina, there is no way to have it returned or withdrawn for testing. You will not be able to withdraw your permission for the use of your blood and urine sample for future use at this time.

 These future studies may be helpful in understanding male infertility and the vitamins used in this trial.

- It is unlikely that these studies will have a direct benefit to you.
- The results of these tests will not have an effect on your care.
- Neither your doctor nor you will receive results of these future research tests, nor will the results be put in your health record.
- It is possible that your blood might be used to develop products or tests that could be patented and licensed. There are no plans to provide financial compensation to you should this occur. If you have any questions, you should contact a member of the research team.

| urine for the repo | esitory: |
|---|---|
| I <b>give</b><br>repository for futo | <b>my permission</b> for my blood sample to be collected and sent to the ure testing. |
| I <b>decl</b> i<br>repository for futu | <b>ne my permission</b> for my blood sample to be collected and sent to the ure testing. |
| | <u>of</u> below to indicate your preference for your leftover blood and urine to be t to the repository: |
| | <b>my permission</b> for my leftover blood and urine sample(s) to be retained epository for future testing. |
| | <b>ine my permission</b> my leftover blood and urine sample(s) to be retained epository for future testing. |

#### Optional Storage of Semen for Future Use in Research

As part of an optional study, we want to obtain a sample of your semen to be stored by the RMN for future testing in the RMN Biologic Repository. If you agree, your semen sample will be collected at the screening visit after informed consent. We are also collecting semen as a part of this study. If you agree, we would like to retain any leftover semen not used for the primary study for future research.

Your sample will be stored for a minimum of 5 years, and perhaps further into the future. Your sample will be tested for the chemicals that make up all of your genes and contain your genetic information. These samples can be used for other research in the future

after this study is over. Your sample will not be labeled with any of your personal information, such as your name or a code number. The sample for the repository is labeled with a bar code and cannot be directly linked back to you. They will be available for use in future research studies indefinitely and cannot be removed due to the inability to identify them.

- These future studies may be helpful in understanding male fertility and the vitamins used in this trial.
- It is unlikely that these studies will have a direct benefit to you.
- The results of these tests will not have an effect on your care.
- Neither your doctor nor you will receive results of these future research tests, nor will the results be put in your health record.
- It is possible that your semen sample might be used to develop products or tests that could be patented and licensed. There are no plans to provide financial compensation to you should this occur. If you have any questions, you should contact a member of the research team.

You should *initial* below to indicate your preference for the collection of your semen

| sample f | or the repository: |
|---|---|
| sent to th | _ I <b>give my permission</b> for a portion of my semen sample to be collected and le repository for future testing. |
| | _ I <b>decline my permission</b> for a portion of my semen sample to be collected and |
| sent to th | e repository for future testing. |

#### 11.2 Informed Consent Template – Female Partners

# University of North Carolina Research Subject Combined Informed Consent and HIPAA Authorization Form

Protocol Title: Males, Antioxidants, and Infertility (MOXI) Trial

Principal Anne Steiner, MD, MPH

Investigator: 4007 Old Clinic Bldg, CB 7570

Chapel Hill, NC 27599

919-966-5283

Emergency 919-966-5283 Monday to Friday, 9AM to 5PM Contact:

919-966-4131 During non-business hours (Ask for

the Reproductive Endocrinologist on call)

# Why am I being asked to volunteer?

You are being invited to participate in a research study. Your participation is voluntary which means you can choose whether or not you want to participate. If you choose not to participate, there will be no loss of benefits to which you are otherwise entitled. Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. The research team is going to talk to you about the research study, and they will give you this consent form to read. You may also decide to discuss it with your family, friends, or family doctor. You may find some of the medical language difficult to understand. Please ask the study doctor and/or the research team about this form. If you decide to participate, you will be asked to sign this form.

#### What is the purpose of this research study?

The purpose of this research study is to learn if taking antioxidants can improve male fertility. After 1 year of trying, some couples will not become pregnant. This is called infertility. Male infertility can be caused by DNA damage in sperm. The DNA damage affects the sperm's ability to move or fuse with the egg. Earlier studies have shown that taking antioxidants such as vitamin C, vitamin E, selenium, N-acetylcysteine, L-carnitine, and Zinc might improve this DNA damage. While we know that taking antioxidants might improve DNA damage, we don't know if taking antioxidants can help couples get pregnant. This study will try to determine if taking antioxidants can help infertile couples achieve pregnancy.

You are being invited to participate in this research study because you are an adult female and you and your partner are currently experiencing infertility. To participate in this study, you must be trying to get pregnant and living with your male partner.

# How many people will take part in this study?

A total of approximately 790 couples at six institutions will take part in this study, including approximately 50 people from this institution.

### How long will I be in the study?

If you achieve pregnancy during this study, you will be enrolled in this study from the time you sign this consent form until you have your early pregnancy ultrasound. Study staff will contact you to obtain information about your pregnancy outcome. If you and your partner do not become pregnant, you will be enrolled in this study from the time you sign this consent form to the time your partner has completed six months of study treatment.

# What am I being asked to do?

If you decide to take part in this study, you and your partner will be asked to complete a brief eligibility questionnaire by phone or in person. If you and your partner qualify to take part in research, you and your partner will be scheduled to come into one of the study centers for a screening visit. This consent form will be reviewed by you and the study coordinator. The purpose of the study, all procedures involved, the risks, and the time commitment related to this study will be discussed. Once all questions have been answered, you will sign this consent form. A copy of this signed consent form will be given to you for your records. Your partner will also sign a separate consent form for participation in this study.

Your <u>screening visit</u> will include the following tests and assessments:

- Your past medical and menstrual history will be recorded. This form will ask a series of questions about your medical health, family health history, reproductive and gynecological history, pregnancy history, and current use of medications.
- Your height, weight, vital signs (blood pressure and pulse) and neck circumference will be collected and your body mass index (BMI) will be calculated.
- You will be given 9 questionnaires to complete. A Risk Factor for Genetic Disorders questionnaire is completed to determine if you have an increased risk of having a baby with a genetic disorder. Any potential problems that may lead to complications during pregnancy will be addressed at this time and we may refer you to a genetics counselor prior to starting the study. The Female Sexual Function Index (FSFI) and Female Sexual Distress Scale (FSDS) will assess your sexual function. A Medical Outcomes Survey (PHQ-9) and the Short Form 12 (SF 12) will assess your daily activities. FertiQOL will assess how your infertility affects your thoughts and feelings. The Stop Bang Questionnaire and Epworth Sleepiness Scale (ESS) will assess your sleep habits. The Dietary History Questionnaire II will be completed to assess your current dietary intake. You will be free to skip any questions that you would prefer not to answer.
- The following tests will be done if you have not had them done previously. If you
  have had them done, you will need to sign a medical record release so that we may
  obtain these results.
  - Blood work may be drawn to determine your eligibility for the study. Tests that may be drawn are a progesterone level, FSH, estradiol, or AMH level.
  - o If you have had not had a test within the past 3 years to determine that your fallopian tubes are open, a sonohysterogram (SHG) or hysterosalpingogram (HSG) will be completed. During the SHG, sterile saline fluid is injected through an intrauterine catheter that contains a balloon. The balloon is inflated and the shape of your uterus can be seen and the fluid that accumulates in the back area of your uterus determines that at least one fallopian tube is open. If it can't be determined by the SHG, it will be necessary for a different procedure to be performed. An HSG procedure is done in the radiology department using radio-opaque contrast dye that is injected into the uterus and is visualized flowing through the fallopian tube. If you have been pregnant within the last three years and your pregnancy and delivery were uncomplicated, the SHG or HSG may not be necessary.
  - A physical exam will be performed by the physician if not done within the past 12 months.
  - A pap smear will be collected if you are 21 or older and have not had one within the time period specified by current guidelines.

If you consent to the optional part of the study, an additional 2 tablespoons of blood will be drawn and a urine sample collected for the biological repository.

If you and your partner are considered eligible for the study, your partner will return to the study center to begin study treatment. Your partner will be randomized by a computer system to receive either an antioxidant formulation or placebo. A placebo is a pill that looks just like the antioxidant tablets but does not contain any active medication.

Neither you, your partner, nor your study team will know which treatment he will receive. Half of participants are expected to receive placebo. He will take the study drug for at least three and up to six months. If you are not pregnant by the end of the third month of study treatment, you will receive up to three cycles of infertility treatment in form of clomiphene citrate and intrauterine insemination (IUI) while he is on treatment.

The following procedures will be performed if you and your partner have **not** become pregnant following the third study visit (after 3 months of study treatment):

#### <u>Baseline Visit – Infertility Treatment (clomiphene citrate + IUI)</u>

You will call on the first day of your next menstrual period following your partner's third study visit to schedule your baseline visit for infertility treatment between menstrual cycle day 1-5. At this visit the following procedures will occur:

- Transvaginal Ultrasound. This involves inserting an ultrasound probe into your vagina to visualize your ovaries and uterus. Measurements and ultrasound pictures will be recorded of your ovaries and uterus.
- Your medications will be given to you at this time. You will receive clomiphene citrate. You will be instructed to begin your medications if your urine pregnancy test is negative and your ultrasound results are within a normal range. You will also receive hCG injection medication to be used when directed by your physician prior to your insemination. You and your partner will be taught the technique for administering an intramuscular injection.

#### Monitor Visits (cycle day 8 to 12 and then beyond as required)

You will be required to return to the clinic within 3 days after completing your 5 day treatment of clomiphene citrate. A transvaginal ultrasound will be performed. You may be required to return to the clinic regularly for additional monitoring visits until you have met the criteria for hCG administration. These visits will be individualized and based on your physician's discretion.

When your main follicle (cyst which contains an egg) gets to a certain size, you will be instructed to self or partner-administer an injection of hCG at a dose of 10,000 IU. A cycle may be cancelled if the lead follicles become too large or too small after 18 days of monitoring.

#### Intrauterine Insemination Visit

You must return to the clinic within 44 hours of the hCG shot. Your partner will provide a semen sample. This sample will be washed and prepared for the insemination. A speculum will be placed in your vagina and a thin flexible catheter will be placed into your cervix. The sperm will be injected through the catheter and into your uterus.

#### **Urine Pregnancy Test**

Two weeks after insemination you will do a urine pregnancy test at home and call the study coordinator with your results.

If you have a positive urine pregnancy test, you will be required to return to the clinic for a blood pregnancy test (quantitative bhCG). If your bhCG is positive you will return 2 days later for repeat bhCG to check for a rising level. If the level is not rising, you will begin the next cycle of treatment with the start of your menstrual cycle. If the bhCG level has risen, you will be schedule for an ultrasound approximately 14-21 days after the positive result.

#### Follow up Initiation of Cycle 2 & 3

If your urine pregnancy test is negative after a cycle, you may start another cycle of treatment. You may participate for a maximum of 3 cycles. A cycle may be cancelled if any significant adverse reactions develop in response to the medications, if you are unable to have the hCG injection, or if you request the cycle to be cancelled. The study coordinator will provide you with instructions to start your medication on cycle day 3 (+ or -2 days). The study physician may change the start dose of your Clomiphene Citrate. You will be scheduled for a return monitoring visit during menstrual cycle day 8-12.

The following study procedures will be performed once you and your partner **have** become pregnant:

- Pregnancy Ultrasound (between 6 to 9 weeks gestation)
- Pregnancy Status Update: Women will be contacted by study staff (usually between 20 and 22 weeks gestation) to get an update on where she is receiving prenatal care and where she expects to deliver her baby.

 Pregnancy Outcome: Study staff will contact you or your partner after the planned delivery date to obtain pregnancy outcome information such as birth weight, date of delivery, or delivery complications.

#### Pregnancy Ultrasound:

This transvaginal ultrasound will determine the location of your pregnancy, number of gestational sacs and to assess fetal heartbeat.

#### **Pregnancy Care:**

You may need additional ultrasounds done to evaluate the progress of the pregnancy if necessary. Pregnancy care is not part of this study. You will be scheduled with your obstetrician for follow up prenatal care. If you do not have a doctor who delivers babies, you will be referred to one. Before being released from the study, you will be asked to sign a medical release form so the study coordinator can obtain your pregnancy and delivery information. You will be contacted between 12 and 22 weeks to see how your pregnancy is progressing.

### What will happen to the blood sample that I donate to the study?

The sample of blood you donate to the study will not have your name on it and will be stored in a freezer with other samples. The samples will be stored until they are used by the investigators at The University of North Carolina, or their collaborators. The blood will be tested for certain reproductive hormones and vitamin levels in your blood. You will not be able to remove your sample once it is donated.

# What are the possible risks or discomforts?

You may experience minimal discomfort, bruising, and a low risk of infection with the blood draw. You may experience abdominal or pelvic discomfort due to the transvaginal ultrasound used in this study.

Risks associated with the sonohystogram/hysterosalpingogram include pain, bleeding, damage to the uterus, pelvic infection, interrupting an unrecognized pregnancy, small amount of radiation exposure, allergic reaction to the radio-opaque dye.

Risks associated with clomiphene citrate: visual changes (such as blurring of vision, double vision, light sensitivity), abdominal pain, nausea, vomiting, constipation, mood changes, depression, headache, hot flashes, respiratory difficulty, fatigue, abnormal endometrial thickening, multiple pregnancies, formation of ovarian cyst causing ovarian hyperstimulation syndrome, ovarian enlargement, breast discomfort, abnormal uterine

bleeding, bloating, hair loss, arrhythmias, chest pain, allergic reaction, palpitations, and stroke or pulmonary embolism.

Risks associated with intrauterine insemination include Vasovagal response (feeling lightheaded, dizzy, sweating); possible infection.

We understand that you may not want others to know that you and your partner are trying to get pregnant. We will do our best to protect your confidentiality. In addition, there may be uncommon or previously unknown risks related to the study medication or study procedures. You should report any problems to the researcher.

#### **Risks of Genetic Testing:**

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information.

This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that
  we get from this research when making a decision to hire, promote, or fire you or
  when setting the terms of your employment.

Be aware that this Federal law does not protect you or your family against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Also, GINA does not prohibit discrimination of individuals with a genetic disorder that has been diagnosed. However, in order to do everything possible to keep this from happening, the results of this test will NOT be given to anyone outside the study staff. This means that it will not be made available to you, your family members, your private physician, your employer, your insurance company or any other party as allowed by law.

## What if new information becomes available about the study?

During the course of this study, we may find more information that could be important to you. This includes information that, once learned, might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

## What are the possible benefits of the study?

You will not benefit personally from being in this research study. Research is designed to benefit society by gaining new knowledge.

### What other choices do I have if I do not participate?

You do not have to participate in this study to receive treatment for your infertility. Choosing not to participate will not have any effect on your clinical care.

#### Will I be paid for being in this study?

You will not be paid to be in this study. You and your partner will receive 6 free pregnancy tests and 21 ovulation strips while participating in this study. If you and your partner do not become pregnant following 3 months of study treatment, you will receive infertility treatment in the form of clomiphene citrate, human chorionic gonadotropin, and intrauterine insemination. If you become pregnant during the study, you will receive an ultrasound of your baby. You will not have to pay for the clomiphene citrate, human chorionic gonadotropin, the IUI procedures, or the pregnancy ultrasound.

# Will I have to pay for anything?

For costs of tests and procedures that are <u>only</u> being done for the research study:

- The Clomiphene Citrate and hCG injection will be provided by RMN at no cost to you.
- You and/or your insurance company will not be charged for the cost of any tests or procedures that are required as part of the research.
- The research-related tests and procedures that will be provided at no cost to you include:
  - All study required blood tests
  - Physical exam
  - Transvaginal ultrasound (s)
  - Tests ordered for the study to determine tubal patency such as a sonohystogram
  - Intrauterine inseminations
  - Ovulation predictor kits
  - Urine pregnancy tests
  - Supplies for injection medication such as; syringes, alcohol swabs, gauze, and band-aids

#### 1 Pregnancy Ultrasound

For costs of medical services for care you would receive even if you were not in this research study:

- You and/or your insurance company will be responsible for the cost of routine medications, tests and procedures that you would receive even if you were not in this research.
- You and/or your insurance company will be billed for the costs of these routine tests and procedures in the usual manner.
- You will be responsible for any co-payments, co-insurance and deductibles that are standard for your insurance coverage.
- You will be responsible for any charges not reimbursed by your insurance company.
- Some insurance companies will not pay for routine costs for people taking part in research studies. Before deciding to be in this research you should check with your insurance company to find out what they will pay for.

The following is a list of the non-covered services related to this study:

- Prior testing
- Rubella, Varicella, & HIV testing
- Pap Smear
- Carrier screening for genetic diseases
- Doxycycline prescription for after the HSG procedure, if necessary
- Remaining obstetrical ultrasounds after the first one
- Pregnancy care and delivery costs

If you have any questions about costs and insurance, ask the research study doctor or a member of the research team about putting you in touch with a financial counselor to determine exactly what the deductible and co-pay will be for you; this is highly variable depending on your type of insurance.

# What happens if I am injured from being in the study?

All research involves a chance that something bad might happen to you. This may include the risk of personal injury. In spite of all safety measures, you might develop a reaction or injury from being in this study.

We will offer you the care needed to treat injuries directly resulting from taking part in this research. We may bill your insurance company or other third parties, if appropriate, for the costs of the care you get for the injury, but you may also be responsible for some of them.

There are no plans for the University of North Carolina to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

If you think you have been injured as a result of taking part in this research study, tell the person in charge of the research study as soon as possible. The researcher's name and phone number are listed in the consent form.

## When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed all visits, and all information has been collected. This study may also be stopped at any time by your physician, the study Sponsor, or the Food and Drug Administration (FDA) without your consent because:

- The Primary Investigator feels it is necessary for your health or safety. Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision.
- You have not followed study instructions.
- The Sponsor, the study Principal Investigator, or the Food and Drug Administration (FDA) has decided to stop the study.

If you decide to participate, you are free to leave the study at anytime. Withdrawal will not interfere with your future care.

# What information about me may be collected, used or shared with others?

The following information may be used or disclosed for this research project:

- Name, address, telephone number, email address, date of birth
- Medical record number
- Information from your medical records pertaining to your medical history, pregnancy outcome, and information related to all assessments and treatments for this pregnancy

# Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

- do the research
- oversee the research
- see if the research was done right.

### Who may use and share information about me?

The following individuals may use or share your information for this research study:

Representatives of the following people/groups <u>within</u> The University of North Carolina may use your health information and share it with other specific groups in connection with this research study.

- The principal investigator, Anne Steiner, MD, MPH
- The University of North Carolina Institutional Review Board
- The University of North Carolina Human Subjects Protection Office
- The members of the research team working with Anne Steiner
- Other authorized personnel at The University of North Carolina who may have access to your information to perform their daily duties (laboratory personnel, financial personnel, etc.)

# Who, outside of the School of Medicine, might receive my information?

The above people/groups may share your health information with the following people/groups <u>outside</u> The University of North Carolina for their use in connection with this research study. These groups, while monitoring the research study, may also review and/or copy your original The University of North Carolina records.

- The Office of Human Research Protections in the U.S. Department of Health and Human Services
- Food and Drug Administration
- Data Coordination Center at Yale University
- Institutional Review board at The University of Pennsylvania
- Reproductive Medicine Network of the Eunice Kennedy Shriver National Institute of Child Health and Human Development
- National Institute of Health
- City of Chapel Hill Health Department/NC Department of Health

Once your personal health information is disclosed to others outside the School of Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to The University of North Carolina procedures developed to protect your privacy.

# How long may the School of Medicine use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire.

Your information may be held in a research database. However, the School of Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- The University of North Carolina's Institutional Review Board grants permission
- As permitted by law
- As permitted by law

# Who is sponsoring this study?

This research is funded by the National Institute of Child Health and Human Development. This means that the research team is being paid by the sponsor for doing the study. The researchers do not, however, have a direct financial interest with the sponsor or in the final results of the study.

# Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigator for the study. If you withdraw your permission, you will not be able to stay in this study.

# Who can see or use my information? How will my personal information be protected?

The investigators and the research team will be able to see your medical records as authorized by you. Results of laboratory tests and clinical procedures done for the

monitoring or treatment of your infertility will be placed in your medical record and will be accessible to employees of the health system that are not part of the research team. This information may also be viewed by your insurance company during routine audits.

#### Privacy and confidentiality measures:

Your records that are used in the research at The University of North Carolina will include your study identification number, your initials, and visit date and will be kept in a secured area in a locked file cabinet. Your samples collected for research purposes will be labeled with your study identification number, initials, and visit date and will be stored in a -80 degree freezer.

For research records sent to the Data Coordination Center at Yale University, you will be identified by your study identification number and study visit date. Your blood specimens will not identify you and you cannot be linked to your specimen. The list that matches your name with your code number will be kept in a secured area in a locked file cabinet or in a password-protected electronic document at University of North Carolina

To help protect your privacy, a Certificate of Confidentiality will be obtained from the federal government. This Certificate means that the researchers cannot be forced (for example by court subpoena) to share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the U.S. government that is used for checking or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate, however, does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information. This means that you and your family should actively protect your own privacy.

The Certificate of Confidentiality does not prevent researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in

the research project under the following circumstances: child abuse, intent to harm yourself or others, or if you have reportable communicable disease that state or federal law requires us to report such as Tuberculosis, HIV infection, or Syphilis.

In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared. Your de-identified information may be used in the future for other research. Your de-identified data will be shared with the National Institute of Child Health and Human Development on the Data and Specimen Hub which is a resource for investigators to share de-identified research data from studies.

A copy of this consent form will go in to your medical record. This will allow the doctors caring for you to know what study medications or tests you may be receiving as a part of the study and know how to take care of you if you have other health problems or needs during the study.

We will do our best to make sure that the personal information obtained during the course of this research study will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. If this study is being overseen by the Food and Drug Administration (FDA), they may review your research records.

If you test positive for reportable infectious diseases, by law we have to report the infection to the City of Chapel Hill Health Department/NC Department of Health. We would report your name, gender, racial/ethnic background, and the month and year you were born.

This is to keep track of how many people in the U.S. have HIV infection. It is also to make sure that states get enough money from the federal government to support the medical care of people living with HIV. The Health Department does not share the names of HIV infected people with anyone else. It removes all personal identifiers, such as your name, before giving information on the number of HIV infections to the federal government.

#### Electronic Medical Records and Research Results

What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of the record of your care within a health system. An EMR is simply a computerized version of a paper medical record.

If you are receiving care or have received care within the University of North Carolina (outpatient or inpatient) and are participating in a University of North Carolina research study, results of research-related procedures (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in your existing EMR maintained by UNC Healthcare.

If you have never received care within UNC and are participating in a University of North Carolina research study that uses UNC services, an EMR will be created for you for the purpose of maintaining any results of procedures performed as part of this research study. The creation of this EMR is required for your participation in this study. In order to create your EMR, the study team will need to obtain basic information about you that would be similar to the information you would provide the first time you visit a hospital or medical facility (i.e. your name, the name of your primary doctor, the type of insurance you have). Results of research procedures performed as part of your participation in the study (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in this EMR.

Once placed in your EMR, these results are accessible to appropriate UNC workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by UNC to be appropriate to have access to your EMR (e.g. health insurance company, disability provider, etc.).

# Optional part(s) of the study

In addition to the main part of the research study, there is another part of the research. You can be in the main part of the research without agreeing to be in this optional part.

#### Optional Collection of Saliva for Biomarkers of Stress

As part of an optional part of the study, you will provide us with a sample of saliva. This saliva sample will be tested for biomarkers of stress such as amylase and cortisol. You will be asked to collect the sample upon wakening using a kit provided to you. There are no risks or pain associated with the collection. The sample can be returned in person or via prepaid overnight shipping. Neither you nor your doctor will receive the results of these tests. There is no cost to you to participate in this optional portion of the study.

| You should testing: | initial below to indicate your preference for the collection of your saliva for |
|---|---|
| l<br>biomarkers. | give my permission for my saliva to be collected and tested for stress |
| | decline my permission for my saliva to be collected and tested for stress |
| biomarkers. | |

#### Optional Storage of Blood and Urine for RMN Biologic Repository

As part of an optional study, we are obtaining a sample of your blood and urine to be stored in a Biologic Repository by the Reproductive Medicine Network for future use. If you agree, approximately 2 tablespoons of your blood will be collected at the randomization visit and shipped to the RMN Biologic Repository (a central location) and stored for a minimum of 5 years, and perhaps into the future. Your sample will be tested for DNA and to measure other substances in your blood and urine. If you agree to allow us to collect and store a blood and urine sample from you for future use in the repository, your sample will be labeled with a bar code label and unique identifier. These samples will be stored in a locked laboratory at The University of North Carolina, until shipment to the repository. If you consent to the collection of your blood and urine for the repository, it will be kept indefinitely or until the sample is exhausted by the Reproductive Medicine Network. Once your blood and urine has left University of North Carolina, there is no way to have it returned or withdrawn for testing. You will not be able to withdraw your permission for the use of your blood and urine sample for future use at this time.

- These future studies may be helpful in understanding male infertility and the vitamins used in this trial.
- It is unlikely that these studies will have a direct benefit to you.
- The results of these tests will not have an effect on your care.
- Neither your doctor nor you will receive results of these future research tests, nor will the results be put in your health record.
- It is possible that your blood might be used to develop products or tests that could be patented and licensed. There are no plans to provide financial compensation to you should this occur. If you have any questions, you should contact a member of the research team.

| You should <u>initial</u> below to indicate your preference for the collection of y urine for the repository: | our blood and |
|---|---|
| I <b>give my permission</b> for my blood and urine sample to be co<br>the repository for future testing. | llected and sent to |
| I <b>decline my permission</b> for my blood and urine sample to be sent to the repository for future testing. | e collected and |
| Who can I call with questions, complaints or if I'm concerr my rights as a research subject? | ned about |
| If you have questions, concerns or complaints regarding your participation research study or if you have any questions about your rights as a resear should speak with the Principal Investigator listed on page one of this form member of the research team cannot be reached or you want to talk to see than those working on the study, you may contact the Institutional Review any question, concerns or complaints at the University of North Carolina 1966-3113 or by email to IRB_subjects@unc.edu. | rch subject, you<br>m. If a<br>omeone other<br>v Board with |
| When you sign this form, you are agreeing to take part in this research is This means that you have read the consent form, your questions have be answered, and you have decided to volunteer. Your signature also mean you are permitting the University of North Carolina to use your personal information collected about you for research purposes within our institution are also allowing the University of North Carolina to disclose that person information to outside organizations or people involved with the operation study. | een<br>ans that<br>health<br>ion. You<br>nal health |
| By signing below, you also indicate that you have read the information write above and have indicated your choices for the optional part(s) of the reseastudy. | |
| A copy of this consent form will be given to you. | |
| Name of Subject (Please Print) Signature of Subject | Date |

Your signature below means that you have explained the optional part(s) to the research to the subject or subject representative and have answered any questions he/she has about the research.

2016.10.12

| Name of Person Obtaining<br>Consent (Please Print) | Signature | Date |
|----------------------------------------------------|-----------|------|

# 12 Appendix A: Male Medical History Questionnaire



**Male Medical History** 

Source Document
Reproductive Medicine Network
Males, Antioxidants, and Infertility (MOXI) Trial

### **MEDICAL HISTORY**

Do you have a history of any of the following medical conditions or problems?

| , | | | | |
|---|---|---|---|---|
| Body System | Response<br>(If NO, skip to<br>next<br>question) | Condition/Problem | Currently<br>Symptomatic | Requires<br>Medication |
| 1. Problems with | Yes | ☐ Hearing loss | Yes | Yes |
| your head, ears,<br>eyes, nose or | □No | Blindness | | |
| throat? | | Sinus | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 2. Problems with | Yes | Stroke | Yes | Yes |
| your brain, nervous system or any psychiatric conditions? | □ No | Migraines | | |
| | | Seizures | | |
| | | ☐ CVA/TIA | | |
| | | ☐ Depression | | |
| | | ☐ Anxiety | | |
| | | ☐ Bipolar disorder | | |
| | | ☐ Schizophrenia/Psychosis | | |
| | | ☐ Obsessive-Compulsive Disorder | | |
| | | ☐ ADD/ADHD | | |
| | | ☐ Eating Disorder (anorexia, bulimia) | | |
| i | l | 1 | 1 | 1 |

| | | ☐ Post-Traumatic Stress | | |
|---|---|---|---|---|
| | | ☐ Acute Stress Disorder | | |
| | | ☐ Substance/Alcohol Abuse | | |
| | | ☐ Phobia/Agoraphobia | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 3. Problems with | Yes | Asthma | Yes | Yes |
| your respiratory system? | □No | ☐ Pneumonia | | |
| | | ☐ COPD | | |
| | | ☐ Emphysema | | |
| | | □тв | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 4. Problems with | Yes | ☐ Previous heart attack | Yes | Yes |
| your heart or cardiovascular | □No | ☐ Congenital heart defect | | |
| system? | | ☐ Palpitations | | |
| | | ☐ Arrhythmias | | |
| | | ☐ Valve disease | | |
| | | ☐ Angina | | |
| | | ☐ CHF | | |
| | | Hypertension | | |
| | | ☐ Syncope | | |
| | | ☐ Blood clot in leg, lung, brain | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |

| 5. Problems with | Yes | ☐ Arthritis | Yes | Yes |
|----------------------------------|------|------------------------|-----|-----|
| your muscles, joints, bones or | ☐ No | Lupus | | |
| musculoskeletal system? | | Osteoporosis | | |
| bystom: | | ☐ Gout | | |
| | | ☐ Disc disease | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 6. Problems with | Yes | ☐ Irritable bowel | Yes | Yes |
| your gastrointestinal system? | ☐ No | ☐ GI cancer | | |
| | | ☐ Liver disease | | |
| | | ☐ Peptic ulcer | | |
| | | ☐ GERD | | |
| | | ☐ Hepatitis | | |
| | | ☐ Pancreatitis | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 7. Problems with | Yes | Clotting | Yes | Yes |
| your blood and metabolic system? | ☐ No | ☐ Anemia | | |
| | | ☐ Hyperlipidemia | | |
| | | ☐ Diabetes | | |
| | | ☐ Hyper/hypothyroidism | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 8. Problems with the | Yes | ☐ Cancer | Yes | Yes |
| whole body? | ☐ No | Alcoholism | | |
| | | ☐ Drug abuse | | |
| | İ | | İ | 1 |

| | Aller | gies | | |
|---|---|---|---|---|
| | ☐ Fatig | gue | | |
| | ☐ Wea | kness | | |
| | | Jery (specify): | | |
| | Othe | er (specify): | | L |
| 9. Have you ever been trea | ted for cancer? | ☐ Yes ☐No → Skip to Ques | etion #10 | |
| 9a. If yes, specify type of | | Testicular | HOIT # 10 | |
| ou. If you, opeony type t | n carroor. | ☐ Hodgkin's | | |
| | | Lymphoma | | |
| | | ☐ Leukemia | | |
| | | <br>☐ Bladder | | |
| | | ☐ Prostate | | |
| | | Other | | |
| (specify): | | | | |
| 9b. Was surgery used fo | or treatment? | ☐ Yes ☐ No | | |
| 9c. Was chemotherapy | used for treatment? | ☐ Yes ☐ No → Skip to Que | stion #9d | |
| 9c1. If yes, specify | v type: (check all that a | pply) ☐ Cisplatinum chemo<br>(Platinol) | otherapy | |
| | | ☐ Cyclophosphamide | e (Cytoxan) | |
| | | y | , - | |
| | | ☐ Nitrosoureas (Carr<br>Lomustine) | nustine, | |
| | | L-phenylalanine m<br>(Alkeran) | ustard | |
| | | ☐ Bleomycin (Blenox<br>Bleomycin) | ane, | |
| | | ☐ Chlorambucil (Leul | keran) | |
| | | <br>☐ Procarbazine (Natı | · | |
| | | ☐ Nitrogen mustard | (Mustargen) | |
| | | Other | | |
| (specify): | | | | |

| | Unknown |
|---|---|
| 9d. Was radiation used for treatment?<br>#10 | ☐ Yes ☐ No → Skip to Question |
| 9d1. If yes, specify location: | ☐ Pelvic |
| | ☐ Brain |
| | ☐ Total body irradiation |
| | Other |
| (specify): | _ |
| 10. Have you had a high fever (≥103 °F) in the last six | x months? ☐ Yes ☐ No |
| 11. Have you ever been diagnosed with a sexually | rtransmitted infection/disease? |
| | ☐ Yes ☐ No → Skip to Question #12 |
| 11a. Type of STD/STI: (check all that apply) | ☐ Gonorrhea |
| | ☐ Chlamydia |
| | ☐ Syphillis |
| | ☐ Herpes Simplex Virus (HSV) |
| | ☐ Human Papillomavirus<br>(HPV) |
| | ☐ Trichomoniasis (Trich) |
| | ☐ Other |
| | (specify): |
| 11b. Did you receive treatment? | ☐ Yes ☐ No |
| 12. Have you ever had a urinary tract infection (bladde | er infection)? |
| 12. Have you ever had a annaly had micetion (wada | ☐ Yes ☐ No → Skip to Question #13 |
| 12a. Indicate number of times: | —— |
| 13. Have you ever had epididymitis? | ☐ Yes ☐ No → Skip to Question #14 |
| 13a. Indicate number of times: | |
| roa. maioato nambor of timos. | |
| 14. Have you ever had prostatitis? | ☐ Yes ☐ No → Skip to Question #15 |
| 14a. Indicate number of times: | |

| 15. Have you ever had testicular torsion (twist)? | ☐ Yes ☐ No → Skip to Question #16 |
|---|---|
| 15a. Indicate number of times: | |
| 16. Have you ever been treated for an undescended tes | |
| | ☐ Yes☐ No → Skip to Question #17 |
| 16a. Indicate type: | ☐ Bilateral ☐ Unilateral |
| 47. Danish kara a saria a ala 0 | T V T N - N Obin to Occasion #40 |
| 17. Do you have a varicocele? | ☐ Yes ☐ No → Skip to Question #18 |
| 17a. Indicate type: | ☐ Unilateral |
| | Bilateral |
| ENVIRONMENTAL EXPOSURES | |
| 18. Have you ever used cigarettes? | Never → Skip to Question #19 |
| | ☐ Current |
| | Former |
| | <del>_</del> |
| →Current or former users, proceed to que | estions 18a through 18g. ← |
| 18a. Are you currently smoking? | ☐ Yes ☐ No |
| 18b. On average, how many cigarettes do/did you sr | moke |
| per day? | ☐ 1-10 ☐ 21-40 |
| | □ 11-20 □ >40 |
| 18c. On days that you can/could smoke cigarettes | |
| freely, how soon after you wake up do you smo | ke |
| your first cigarette of the day? | ☐ minutes ☐ hours |
| 40.4.11 | □ .4 □ 0.40 |
| 18d. How many years have/had you smoked? | ☐ <1 year ☐ 6-10 years |
| | ☐ 1-5 years ☐ >15 years |

| 18e. How many of times have you tried to quit smok | ing |
|---|---|
| (ever)? | times |
| 18f. How long ago did you quit smoking? | |
| | ☐ 6-10 years ☐ NA- currently smoking |
| 18g. Do/did you use any other forms of tobacco? Question #19 | ☐ Yes ☐ No → Skip to |
| 18g1. If yes, please indicate other tobacco produ | ucts: ☐ Cigars ☐ Pipes |
| | ☐ Snus/snuff/dip ☐ Chew |
| | ☐ Electric Cigarettes |
| | Dissolvables |
| | ☐ Hookah/water pipe |
| | Other (specify): |
| 19. On a scale of 1 thru 7, are you around smokers muc | th of the time? |
| To. Off a socie of Talla T, allo you around officiol flac | 1- Not at all true of me |
| | □ 2 |
| | □ 3 |
| | ☐ 4 |
| | □ 5 |
| | □ 6 |
| | ☐ 7- Extremely true of me |
| 20. How many people who live in your household use | |
| tobacco? (Do not count yourself) | people |
| 21. Does your spouse or partner currently use | tobacco? ☐ Yes ☐ No |
|---|---|
| 22. Have you used any recreational drugs or no months? | on-prescribed prescription medicines in the last 3<br>☐ Yes ☐ No → Skip to Question #23 |
| 22a. If yes, indicate what type: | ☐ Marijuana |
| | ☐ Cocaine |
| | ☐ Methadone / Narcotics |
| | Other (specify): |
| 23. During the last 12 months, how often did you alcohol? Choose only one. (By a drink we meat can or glass of beer or cooler, a 5 ounce glass of with the cooler of the c | an half an ounce of absolute alcohol (e.g. a 12 ounce |
| | ☐ Everyday |
| | ☐ 5 to 6 times a week |
| | 3 to 4 times a week |
| | ☐ twice a week |
| | once a week |
| | ☐ 2 to 3 times a month☐ once a month |
| | ☐ 3 to 11 times in the past year |
| | 1 or 2 times in the past year |
| →If any of the responses are check | red above, proceed to Question #24. ← |
| ☐ I did not drink any alcohol in the past year, b | out I did drink in the past |
| → Skip to Question #23a. | |
| ☐ I never drank any alcohol in my life | |
| → Skip to Question #23b. | |

| 23a. During your <u>lifetime</u> , what is the maximum number of drinks containing alcohol that you drank within a 24-hour period? | |
|---|---|
| | ☐ 36 drinks or more |
| | 24 to 35 drinks |
| | ☐ 18 to 23 drinks |
| | 12 to 17 drinks |
| | ☐ 8 to 11 drinks |
| | ☐ 5 to 7 drinks |
| | 4 drinks |
| | 3 drinks |
| | 2 drinks |
| | 1 drink |
| →STOP HERE, and proced | ed to Question #26. ← |
| 23b. So you have never had a drink containing | alcohol in your entire life? |
| ☐ Yes, I never drank →Skip to Question #26 | |
| No, I did drink. → Return to Question #23 | |
| 24. During the last 12 months, how <u>many</u> alcoholic you drank alcohol? Choose only one. | drinks did you have on a typical day when |
| | 25 or more drinks |
| | ☐ 19 to 24 drinks |
| | ☐ 16 to 18 drinks |
| | ☐ 12 to 15 drinks |
| | ☐ 9 to 11 drinks |
| | ☐ 7 to 8 drinks |

| | 5 to 6 drinks |
|---|---|
| | 3 to 4 drinks |
| | 2 drinks |
| | 1 drink |
| 25. During the last 12 months, how often did you halcohol within a two-hour period? Choose only ounce cans or bottles of beer, 4 five ounce glasses of waspirits.) | one. (That would be equivalent of a least 4 12- |
| | ☐ Everyday |
| | ☐ 5 to 6 days a week |
| | ☐ 3 to 4 days a week |
| | 2 days a week |
| | ☐ one day a week |
| | 2 to 3 days a month |
| | one day a month |
| | ☐ 3 to 11 days in the past year |
| | ☐ 1 or 2 days in the past year |
| | ☐ 0 days in the past year |
| 26. Are you exposed to pesticides on a regular bas | sis? |
| 27. Have you been exposed to toxic chemicals? 27a. If yes, what types: | ☐ Yes ☐ No → Skip to Question #28 |
| 28. Are you exposed to radiation (x-rays) regularly | ? ☐ Yes□ No |

| 29. Are you exposed to prolonged heat regularly? | |
|---|---|
| (e.g. hot tubs, saunas)? | ☐ Yes ☐ No |
| 30. Have you ever taken testosterone or anabolic steroic | ds? ☐ Yes ☐ No → Skip to Question #31 |
| 30a. Are you currently using steroids? | ☐ Yes ☐ No → Skip to Question #31 |
| 30b. Please list: | |
| PATERNITY/FERTILITY HISTORY | |
| 31. Have you ever created a pregnancy with anyone? | ☐ Yes ☐ No |
| 32. Have you ever had any infertility treatment and/or su | rgery in the past?<br>☐ Yes ☐ No <i>→ Skip to Question #33</i> |
| 32a.What type of treatment/surgery did you have | ? |
| (check all that apply) | <ul><li>☐ Varicocele Repair</li><li>☐ Vasectomy Reversal</li><li>☐ In Vitro Fertilization</li></ul> |
| | ☐ In Vitro Fertilization with |
| | Intracytoplasmic<br>Sperm Injection (IVF<br>with ICSI) |
| | ☐ Viagra/Cialis/Levitra |
| | ☐ Intrauterine Insemination (IUI) |
| | ☐ Intrauterine Insemination with ICSI (IUI with ICSI) |
| | ☐ Inguinal hernia repair |
| | ☐ Prostate Surgery |
| | Other |
| | (specify): |

| 33. During the time you have been trying examination? | - | d a male genital o → Skip to Question #34 |
|---|---|---|
| 33a. If yes, were you told that yo | ou have dilated scrotal veins? (e<br>☐ Yes☐ N | |
| 34. How long have you and your partner ———— | | ☐ Unknown |
| 35. Have you achieved pregnancy with y | your current partner? 🗌 Yes 🗌 | No → Skip to Question #36 |
| 35a. If yes, complete the table below | V: | |
| Pregnancy | Date | |
| <u> </u> | // | |
| <u> </u> | // | |
| #3 | // | |
| <u> </u> | // | |
| #5 | // | |
| 36. Currently, what is your average frequency | <u> </u> | artner?<br>1 per month |
| | □ 1- | -2 times per month |
| | □1 | time per week |
| | _ 2- | -3 times per week |
| | □ D | aily |

| 37. Do you know how to time intercourse to your partner's | menstrual cycle? |
|---|---|
| 38. Do you use any lubrication during intercourse? | ☐ Yes ☐ No |
| MEDICATION INFORMATION | |
| 39. Are you currently taking any medications? | ☐ Yes ☐ No |
| (include prescription medications and over the counter med | ications, do not include supplements here) |
| →If Yes, please list all medications on the Co | oncomitant Medications CRF← |
| 40. Are you taking any vitamins, multivitamins, or herbal s | upplements?<br>☐ Yes ☐ No |
| →If Yes, please speak with the stud | y staff immediately ← |
| 41. Have you taken any vitamins, multivitamins, or herbal months? | supplements over the past six<br>☐ Yes ☐ No |
| DEMOGRAPHICS | |
| 42. What is your age? | years old |
| 43. What is your marital status? (check only one) | Single |
| | Married |
| | Divorced |
| | Separated |
| | Widowed |

| 44. What is your highest level of education? | ☐ 8 <sup>th</sup> grade or less |
|---|---|
| | ☐ Some high school |
| | ☐ High school graduate |
| | ☐ Some college |
| | ☐ College graduate |
| | ☐ Graduate degree |
| 45. What is your occupation? (check only one) | ☐ Management, Business & Financial Occupations |
| | ☐ Computer, Engineering & Science Occupations |
| | ☐ Education, Legal, Community Service, Arts, & Media Occupations |
| | ☐ Healthcare Practitioners and Technical Occupations |
| | ☐ Service Occupations |
| | ☐ Sales and Related Occupations |
| | ☐ Office & Administrative Support Occupations |
| | ☐ Farming, Fishing, & Forestry Occupations |
| | ☐ Construction & Extraction Occupations |
| | ☐ Installation, Maintenance, & Repair Occupations |
| | ☐ Production Occupations |
| | ☐ Transportation & Material Moving Occupations |
| | ☐ Military Specific Occupations |
| | ☐ Student |

| | Retired |
|---|---|
| | Unemployed |
| | Disabled |
| 46. What is your annual Household Income? | |
| (check only one) | |
| | ☐ \$25,000 to \$49,999 |
| | ☐ \$50,000 to \$74,999 |
| | ☐ \$75,000 to \$100,000 |
| | ☐ Wish to not answer |
| 47. What type(s) of Insurance coverage do you have? (che | eck all that apply) |
| | ☐ Managed Care Plan or HMO |
| | Other Private Insurance |
| | ☐ Medicaid |
| | ☐ Medicare |
| | ☐ Self-pay/Uninsured |
| 48. Are you currently participating in any other clinical trial | |
| | ∐ Yes ∐ No |
| SIGNATURE | |
| ☐ Patient completed form ☐ Study coordinator perform | ned an interview of this questionnaire |
| _ , _ , | · |
| I have reviewed the data captured on this form and to the I Signature: | Date:// |
| Oignature. | Month Day Year |

## 13 Appendix B: Female Medical History Questionnaire



### Males, Antioxidants, and Infertility (MOXI) Trial

| W | J | | HIST | OB | V |
|---|----|------|------|----|---|
| ľ | עם | ICAL | ПΟІ | UR | • |

Do you have a history of any of the following medical conditions or problems?

| Body System | Response<br>(If NO, skip to<br>next question) | Condition/Problem | Currently<br>Symptomatic | Requires<br>Medication |
|---|---|---|---|---|
| 1. Problems with your head, ears, | Yes | ☐ Hearing loss | Yes | ☐ Yes |
| eyes, nose or | □ No | Blindness | | |
| throat? | | Sinus | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 2. Problems with | Yes | Stroke | Yes | ☐ Yes |
| your brain, nervous system or any | □No | Migraines | | |
| psychiatric conditions? | | Seizures | | |
| conditione. | | ☐ CVA/TIA | | |
| | | Depression | | |
| | | ☐ Anxiety | | |
| | | ☐ Bipolar disorder | | |
| | | Schizophrenia/Psychosis | | |

| | | ☐ Obsessive-Compulsive Disorder | | |
|---|---|---|---|---|
| | | ☐ ADD/ADHD | | |
| | | ☐ Eating Disorder (anorexia, bulimia) | | |
| | | ☐ Post-Traumatic Stress | | |
| | | ☐ Acute Stress Disorder | | |
| | | ☐ Substance/Alcohol Abuse | | |
| | | ☐ PMS/PMDD | | |
| | | ☐ Phobia/Agoraphobia | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 3. Problems with | Yes | Asthma | Yes | Yes |
| 3. Problems with your respiratory system? | ☐ Yes | | ☐ Yes | ☐ Yes |
| your respiratory | _ | Asthma | _ | ☐ Yes |
| your respiratory | _ | ☐ Asthma ☐ Pneumonia | _ | ☐ Yes ☐ ☐ |
| your respiratory | _ | ☐ Asthma ☐ Pneumonia ☐ COPD | | ☐ Yes ☐ ☐ ☐ ☐ ☐ ☐ ☐ |
| your respiratory | _ | ☐ Asthma ☐ Pneumonia ☐ COPD ☐ Emphysema | | ☐ Yes ☐ |
| your respiratory | _ | ☐ Asthma ☐ Pneumonia ☐ COPD ☐ Emphysema ☐ TB | | Yes Yes |
| your respiratory | _ | □ Asthma □ Pneumonia □ COPD □ Emphysema □ TB □ Surgery (specify): | | |

| 4. Problems with | ☐ Yes | ☐ Previous heart attack | ☐ Yes | ☐ Yes |
|---|---|---|---|---|
| your heart or cardiovascular | ☐ No | ☐ Congenital heart defect | | |
| system? | | ☐ Palpitations | | |
| | | ☐ Arrhythmias | | |
| | | ☐ Valve disease | | |
| | | ☐ Angina | | |
| | | ☐ CHF | | |
| | | Hypertension | | |
| | | Syncope | | |
| | | ☐ Blood clot in leg, lung, brain | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 5. Problems with | Yes | Arthritis | Yes | Yes |
| your muscles, joints, bones or | ☐ No | Lupus | | |
| musculoskeletal system? | | Osteoporosis | | |
| | | ☐ Gout | | |
| | | ☐ Disc disease | | |
| | | Surgery (specify): | | |
| | | Other (specify): | | |
| 6. Problems with | Yes | ☐ Irritable bowel | Yes | Yes |
| your gastrointestinal system? | □No | ☐ GI cancer | | |
| | | Liver disease | | |
| | | ☐ Peptic ulcer | | |
| | | GERD | | |
| | | ☐ Hepatitis | | |
| | | ☐ Pancreatitis | | |

| | | | Surgery (specify): | | | |
|---|---|---|---|---|---|---|
| | | | Other (specify): | | | |
| 7. Problems with | Yes | | ☐ Clotting | | Yes | Yes |
| your blood and metabolic system? | | | ☐ Anemia | | | |
| | ☐ No | | ☐ Hyperlipidemia | | | |
| | | | ☐ Diabetes | | | |
| | | | ☐ Hyper/hypothyroidism | | | |
| | | | Surgery (specify): | | | |
| | | | Other (specify): | | | |
| | | | I | | | |
| 8. Problems with | ] Yes | _ | ncer | Yes | Yes | |
| the whole body? | ] No | (specif | fy): | | | |
| | • | ☐ Alc | coholism | | | |
| | | ☐ Dru | ug abuse | | | |
| | | ☐ Alle | ergies | | | |
| | | ☐ Fat | tigue | | | |
| | | □ We | eakness | | | |
| | | ☐ Adı | renal or Ovarian androgen | | | |
| | | sec | creting tumor | | | |
| | | ☐ Cu | shing's Syndrome | | | |
| | | Sur | rgery<br>'y): | | | |
| | | ☐ Oth | | | | |
| | | | | • | 1 | |

→If any of these conditions require medication treatment, record medications on the concomitant medication log ←

# **ENVIRONMENTAL EXPOSURES**

| 9. Have you ever used cigarettes? | ☐ Never → Skip to Question #10 | |
|---|---|---|
| | ☐ Current | |
| | Former | |
| →Current or former users, proceed to que | estions 9a thro | ough 9g← |
| 9a. Are you currently smoking? | ☐ Yes ☐ No | |
| 9b. On average, how many cigarettes do/did you smok | ke per day?<br>☐ 1-10 | <u>21-40</u> |
| | <u> </u> | |
| 9c. On days that you can/could smoke cigarettes freely smoke your first cigarette of the day? | y, how soon aft<br>☐ minutes | er you wake do you<br>☐ hours |
| 9d. How many years have/had you smoked? | ☐ <1 year | ☐ 6-10 years |
| | ☐ 1-5 years | ☐ >15 years |
| 9e. How many times have you tried to quit smoking (e | ver)? | times |
| 9f. How long ago did you quit smoking? | ☐ <1 year | ☐ 11-15 years |
| | ☐ 1-5 years | ☐ >15 years |
| | ☐ 6-10 years | 3 |
| | ☐ NA- currer | ntly smoking |

| 9g. Do/did you use any other forms of tobacco? | ☐ Yes ☐ No → Skip to Question #10 |
|---|---|
| 9g1. If yes, please indicate other tobacco products | : Cigars |
| | ☐ Pipes |
| | ☐ Snus/snuff/dip |
| | ☐ Electric Cigarettes |
| | Dissolvables |
| | ☐ Hookah/water pipe |
| | Other |
| | (specify): |
| 10. On a scale of 1 thru 7, are you around smokers much | |
| | ☐ 1- Not at all true of me |
| | <u> </u> |
| | □ 3 |
| | ☐ 4 |
| | □ 5 |
| | □ 6 |
| | ☐ 7- Extremely true of me |
| 11. How many people who live in your household use toba | acco? (Do not count yourself) people |
| <del>_</del> | , . |
| 12. Does your spouse or partner currently use tobacco? | ☐ Yes ☐ No |
| 13. Have you used any recreational drugs or non-prescribe months? | ed prescription medicines in the last 3 ☐ Yes ☐ No → Skip to Question #14 |
| 13a. If yes, indicate what type(s): (check all that apply) | ☐ Marijuana |

| | ☐ Cocaine |
|---|---|
| | ☐ Methadone/Narcotics |
| | Other (specify): |
| 14. During the last 12 months, how <u>often</u> did you us<br>alcohol? Choose only one. (By a drink we mean ha<br>ounce can or glass of beer or cooler, a 5 ounce glass of | alf an ounce of absolute alcohol (e.g. a 12 |
| | ☐ Everyday |
| | ☐ 5 to 6 times a week |
| | ☐ 3 to 4 times a week |
| | ☐ twice a week |
| | once a week |
| | ☐ 2 to 3 times a month☐ once a month |
| | ☐ 3 to 11 times in the past year |
| | ☐ 1 or 2 times in the past year |
| →If any of the responses are checked a | above, proceed to Question #15. |
| I did not drink any alcohol in the past year, but I did | drink in the past 🗌 |
| → Skip to Question #14a. | |
| I never drank any alcohol in my life | |
| → Skip to Question #14b. | |
| 14a. During your <u>li<b>fetime</b>,</u> what is the maximum nu<br>drank within a <u>24-hour period</u> ? | mber of drinks containing alcohol that you |
| | ☐ 36 drinks or more |
| | ☐ 24 to 35 drinks |
| | ☐ 18 to 23 drinks |

| | 12 to 17 drinks |
|---|---|
| | ☐ 8 to 11 drinks |
| | 5 to 7 drinks |
| | 4 drinks |
| | 3 drinks |
| | 2 drinks |
| | 1 drink |
| →STOP HERE, and proceed to Menstrual History | ory Section.← |
| 14b. So you have never had a drink containing alcohol in y ☐ Yes, I neve | your entire life?<br>er drank <i>→Skip to next section</i> |
| ☐ No, I did d | rink. → Return to Question #14 |
| 15. During the last 12 months, how <u>many</u> alcoholic drinks did you you drank alcohol? Choose only one. | have on a typical day when |
| | 25 or more drinks |
| | ☐ 19 to 24 drinks |
| | ☐ 16 to 18 drinks |
| | 12 to 15 drinks |
| | 9 to 11 drinks |
| | ☐ 7 to 8 drinks |
| | ☐ 5 to 6 drinks |
| | O to A defector |
| | 3 to 4 drinks |
| | 2 drinks |

16. During the last 12 months, how <u>often did you have 4 or more drinks</u> containing any kind of alcohol within a two-hour period? Choose only one. (That would be equivalent of a least 4 12-

| ounce cans or bottles of beer, 4 five ounce glasses of wine, 4 drinks each containing one shot of liquor or spirits.) | |
|---|---|
| | ☐ Everyday |
| | ☐ 5 to 6 days a week |
| | ☐ 3 to 4 days a week |
| | ☐ two days a week |
| | ☐ one day a week |
| | ☐ 2 to 3 days a month |
| | ☐ one day a month |
| | ☐ 3 to 11 days in the past year |
| | ☐ 1 or 2 days in the past year |
| | ☐ 0 days in the past year |
| MENSTRUAL HISTORY | |
| 17. On average, how many periods do you have per year? | periods OR Unknown |
| 18. What is the average number of days between your period? | days OR 🗌 Unknown |
| 19. What is the number of days of bleeding per cycle? | days OR 🗌 Unknown |
| 20. Date of last menstrual period:/ | / OR |
| Month | Day Year |
| GYNECOLOGICAL HISTORY | |
| 21. Have you ever used medication to regulate your period? Question #22 | ☐ Yes ☐ No → Skip to |
| If yes, check below types of medications previously used: (che | eck all that apply) |

| | used | Medication | | Duration (months) |
|---|---|---|---|---|
| | | 21a.Birth control pills | | Unknown |
| | | 21b. Progesterone (e.g. Provera) | | Unknown |
| | | 21c. Letrozole | | Unknown |
| | | 21d. Anastrozole | | Unknown |
| | | 21e. Cabergoline (Dostinex) | | Unknown |
| | | 21f. GnRH agonist (e.g. any form- Lupron, Synnarel) | | Unknown |
| | | 21g. Metformin (Glucophage) | | Unknown |
| | | 21h. Rosiglitazone (Avandia) | | Unknown |
| | | 21i. Other (specify): | | Unknown |
| - | | 21j. Other (specify): | | Unknown |
| | | 21k. Other (specify): | _ | Unknown |
| | | 21I. Other (specify): | _ | Unknown |
| Questi | on #23 | d a pap smear? | □ Y | es No → Skip to |
| 22 | a. Date of last p | pap smear: | | |
| 22 | b. Was the resu | ılt of this pap smear abnormal? | ΠY | ′es |
| 23. Ha | ave you ever be | en diagnosed with a sexually transmitted dis | | infection?<br>es |
| Questi | on #24 | | | |
| 23 | a. Type of STD | /STI: (check all that apply) | □G | Gonorrhea |
| | | | □С | chlamydia |
| | | | □s | yphillis |

| | 27c. Sonohysterogram (SHG) | / |
|---|---|---|
| | 27b. Hysterosalpingogram (HSG) | / |
| | 27a. Ultrasound (transvaginal or abdominal) | /Unknown |
| ever had | Type of Procedure or Surgery | (MM/YYYY) |
| Check if | production types of production of ourgonous do | Date |
| | neck below types of procedures or surgeries do | ☐ Yes ☐ No → Skip to Question #28 |
| 27. Have you | u ever had any gynecological procedures or su | rgeries done with the past? |
| 26a. Did you receive treatment? | | ☐ Yes ☐ No |
| 26. Have yoւ | u ever been diagnosed with Endometriosis? | ☐ Yes ☐ No → Skip to Question #27 |
| 25a. Did | you receive treatment? | ☐ Yes ☐ No |
| 25. Have you | u ever been diagnosed with Fibroids? | ☐ Yes ☐ No → Skip to Question #26 |
| 24a. Did | you receive treatment? | ☐ Yes ☐ No |
| · | , | ☐ Yes ☐ No → Skip to Question #25 |
| 24. Have you | u been diagnosed with Pelvic Inflammatory dise | ease? |
| 23b. Did | you receive treatment? | ☐ Yes ☐ No |
| | | Other (specify): |
| | | ☐ Trichomoniasis (Trich) |
| | | ☐ Human Papillomavirus<br>(HPV) |
| | | ☐ Herpes Simplex Virus (HSV) |

| 27d. Hysteroscopy | / | Unknown |
|------------------------------------------------|---|---------|
| 27e. Colposcopy | / | Unknown |
| 27f. Salpingo-oophorectomy | / | Unknown |
| 27g. Tubal ligation | / | Unknown |
| 27h. Endometrial ablation | / | Unknown |
| 27i. Polypectomy | / | Unknown |
| 27j. Oophorectomy | / | Unknown |
| 27k. Uterine dilation & curettage | / | Unknown |
| 27l. Salpingectomy | / | Unknown |
| 27m. Ovarian surgery | / | Unknown |
| 27n. Hysterectomy with or without oophorectomy | / | Unknown |
| 27o. Unilateral or bilateral oophorectomy | / | Unknown |
| 27p. Ovarian cyst removal | / | Unknown |
| 27q. Endometriosis | / | Unknown |
| 27r. Lysis of adhesions | / | Unknown |
| 27s. Myomectomy | / | Unknown |
| 27t. UAE (uterine artery embolization) | / | Unknown |
| 27u. Diagnostic laparoscopy | | Unknown |
| 27v. IUD removal | | Unknown |
| 27w. Caesarean section | / | Unknown |
| 27x. LEEP | / | Unknown |
| 27y. Other (specify): | / | Unknown |
| 27z. Other (specify): | / | Unknown |

| INFERTI | LITY HISTORY | | | |
|---|---|---|---|---|
| 28. How I | ong have you been trying to get pregnant? | | months | OR Unknown |
| 29. Have you ever received a diagnosis from a physician for why pregnant? | | | · | uble getting<br>sip to Question #30 |
| 29a. \ | What was your diagnosis? (Check all that apply) | | vulatory dysfu | nction (e.g. PCOS) |
| | | □ Τι | ıbal factor (e.ç | g. blocked tubes) |
| | | ☐ Er | ndometriosis | |
| | | ☐ Ut | erine factor (e | e.g. fibroids) |
| | | ☐ Ma | ale factor infe | rtility |
| | | ☐ Ur | nexplained | |
| | | ☐ In | tra-abdominal | adhesions |
| | | ☐ Ce | ervical factor | |
| 30. Have you ever received therapy for infertility? ☐ Yes ☐ No → Skip to Question #31 | | | kip to Question #31 | |
| If yes | , check below types of therapies previously used | : (check | all that apply) | |
| Check if ever | | | Number of times received | |
| used | Name of Therapy | | (enter<br>"99" if<br>unknown) | Date<br>(MM/YYYY) |
| | 30a. Clomiphene Citrate (Clomid) | | | / Unknow |
| | 30b. Clomid and Intrauterine Insemination (IUI) | | | / Unknow |
| | 30c. Letrozole (Femara) | | | / Unknow |
| | 30d. Letrozole and Intrauterine Insemination (II | JI) | | / Unknow |
| | 30e. Intrauterine Insemination with no medicati | on . | | / Unknow |

| | | 30f. Clomid/gonadatropins/IUI | | / | Unknov |
|---|---|---|---|---|---|
| | | 30g. Gonadatropins (infertility shots) | | | Unknov |
| | | . , , , | —— | / | |
| | | 30h. Gonadatropins with IUI | | / | _ |
| | | 30i. Lupron/gonadotropins/IUI | | / | _ Unknov |
| | | 30j. In Vitro Fertilization (IVF) | | | _ Unknov |
| | | 30k. IVF with Intracytoplasmic Sperm Injection (ICSI) | | / | Unknov |
| | | 30l. Frozen Transfer | | / | _ Unknov |
| | | 30m. Donor sperm | | / | _ Unknov |
| | | 30n. Donor egg | | / | _ Unknov |
| | | 30o. Donor embryo | | / | _ Unknov |
| | | 30p. Other (specify): | | / | _ Unknov |
| | | 30q. Other (specify): | | / | _ Unknov |
| CC | ONCO | MITANT MEDICATIONS | | | |
| 21 | ۸re v | ou allergic to any medications? | sc□No→S | kip to Question #32 | |
| 51. | | | .5 <u> NO 7</u> 31 | NP to Question #32 | |
| | Pleas | e list these medications: | | | |
| 32. | Are y | ou currently taking any medications on a daily basis? | ☐ Yes ☐ I | No | |
| | • | | | | |
| 33 | Are v | ou currently taking any vitamins or supplements on a da | ilv basis? | | |
| -0. | <b>.</b> y | - a carpionionio di dappionionio di di di | ☐ Yes ☐ I | No. | |
| | | | resI | NU | |

→If YES to Question #32 & #33, complete Concomitant Medication CRF ←

# **SIGNATURE**

| ☐ Patient completed form | |
|---|---|
| ☐ Study coordinator performed an interview of this ques | tionnaire |
| To the best of your knowledge the above information | is correct. |
| Signature of Patient: | Date:/// |
| | Month Day Year |
| The above information has been verified with the pati | ient and is complete. |
| Signature: | Date: / / |
| | Month Day Year |

## 14 Appendix C: List of Prohibited Concomitant Medications

#### **Female**

```
Progestins (Oral or Cyclic)
       medroxyprogesterone acetate (Provera, Cycrin, Amen, Curretab)
       megestrol (Megase) norethindrone (Aygestin)
       progesterone gel (Crinone)
       Micronized progesterone (Prometrium)
GnRH Agonists/Antagonists Leuprolide (Lupron)
nafarelin (Synarel)
buserelin gosarelin (Zoladex)
ganarelix (Antagon) cetrorelix
(Cetrotide) Gonadotropins
Pergonal
Repronex
Follistim
Gonal-F
Fertinex
Metrodin
Injectable Contraceptives
       medroxyprogesterone acetate (Depo Provera)
Oral Contraceptives Any Brand
Continuous Progestins (Not including cyclic)
       Any Brand
Contraceptive Implants
       Norplant (levonorgestrel implants)
       Implanon
Clomiphene
Letrozole (femara)
Tamoxifen
```

#### Male

```
Inflammatory bowel disease medications - Need 3 month washout
Sulfasalazine
       Azulfidine
       Azulfidine EN
       Azathioprine
Infliximab
Antihypertensives - Need 3 month washout
Calcium channel blockers
       Nifedipine
       Adalat
       Afeditab
       Nifediac
       Nifedical
       Procardia
Spironolactone
5 alpha reductase medications
       Finasteride (Propecia, Proscar)
       Alfatradiol (Ell-Cranell Alpha, Pantostin)
       Dutasteride (Avodart)
       Flutamide
Cimetidine (Tagamet) - Need 3 month washout
Immunosuppressive agents within the past 1 year
Chemotherapeutic agents within the past 1 year
Androgens - Need 6 month washout
       DHEA or DHEAS, androstenedione
       OTC "testosterone boosting" herbals and supplements
       OTC workout enhancing supplements
Synthetic testosterone or anabolic steroids - Need 6 month washout
       Testred
Android
Axiron
```

```
Androgel 1%
Androgel 1.62%
Tesetim
      Fortesta
      Vogelxo
      Striant
      Androderm
      Natesto
      Aveed
      Testosterone cypionate
      Testosterone enanthate
      Testopel
Testosterone modulating medications - Need 3 month washout
      Clomid
      Anastrazole
      HCG
             Profasi
             Ovidrel
      Lupron
      Zoladex
```

Cannabis (Marijuana) - Need 3-month washout

# 15 Appendix D: Review of Antioxidant Formulations

# 15.1 Commercially Available Formulations

| | | I . | I | T | I . | T | I | | | - | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Coast | Countboost 2 | ProCreation 2 | | Fertilsan 3 | MotilityBoost 2 | Proceptin 4 | Proxeed 1 | Popmen 3 | | Blend 2 |
| Ingredient | 4 Caps | Caps | Caps | Caps | Caps | Caps | Caps | packet | Caps | XR 4 caps | caps |
| Acetyl-L-Carnitine | | | | | | | x | 500 mg | | | |
| Calcium (as amino acid chelate) | | | 50 mg | | | | | | | | |
| Chromium (as polynicotinate) | | | .12 mg | .12 mg | | | | | .12 mg | | |
| Coenzyme Q10 (Ubiqonone) | | x | | Х | 15 mg | х | x | 20 mg | | | |
| Copper (as gluconate) | | | 2 mg | | | | | | 2 mg | | |
| Folate (as folic acid) | 1 mg | | 400 mcg | 500 mcg | .8 mg | | 533 mg | .2 mg | .5 mg | 1mg | 0.4mg |
| Glutathione | | | | | | | | | | | |
| lodine | | | | 150 mcg | | | | | .15 mg | | |
| Iron (as amino acid chelate) | | | 5 mg | | | | | | | | |
| L-Arginine (free from amino acid) | | | 100 mg | | 500 mg | х | x | | | | |
| L-Carnitine (as L-carnitine-L-tartrate) | | | 50 mg | х | 500 mg | х | x | 1000 mg | | 1000mg | |
| L-Glutathione | | х | | | | | x | | | | |
| L-Methionine | 25 mg | | | | | | x | | | | |
| L-taurine | | | 50 mg | | | | | | | | |
| Lycopene | 100 mg | | | | | | x | | | 10mg | |
| Manganese (as amino acid chelate) | | | 5 mg | 120 mg | | | | | 2 mg | | |
| N-acetyl-I-cystine | | | | | 80 mg | х | | | | | |
| Niacin (as Inositol Hexanicotinate) | | 25 mg | 20 mg | 20 mg | | | | | 20 mg | | |
| Pantothenic Acid (as calcium pantothenate) | | | 10 mg | 10 mg | | | | | 10 mg | | |
| Relora® (U.S. Patent 6,582,735) | 250 mg | | | | | | | | | | |
| Selenium (as L-selenomethionine) | 0.25 mg | | .1 mg | 0.1mg | .06 mg | | .133 mg | .05 mg | .1 mg | 0.2mg | 0.07mg |
| Thiamin (as thiamine HCI) (vitamin B1) | | | 20 mg | 1.5 mg | | | | | 1.5 mg | | |
| Turmeric (curcuma longa rhizome) | | | 50 mg | | | | | | | | |
| Vitamin A (as beta carotene) | 5000 IU | | 5000 IU | 5000IU | | | 200 IU | | 5000 IU | | |
| Vitamin B12 (as cyanocobalamin) | 0.015 mg | 0.5 mg | .02 mg | .025 mg | | .5 mg | 1 mg | 1.5 mcg | 25 mcg | | 0.006mg |
| Vitamin B2 (as Riboflavin) | | 15 mg | 20 mg | 1.7 mg | | | | | 1.7 mg | | |
| Vitamin B6 (as pyridoxine HCI) | | | 20 mg | | 25 mg | | 1.3 mg | | 2 mg | | 2mg |
| Vitamin C (as ascorbic acid) | 200 mg | 500 mg | 60 mg | | 200 mg | | | 90 mg | 250 mg | 500mg | 120mg |
| Vitamin D3 (cholcalciferol) | | | 400 IU | 400 IU | .01 mg | | 267 IU | | 400 IU | 2000IU | |
| Vitamin E (as d-alpha tocopheryl acid succinate) | 400IU | | 150 IU | 150 IU | 120 mg | | 267 IU | | 150 IU | 400IU | 150IU |
| Vitamin K2 (as menatetrenone) | | | .1 mg | .08 mg | | | | | .08 mg | | |
| , | 70 mg | | 25 mg | 30 mg | 40 mg | | 27mg | 10 mg | 30 mg | 20mg | 15mg |

## 15.2 Research Formulations

| | Akiyama | Balercia | Balercia | Biagotti | Cavallini | Ciftci | Conquer | Dawson | Galatioto | Greco | Keskes-Ammar |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Ingredient | 1999 | 2005 | 2009 | 2003 | 2004 | 2009 | 2000 | 1990 | 2008 | 2005 | 2003 |
| Acetyl-L-Carnitine | | 3g (1) | | 1g | 1g | | | | | | |
| Calcium (as amino acid chelate) | | | | | | | | | х | | |
| Chromium (as polynicotinate) | | | | | | | | | | | |
| Coenzyme Q10 (Ubiqonone) | | | 200 mg | | | | | | | | |
| Copper (as gluconate) | | | | | | | | | | | |
| Folate (as folic acid) | | | | | | | | | | | |
| Glutathione | | | | | | | | | | | |
| lodine | | | | | | | | | | | |
| Iron (as amino acid chelate) | | | | | | | | | | | |
| L-Arginine (free from amino acid) | | | | | | | | | | | |
| L-Carnitine (as L-carnitine-L-tartrate) | | 3g (2) | | 2g | 2g | | | | | | |
| L-Glutathione | | | | | | | | | | | |
| L-Methionine | | | | | | | | | | | |
| L-taurine | | | | | | | | | | | |
| Lycopene | | | | | | | | | | | |
| Manganese (as amino acid chelate) | | | | | | | | | | | |
| N-acetyl-l-cystine | | | | | | 600mg | | | 600mg | | |
| Niacin (as Inositol Hexanicotinate) | | | | | | | | | | | |
| Pantothenic Acid (as calcium pantothenate) | | | | | | | | | | | |
| Relora® (U.S. Patent 6,582,735) | | | | | | | | | | | |
| Selenium (as L-selenomethionine) | | | | | | | | | | | 0.225mg |
| Thiamin (as thiamine HCI) (vitamin B1) | | | | | | | | | х | | х |
| Turmeric (curcuma longa rhizome) | | | | | | | | | | | |
| Vitamin A (as beta carotene) | | | | | | | | | х | | |
| Vitamin B12 (as cyanocobalamin) | | | | | | | | | | | х |
| Vitamin B2 (as Riboflavin) | | | | | | | | | | | |
| Vitamin B6 (as pyridoxine HCI) | | | | | | | | | | | х |
| Vitamin C (as ascorbic acid) | | | | | | | | 1000mg | х | 1000mg | |
| Vitamin D3 (cholcalciferol) | | | | | | | | | | | |
| Vitamin E (as d-alpha tocopheryl acid succinate) | 600mg | | | | | | | | х | 1000mg | 400mg |
| Vitamin K2 (as menatetrenone) | | | | | | | | | | | |
| Zinc (as zinc amino acid chelate) | | | | | | | | | | | |
| Zinc (as zinc sulfate) | | | | | | | | | | | |
| Cinnoxicam | | | | ? | 30mg q4day | | | | | | |
| Docosahexaenoic acid (DHA) | | | | | | | 800mg | | | | |

## 16 Appendix E: Risk Factors for Genetic Disorders

The following questions are designed to determine if you have an increased risk of having a baby with a genetic disorder. Sometimes genetic disorders occur even when there is no history of problems in your family. The following questions are related to you and your immediate family including mother, father, sister, brother, child, or grandparent. If you answer "yes" to any of the following questions and would like more information, please discuss this with your physician.

| Questions | Yes | No | Unknown | N/A |
|---|---|---|---|---|
| 1. If you conceive during this study, will you be 35 or older | | | | |
| when your baby is due? | | | | |
| 2 If you are of Meditorranean or Asian descent does | | | | |
| 2. If you are of Mediterranean or Asian descent, does | | | | |
| anyone in your family have thalassemia? | | | | |
| (a blood disorder that causes anemia) | | | | |
| 3. Is there a family history of neural tube defects? | | | | |
| 4. Have you had a child with a neural tube defect? | | | | |
| 5. Does anyone in your family have a history of congenital | | | | |
| heart defects? (heart problems when they were born) | | | | |
| 6. Does anyone in your family have Down Syndrome? | | | | |
| 7. Have you ever had a child with Down Syndrome? | | | | |
| 8. If you are of Eastern European Jewish or French Canadian | | | | |
| descent, does anyone in your family have a history of Tay- | | | | |
| Sachs disease? (a disorder of the central nervous system) | | | | |
| 9. If you are of Eastern European Jewish descent, does | | | | |
| anyone in your family have a history of Canavan disease? | | | | |
| (a disorder of the central nervous system that leads to blindness and muscle weakness) | | | | |
| 10. If you are of African American descent, is there any | | | | |
| history of sickle cell trait? (a type of anemia) | | | | |

| 11. If you are of African American descent, is there any |
|------------------------------------------------------------------------|
| history of sickle cell disease? (a type of anemia) |
| (4-), [ |
| 12. Do you or anyone in your family have a history of |
| hemophilia? (a disorder that causes bleeding) |
| 13. Do you or anyone in your family have a history of |
| muscular dystrophy? (a neuromuscular disorder) |
| 14. Do you or anyone in your family have a history of cystic |
| fibrosis? ( a disorder that causes thick mucous in the lungs and other |
| organs) |
| 15. Do you or anyone in your family have a history of |
| Huntington's disease? (a degenerative brain disease) |
| 16. Do you or anyone in your family have a history of alpha-1 |
| antitrypsin deficiency? (lack of a liver protein) |
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| 17. Do you or anyone in your family have a history of mental |
| retardation? |
| 17a. If yes to Question #17, was the person ever tested |
| for fragile-x syndrome? (a condition which can cause mild to severe |
| mental retardation) |
| mental retardation/ |
| 18. Do you or anyone in your family have a history of any |
| other genetic disease, chromosomal disorder or birth |
| defect? |
| 10. Do you have any matchalic discarders such as disk the same |
| 19. Do you have any metabolic disorders such as diabetes or |
| phenylketonuria (PKU)? |
| (a disorder which prevents the normal use of protein foods) |
| 20. Have you ever had 3 or more miscarriages in a row? |
| 21. Have you ever had a baby that was stillborn? |
| , |

# 17 Appendix F: Female Sexual Function Index (FSFI)

# Female Sexual Function Index (FSFI) ©

| Subject Iden | ntifier | Date |
|---|---|---|
| - | | |
| during the pa<br>clearly as po | ONS: These questions ask about your sexual<br>ast 4 weeks. Please answer the following que<br>ossible. Your responses will be kept completel<br>nese questions the following definitions apply: | stions as honestly and |
| Sexual activ | <u>ity</u> can include caressing, foreplay, masturbati | on and vaginal intercourse |
| Sexual inter | <u>course</u> is defined as penile penetration (entry) | of the vagina. |
| | ulation includes situations like foreplay with a pon), or sexual fantasy. | partner, self-stimulation |
| CHECK ON | LY ONE BOX PER QUESTION. | |
| experience, | re or <u>interest</u> is a feeling that includes wanting<br>feeling receptive to a partner's sexual initiatior<br>about having sex. | |
| 1. Over the | past 4 weeks, how often did you feel sexual o | tesire or interest? |
| | Almost always or always<br>Most times (more than half the time)<br>Sometimes (about half the time)<br>A few times (less than half the time)<br>Almost never or never | |
| 2. Over the or interes | past 4 weeks, how would you rate your <b>level</b><br>st? | (degree) of sexual desire |
| | Very high<br>High<br>Moderate<br>Low<br>Very low or none at all | |

Sexual arousal is a feeling that includes both physical and mental aspects of sexual excitement. It may include feelings of warmth or tingling in the genitals, lubrication (wetness), or muscle contractions.

| 3. | past 4 weeks, now <b>orten</b> did you feel sexually aroused ("turned on")<br>xual activity or intercourse? |
|---|---|
| | No sexual activity Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never |
| 4. | past 4 weeks, how would you rate your <b>level</b> of sexual arousal ("turn<br>ng sexual activity or intercourse? |
| | No sexual activity Very high High Moderate Low Very low or none at all |
| 5. | past 4 weeks, how <b>confident</b> were you about becoming sexually during sexual activity or intercourse? |
| | No sexual activity Very high confidence High confidence Moderate confidence Low confidence Very low or no confidence |
| 6. | past 4 weeks, how <b>often</b> have you been satisfied with your arousal ent) during sexual activity or intercourse? |
| | No sexual activity Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never |

| past 4 weeks, how <b>often</b> did you become lubricated ("wet") during ctivity or intercourse? |
|---|
| No sexual activity Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never |
| past 4 weeks, how <b>difficult</b> was it to become lubricated ("wet") during ctivity or intercourse? |
| No sexual activity Extremely difficult or impossible Very difficult Difficult Slightly difficult Not difficult |
| past 4 weeks, how often did you maintain your lubrication ("wetness") pletion of sexual activity or intercourse? |
| No sexual activity Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never |
| e past 4 weeks, how <b>difficult</b> was it to maintain your lubrication<br>ss") until completion of sexual activity or intercourse? |
| No sexual activity Extremely difficult or impossible Very difficult Difficult Slightly difficult Not difficult |

| past 4 weeks, when you had sexual stimulation or intercourse, how<br>I you reach orgasm (climax)? |
|---|
| No sexual activity Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never |
| past 4 weeks, when you had sexual stimulation or intercourse, how was it for you to reach orgasm (climax)? |
| No sexual activity Extremely difficult or impossible Very difficult Difficult Slightly difficult Not difficult |
| past 4 weeks, how satisfied were you with your ability to reach orgasm during sexual activity or intercourse? |
| No sexual activity Very satisfied Moderately satisfied About equally satisfied and dissatisfied Moderately dissatisfied Very dissatisfied |
| past 4 weeks, how satisfied have you been with the amount of a closeness during sexual activity between you and your partner? |
| No sexual activity Very satisfied Moderately satisfied About equally satisfied and dissatisfied Moderately dissatisfied Very dissatisfied |
| | past 4 weeks, how <b>satisfied</b> have you been with your sexual<br>nip with your partner? | | |
|---|---|---|--|
| | Very satisfied<br>Moderately satisfied<br>About equally satisfied and dissatisfied<br>Moderately dissatisfied<br>Very dissatisfied | | |
| 16. Over the | past 4 weeks, how <b>satisfied</b> have you been with your overal | sexual life? | |
| | Very satisfied<br>Moderately satisfied<br>About equally satisfied and dissatisfied<br>Moderately dissatisfied<br>Very dissatisfied | | |
| 17. Over the past 4 weeks, how <b>often</b> did you experience discomfort or pain <u>during</u> vaginal penetration? | | | |
| | Did not attempt intercourse Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never | | |
| | past 4 weeks, how <b>often</b> did you experience discomfort or pa<br>enetration? | ain <u>following</u> | |
| | Did not attempt intercourse Almost always or always Most times (more than half the time) Sometimes (about half the time) A few times (less than half the time) Almost never or never | | |
| | past 4 weeks, how would you rate your <b>level</b> (degree) of disc<br>ng or following vaginal penetration? | omfort or | |
| | Did not attempt intercourse<br>Very high<br>High<br>Moderate<br>Low<br>Very low or none at all | | |
| - | for completing this questionnaire | | |
| Copyright ©200 | Copyright © 2000 All Rights Reserved Page 5 (of 5) | | |

# Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey!

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:



2. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not limited at all |
|---|---|---|---|---|
| | Moderate activities, such as moving a table, pushing | | | |
| | a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 |
| , | Climbing several flights of stairs | 1 | 2 | 3 |

| 3. | During the <u>past 4 weeks</u> following problems with result of your physical l | ı your wor | | | | |
|---|---|---|---|---|---|---|
| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| a | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| ъ | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 🗆 4 | 5 |
| 4. | During the <u>past 4 weeks</u> following problems with <u>result of any emotional</u> | ı your wor | k or other | regular da | ily activitie | s <u>as a</u> |
| | | All of the time | Most of the time | Some of the time | A little of the time | None of<br>the time |
| a | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| ъ | Did work or other activities less carefully than usual | | 2 | 3 | 4 | 5 |
| | AV | | | | | |
| 5. | During the past 4 weeks<br>work (including both w | | | | | ormal |
| | Not at all A little | bit Mod | derately ( | Quite a bit | Extremely | |
| | 1 | 2 | 3 | 4 | 5 | |

| 6. | . These questions are about how | you f | eel and | how thi | ngs l | have be | en ' | with y | you |
|---|---|---|---|---|---|---|---|---|---|
| | during the past 4 weeks. For e | ach qu | iestion, | please | give 1 | the one | ans | swer 1 | that |
| | comes closest to the way you ha | ave be | en feeli | ng. Ho | v mu | ich of t | he t | ime | |
| | during the past 4 weeks | | | | | | | | |
| | | | | _ | _ | | _ | | _ |

| | | All of<br>the time | Most of<br>the time | Some of<br>the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | ' | | lacksquare | | | |
| 1 | Have you felt calm and peaceful? | 1 | 2 | 3 | | 5 |
| , | Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 |
| | Have you felt downhearted and depressed? | 1 | 2.,, | 3 | | ,, <u> </u> |

7. During the <u>past 4 weeks</u>, how much of the time has your <u>physical health or emotional problems</u> interfered with your social activities (like visiting with friends, relatives, etc.)?



Thank you for completing these questions!

# 19 Appendix H: Patient Health Questionnaire (PHQ-9)

#### PATIENT HEALTH QUESTIONNAIRE (PHQ-9)

| NAME: | ME: DATE: | | | |
|---|---|---|---|---|
| Over the last 2 weeks, how often have you been bothered by any of the following problems? | | | | |
| (use "✓" to indicate your answer) | Not at all | Several<br>days | More than half the days | Nearly<br>every day |
| 1. Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| 2. Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| 3. Trouble falling or staying asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. Feeling tired or having little energy | 0 | 1 | 2 | 3 |
| 5. Poor appetite or overeating | 0 | 1 | 2 | 3 |
| Feeling bad about yourself—or that you are a failure or have let yourself or your family down | 0 | 1 | 2 | 3 |
| 7. Trouble concentrating on things, such as reading the newspaper or watching television | 0 | 1 | 2 | 3 |
| 8. Moving or speaking so slowly that other people could have noticed. Or the opposite — being so figety or restless that you have been moving around a lot more than usual | 0 | 1 | 2 | 3 |
| 9. Thoughts that you would be better off dead, or of hurting yourself | 0 | 1 | 2 | 3 |
| | add columns | | + | + |
| (Healthcare professional: For interpretation of TOTA please refer to accompanying scoring card). | AL, TOTAL: | | | |
| If you checked off any problems, how difficult have these problems made it for you to do | | | cult at all | |
| your work, take care of things at home, or get along with other people? | | Very dif | | |

Copyright  $\ ^{\circ}$  1999 Pfizer Inc. All rights reserved. Reproduced with permission. PRIME-MD $\ ^{\circ}$  is a trademark of Pfizer Inc. A2663B 10-04-2005

#### PHQ-9 Patient Depression Questionnaire

#### For initial diagnosis:

- 1. Patient completes PHQ-9 Quick Depression Assessment.
- If there are at least 4 √s in the shaded section (including Questions #1 and #2), consider a depressive disorder. Add score to determine severity.

#### Consider Major Depressive Disorder

- if there are at least 5 √s in the shaded section (one of which corresponds to Question #1 or #2)

#### Consider Other Depressive Disorder

- if there are 2-4 √s in the shaded section (one of which corresponds to Question #1 or #2)

Note: Since the questionnaire relies on patient self-report, all responses should be verified by the clinician, and a definitive diagnosis is made on clinical grounds taking into account how well the patient understood the questionnaire, as well as other relevant information from the patient.

Diagnoses of Major Depressive Disorder or Other Depressive Disorder also require impairment of social, occupational, or other important areas of functioning (Question #10) and ruling out normal bereavement, a history of a Manic Episode (Bipolar Disorder), and a physical disorder, medication, or other drug as the biological cause of the depressive symptoms.

### To monitor severity over time for newly diagnosed patients or patients in current treatment for depression:

- Patients may complete questionnaires at baseline and at regular intervals (eg, every 2 weeks) at home and bring them in at their next appointment for scoring or they may complete the questionnaire during each scheduled appointment.
- 2. Add up √s by column. For every √: Several days = 1 More than half the days = 2 Nearly every day = 3
- 3. Add together column scores to get a TOTAL score.
- 4. Refer to the accompanying PHQ-9 Scoring Box to interpret the TOTAL score.
- Results may be included in patient files to assist you in setting up a treatment goal, determining degree of response, as well as guiding treatment intervention.

#### Scoring: add up all checked boxes on PHQ-9

For every ✓ Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3

#### Interpretation of Total Score

| Total Score | Depression Severity |
|-------------|------------------------------|
| 1-4 | Minimal depression |
| 5-9 | Mild depression |
| 10-14 | Moderate depression |
| 15-19 | Moderately severe depression |
| 20-27 | Severe depression |

PHQ9 Copyright © Pfizer Inc. All rights reserved. Reproduced with permission. PRIME-MD ® is a trademark of Pfizer Inc.

A2662B 10-04-2005

FertiQoL International
Fertility Quality of Life Questionnaire (2008)
For each question, kindly check (tick the box) for the response that most closely reflects how you think and feel. Relate your answers to your current thoughts and feelings. Some questions may relate to your private life, but they are necessary to adequately measure all aspects of your life.

Please complete the items marked with an asterisk (\*) only if you have a partner.

| | Please complete the items marked with a | n asterisk ( | ) only if yo | u nave a partn | er. | |
|---|---|---|---|---|---|---|
| | For each question, check the response that is closest to your<br>current thoughts and feelings | Very Poor | Poor | Nor good nor<br>poor | Good | Very<br>Good |
| Α | How would you rate your health? | | | | | |
| | For each question, check the response that is closest to your current thoughts and feelings | Very<br>Dissatisfied | Dissatisfied | Neither Satisfied<br>Nor Dissatisfied | Satisfied | Very<br>Satisfied |
| В | Are you satisfied with your quality of life? | | | | | |
| | For each question, check the response that is closest to your current thoughts and feelings | Completely | A Great<br>Deal | Moderately | Not<br>Much | Not At All |
| Q1 | Are your attention and concentration impaired by thoughts of infertility? | | _ | | | |
| Q2 | Do you think you cannot move ahead with other life goals and plans because of fertility problems? | | | | | |
| Q3 | Do you feel drained or worn out because of fertility problems? | | | | | |
| Q4 | Do you feel able to cope with your fertility problems? | | | | | |
| | For each question, check the response that is closest to your current thoughts and feelings | Very<br>Dissatisfied | Dissatisfied | Neither Satisfied<br>Nor Dissatisfied | Satisfied | Very<br>Satisfied |
| Q5 | Are you satisfied with the support you receive from friends with regard to your fertility problems? | | | | | |
| *Q6 | Are you satisfied with your sexual relationship even though you have fertility problems? | | | | | |
| | For each question, check the response that is closest to your<br>current thoughts and feelings | Always | Very Often | Quite Often | Seldom | Never |
| Q7 | Do your fertility problems cause feelings of jealousy and resentment? | | | | | |
| Q8 | Do you experience grief and/or feelings of loss about not being able to have a child (or more children)? | | | | | |
| Q9 | Do you fluctuate between hope and despair because of fertility problems? | | | | | |
| Q10 | Are you socially isolated because of fertility problems? | | | | | |
| *Q11 | Are you and your partner affectionate with each other even though you have fertility problems? | | | | | _ |
| Q12 | Do your fertility problems interfere with your day-to-day work or obligations? | | | | | |
| Q13 | Do you feel uncomfortable attending social situations like holidays and celebrations because of your fertility problems? | | 0 | | 0 | 0 |
| Q14 | Do you feel your family can understand what you are going through? | | | | | |
| | For each question, check the response that is closest to your current thoughts and feelings | An<br>Extreme<br>Amount | Very Much | A Moderate<br>Amount | A Little | Not At All |
| *Q15 | Have fertility problems strengthened your commitment to your partner? | | | | | |
| Q16 | Do you feel sad and depressed about your fertility problems? | | | | | |
| Q17 | Do your fertility problems make you inferior to people with children? | | | | | |
| Q18 | Are you bothered by fatigue because of fertility problems? | | | | | |
| *Q19 | Have fertility problems had a negative impact on your relationship with your partner? | 0 | 0 | 0 | | |
| *Q20 | Do you find it difficult to talk to your partner about your feelings related to infertility? | | | | | |
| *Q21 | Are you content with your relationship even though you have fertility problems? | 0 | 0 | 0 | 0 | |
| Q22 | Do you feel social pressure on you to have (or have more) children? | | | | | |
| Q23 | Do your fertility problems make you angry? | | | | | |
| Q24 | Do you feel pain and physical discomfort because of your fertility problems? | | | | | |

<sup>©</sup> European Society of Human Reproduction & Embryology and American Society of Reproductive Medicine

Revised 09/25/08

#### **EPWORTH SLEEPINESS SCALE (ESS)**

The following questionnaire will help you measure your general level of daytime sleepiness. You are to rate the chance that you would *doze off or fall asleep* during different routine daytime situations. Answers to the questions are rated on a reliable scale called the Epworth Sleepiness Scale (ESS). Each item is rated from 0 to 3: with 0 meaning you would never *doze or fall asleep* in a given situation; and 3 meaning that there is a very high chance that you would *doze or fall asleep* in that situation.

How likely are you to *doze off or fall asleep* in the following situations, in contrast to just feeling tired? Even if you haven't done some of the activities recently, think about how they would have affected you.

Use this scale to choose the most appropriate number for each situation:

0 = would never doze
2 = moderate chance of dozing
1 = slight chance of dozing
3 = high chance of dozing
It is important that you circle a number (0 to 3) for EACH situation.

| SITUATION | CHA | NCE | OF DO | ZING |
|---|---|---|---|---|
| Sitting and Reading | 0 | 1 | 2 | 3 |
| Watching Television | 0 | 1 | 2 | 3 |
| Sitting inactive in a public place (theater/meeting) | 0 | 1 | 2 | 3 |
| As a passenger in a car for an hour without a break | 0 | 1 | 2 | 3 |
| Lying down to rest in the afternoon | 0 | 1 | 2 | 3 |
| Sitting and talking to someone | 0 | 1 | 2 | 3 |
| Sitting quietly after lunch (with no alcohol) | 0 | 1 | 2 | 3 |
| In a car, while stopped in traffic | 0 | 1 | 2 | 3 |
| | TOTAL SO | ORE . | | |
| Name: | | | | |
| Date: | | | | |

#### STOP BANG Questionnaire

| Height inches/cm Weight lb/kg |
|---|
| Age<br>Male/Female<br>BMI |
| Collar size of shirt: S, M, L, XL, or inches/cm Neck circumference* cm |
| <del></del> |
| 1. Shoring Do you snore loudly (louder than talking or loud enough to be heard through closed doors)? |
| Yes No |
| 2. Tired Do you often feel tired, fatigued, or sleepy during daytime? |
| Yes No |
| 3. Observed Has anyone observed you stop breathing during your sleep? |
| Yes No |
| 4. Blood pressure |
| Do you have or are you being treated for high blood pressure? Yes No |
| 5. <i>B</i> MI |
| BMI more than 35 kg/m <sup>2</sup> ?<br>Yes No |
| 6. Age |
| Age over 50 yr old? Yes No |
| ies no |
| 7. Neck circumference Neck circumference greater than 40 cm? |
| Yes No |
| 8. Gender |
| Gender male? Yes No |
| * Neck circumference is measured by staff |
| High risk of OSA: answering yes to three or more items Low risk of OSA: answering yes to less than three items |
| Adapted from: |

#### STOP Questionnaire

A Tool to Screen Patients for Obstructive Sleep Apnea
Frances Chung, F.R.C.P.C.,\* Balaji Yegneswaran, M.B.B.S., † Pu Liao, M.D., ‡ Sharon A. Chung, Ph.D.,
\$
Santhira Vairavanathan, M.B.B.S., Sazzadul Islam, M.Sc., Ali Khajehdehi, M.D., † Colin M. Shapiro, F.R.C.P.C.#
Anesthesiology 2008; 108 812–21 Copyright © 2008, the American Society of Anesthesiologists, Inc. Lippincott Williams & Wilkins, Inc.

#### 23 Appendix L: Female Sexual Distress Scale (FSDS- Revised 2005)

#### **INSTRUCTIONS**

Below is a list of feelings and problems that women sometimes have concerning their sexuality. Please read each item carefully, and circle the number that best describes HOW OFTEN THAT PROBLEM HAS BOTHERED YOU OR CAUSED YOU DISTRESS DURING THE PAST 7 DAYS INCLUDING TODAY. Circle only one number for each item, and take care not to skip any items. If you change your mind, erase your first circle carefully. Read the example before beginning, and if you have any questions please ask about them.

Example: How often did you feel: Personal responsibility for your sexual problems.

| NEVER | RARELY | OCCASIONALLY | FRE | QUEN | TLY | ALW | /AYS |
|---|---|---|---|---|---|---|---|
| 0 | 1 | 2 | | 3 | | 4 | 4 |
| HOW OFTE | N DID YOU FE | EL: | | | | | |
| 1. Distresse | d about your se | ex life | 0 | 1 | 2 | 3 | 4 |
| 2. Unhappy | about your sex | ual relationship | 0 | 1 | 2 | 3 | 4 |
| 3. Guilty abo | out sexual diffic | ulties | 0 | 1 | 2 | 3 | 4 |
| 4. Frustrated | d by your sexua | al problems | 0 | 1 | 2 | 3 | 4 |
| 5. Stressed about sex | | | 0 | 1 | 2 | 3 | 4 |
| 6. Inferior be | ecause of sexua | al problems | 0 | 1 | 2 | 3 | 4 |
| 7. Worried a | bout sex | | 0 | 1 | 2 | 3 | 4 |
| 8. Sexually i | inadequate | | 0 | 1 | 2 | 3 | 4 |
| 9. Regrets a | about your sexu | ality | 0 | 1 | 2 | 3 | 4 |
| 10. Embarra | assed about sex | kual problems | 0 | 1 | 2 | 3 | 4 |
| 11. Dissatis | fied with your s | ex life | 0 | 1 | 2 | 3 | 4 |
| 12. Angry about your sex life | | | 0 | 1 | 2 | 3 | 4 |
| 13. Bothere | d by low sexual | desire | 0 | 1 | 2 | 3 | 4 |

Copyright ■ □2000 by American Foundation for Urological Disease Inc.

# 24 Appendix M: International Index of Erectile Function (IIEF)

(Write the number that best describes your erectile function <u>for the past 4 weeks</u> in the spaces provided.)

| Over the past four weeks: 1. How often were you able to get an erection during sexual activity? | <ul> <li>0 = No sexual activity</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
|---|---|
| 2. When you had erections with sexual stimulation, how often were your erections hard enough for penetration? | <ul> <li>0 = No sexual activity</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 3. When you attempted sexual intercourse, how often were you able to penetrate (enter) your partner? | <ul> <li>0 = Did not attempt intercourse</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 4. During intercourse, <u>how often</u> were you able to maintain your erection after you had penetrated (entered) your partner? | <ul> <li>0 = Did not attempt intercourse</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 5. During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse? | <ul> <li>0 = Did not attempt intercourse</li> <li>1 = Extremely difficult</li> <li>2 = Very difficult</li> <li>3 = Difficult</li> <li>4 = Slightly difficult</li> <li>5 = Not difficult</li> </ul> |
| 6. How many times have you attempted sexual intercourse? | 0 = No attempts 1 = One to two attempts 2 = Three to four attempts |

| | 4 = Seven to ten attempts 5 = Eleven or more attempts |
|---|---|
| 7. When you attempted sexual intercourse, how often was it satisfactory for you? | <ul> <li>0 = Did not attempt intercourse</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 8. How much have you enjoyed sexual intercourse? | <ul> <li>0 = No intercourse</li> <li>1 = No enjoyment</li> <li>2 = Not very enjoyable</li> <li>3 = Fairly enjoyable</li> <li>4 = Highly enjoyable</li> <li>5 = Very highly enjoyable</li> </ul> |
| 9. When you had sexual stimulation <u>or</u> intercourse, how often did you ejaculate? | <ul> <li>0 = No sexual stimulation/intercourse</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 10. When you had sexual stimulation <u>or</u> intercourse, how often did you have the feeling of orgasm or climax? | <ul> <li>0 = No sexual stimulation/intercourse</li> <li>1 = Almost never/never</li> <li>2 = A few times (much less than half the time)</li> <li>3 = Sometimes (about half the time)</li> <li>4 = Most times (much more than half the time)</li> <li>5 = Almost always/always</li> </ul> |
| 11. How often have you felt sexual desire? | 1 = Almost never/never 2 = A few times (much less than half the time) 3 = Sometimes (about half the time) 4 = Most times (much more than half the time) 5 = Almost always/always |
| 12. How would you rate your sexual desire? | 1 = Very low/none at all<br>2 = Low<br>3 = Moderate |

3 = Five to six attempts

| | 4 = High<br>5 = Very high |
|---|---|
| 13. How satisfied have you been with your overall sex life? | <ul> <li>1 = Very dissatisfied</li> <li>2 = Moderately dissatisfied</li> <li>3 = About equally satisfied and dissatisfied</li> <li>4 = Moderately satisfied</li> <li>5 = Very satisfied</li> </ul> |
| 14. How satisfied have you been with your sexual relationship with your partner? | <ul> <li>1 = Very dissatisfied</li> <li>2 = Moderately dissatisfied</li> <li>3 = About equally satisfied and dissatisfied</li> <li>4 = Moderately satisfied</li> <li>5 = Very satisfied</li> </ul> |
| 15. How would you rate your <u>confidence</u> that you could get and keep an erection? | 1 = Very low 2 = Low 3 = Moderate 4 = High 5 = Very high |

\*RC Rosen, A Riley, G Wagner et al. The international index of erectile dysfunction (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology 1997 49: 822-30.

Copyright © 2004 Urology Specialists, S.C. All rights reserved. Last Updated: 18 May 2004

NATIONAL INSTITUTES OF HEALTH

#### Diet History Questionnaire II



#### **GENERAL INSTRUCTIONS**

- Answer each question as best you can. Estimate if you are not sure. A guess is better than leaving a blank.
- Use only a black ball-point pen. Do not use a pencil or felt-tip pen. Do not fold, staple, or tear the pages.
- Put an X in the box next to your answer.
- If you make any changes, cross out the incorrect answer and put an  $\boldsymbol{X}$  in the box next to the correct answer. Also draw a circle around the correct answer.
- If you mark NEVER, NO, or DON'T KNOW for a question, please follow any arrows or instructions that direct you to the next question.

BEFORE TURNING THE PAGE, PLEASE COMPLETE THE FOLLOWING QUESTIONS.

#### Today's date:

| MONTH | DAY | YEAR |
|---|---|---|
| Jan Feb Mar Apr Jun Jul Sep Oct Noc | | ☐ 2012<br>☐ 2013<br>☐ 2014<br>☐ 2015<br>☐ 2016<br>☐ 2017 |

| DHQ | II | Pas | stY | ea |
|-----|----|-----|-----|----|

| In what month | were |
|---------------|------|
| you born? | |
| you boilir | |

| | Jan |
|---|------------|
| | Feb |
| | Mar |
| | • |
| | May |
| | Jun |
| _ | Jul |
| _ | Aug |
| | Sep |
| | Oct |
| | Nov<br>Dec |

#### In what year were you born?



#### Are you male or female?

| <b>∐Male</b> |
|--------------|
| □Female |

| BAR CODE LABEL OR SUBJECT ID<br>HERE |
|--------------------------------------|

| 1 | . Over the <u>past 12 months</u> , how often did you drink carrot juice? | 3b. How often was the orange juice or grapefruit juice you drank calcium-fortified? |
|---|---|---|
| | NEVER (GO TO QUESTION 2) ☐ 1 time per month or less ☐ 1 time per day ☐ 2–3 times per month ☐ 2–3 times per day ☐ 1–2 times per week ☐ 4–5 times per day ☐ 3–4 times per week ☐ 6 or more times per day ☐ 5–6 times per week | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 33 | □ 5-6 times per week 1a. Each time you drank carrot juice, how much did you usually drink? □ Less than ½ cup (4 ounces) □ ½ to 1½ cups (4 to 10 ounces) □ More than 1½ cups (10 ounces) 2. Over the past 12 months, how often did you drink tomato juice or other vegetable juice? (Please do not include carrot juice.) □ NEVER (GO TO QUESTION 3) □ 1 time per month or less □ 1 time per day □ 2-3 times per month □ 2-3 times per day □ 1-2 times per week □ 4-5 times per day □ 3-4 times per week □ 6 or more times per day □ 5-6 times per week 2a. Each time you drank tomato juice or other vegetable juice, how much did you usually drink? □ Less than ¾ cup (6 ounces) □ ⅓ to 1⅓ cups (6 to 10 ounces) □ More than 1⅓ cups (10 ounces) | 4. Over the past 12 months, how often did you drink other 100% fruit juice or 100% fruit juice mixtures (such as apple, grape, pineapple, or others)? NEVER (GO TO QUESTION 5) |
| ₩ | , | ▼ |

| Over the <u>past 12 months</u> | 7a. Each time you drank chocolate milk, how |
|---|---|
| 5a. Each time you drank <b>fruit drinks</b> , how much did you usually drink? Less than 1 cup (8 ounces) 1 to 2 cups (8 to 16 ounces) More than 2 cups (16 ounces) | much did you usually drink? Less than 1 cup (8 ounces) 1 to 1½ cups (8 to 12 ounces) More than 1½ cups (12 ounces) Tb. How often was the chocolate milk reduced-fat or fat-free? |
| 5b. How often were your fruit drinks diet or sugar-free? Almost never or never About ¼ of the time About ½ of the time About ¾ of the time About ¾ of the time About ¾ of the time Almost always or always 6. How often did you drink milk as a beverage (NOT in coffee, NOT in cereal)? (Please do not include chocolate milk and hot chocolate.) NEVER (GO TO QUESTION 7) 1 time per month or less 1 time per day | □ Almost never or never □ About 1/4 of the time □ About 1/2 of the time □ About 1/4 of the time □ Almost always or always 8: How often did you drink meal replacement or high-protein beverages (such as Instant Breakfast, Ensure, Slimfast, Sustacal or others)? □ NEVER (GO TO QUESTION 9) □ 1 time per month or less □ 1 time per day □ 2-3 times per month □ 2-3 times per day □ 1-2 times per week □ 4-5 times per day |
| 2-3 times per month 2-3 times per day 1-2 times per week 4-5 times per day 3-4 times per week 6 or more times per day 5-6 times per week 6 or more times per day 5-6 times per week 6 or more times per day 5-6 times per week 6 or more times per day 7 or more times 7 or more | 3-4 times per week 6 or more times per day 5-6 times per week 8a. Each time you drank meal replacement or high-protein beverages, how much did you usually drink? Less than 1 cup (8 ounces) 1 to 1½ cups (8 to 12 ounces) More than 1½ cups (12 ounces) More than 1½ cups (12 ounces) 9. Over the past 12 months, did you drink soda or pop? NO (GO TO QUESTION 10) YES 9a. How often did you drink soda or pop IN THE SUMMER? 1 time per month or less 1 time per day 2-3 times per month 2-3 times per day 1-2 times per week 4-5 times per day 3-4 times per week 6 or more times per day 5-6 times per week per day per day 5-6 times per week per day per day 5-6 times per week per day per day 5-6 times per week per day 5-6 t |

| ( | Over th | ne <u>past 12 months</u> | 1 | 0b. | How often did you drink sports drinks DURING THE REST OF THE YEAR? |
|---|---|---|---|---|---|
| | 9b. | How often did you drink soda or pop DURING THE REST OF THE YEAR? | | | □NEVER |
| | | □ NEVER □ 1 time per month or less □ 1 time per day | | | ☐ 1 time per month or less ☐ 1 time per day ☐ 2–3 times per month ☐ 2–3 times per day ☐ 1–2 times per week ☐ 4–5 times per day ☐ 3–4 times per week ☐ 6 or more times |
| | | ☐ 2–3 times per month ☐ 1–2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 5 fimes per week ☐ 2–3 times per day ☐ 4–5 times per day ☐ 6 or more times ☐ per day | 1 | 0c. | □ 5–6 times per week per day Each time you drank sports drinks, how much did you usually drink? |
| | 9c. | Each time you drank <b>soda</b> or <b>pop</b> , how much did you usually drink? | | | Less than 12 ounces or less than 1 bottle 12 to 24 ounces or 1 to 2 bottles |
| | | ☐ Less than 12 ounces or less than 1 can or bottle☐ 12 to 16 ounces or 1 can or bottle☐ More than 16 ounces or more than 1 can or bottle | 11. | | More than 24 ounces or more than 2 bottles ver the past 12 months, did you drink energy |
| | 9d. | How often were these sodas or pop <b>diet</b> or <b>sugar-free</b> ? | _ | | inks (such as Red Bull or Jolt)? NO (GO TO QUESTION 12) |
| | 9e. | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ Almost always or always How often were these sodas or pop caffeine-free? ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ About ¾ of the time ☐ About ¾ of the time | | | How often did you drink energy drinks IN THE SUMMER? NEVER 1 time per month or less 2-3 times per month 1-2 times per week 3-4 times per week 5-6 times per week per day |
| | dr | Almost always or always ver the <u>past 12 months</u> , did you drink <b>sports</b> inks (such as Propel, PowerAde, or atorade)? | 1 | 1b. | How often did you drink energy drinks DURING THE REST OF THE YEAR? NEVER 1 time per month or less 1 time per day |
| | ₽□ | NO (GO TO QUESTION 11)<br>YES | | | □ 2–3 times per month □ 1–2 times per week □ 3–4 times per week □ 5–6 times per week □ 5–6 times per week |
| | 10a. | How often did you drink sports drinks IN THE SUMMER? | 1 | 1c. | Each time you drank energy drinks, how much did you usually drink? |
| | | □ NEVER □ 1 time per month or less □ 2–3 times per month □ 1–2 times per week □ 3–4 times per week □ 5–6 times per week □ 5–6 times per week □ 1 time per day □ 2–3 times per day □ 4–5 times per day □ 6 or more times □ per day | | | ☐ Less than 8 ounces or less than 1 cup ☐ 8 to 16 ounces or 1 to 2 cups ☐ More than 16 ounces or more than 2 cups |

| bottled, and carbonated water) <b>DURING</b> |
|---|
| THE REST OF THE YEAR? |
| □NEVER |
| ☐ 1 time per month or less ☐ 1 time per day ☐ 2–3 times per month ☐ 2–3 times per day ☐ 1–2 times per week ☐ 4–5 times per day ☐ 6 or more times ☐ 5–6 times per week ☐ per day ☐ 6 or more times ☐ 5–6 times per week ☐ 6 or more times ☐ 5–6 times per week ☐ 6 or more times ☐ 5–6 times per week ☐ 6 or more times ☐ 5–6 times per week ☐ 6 or more times ☐ 5–6 times per week ☐ 5 or more times ☐ 5–6 times per week ☐ 5 or more times ☐ 5 or more tim |
| <ul> <li>13c. Each time you drank water, how much did you usually drink?</li> <li>Less than 12 ounces or less than 1 bottle</li> <li>12 to 24 ounces or 1 to 2 bottles</li> <li>More than 24 ounces or more than 2 bottles</li> <li>13d. How often was the water you drank tap</li> </ul> |
| water? Almost never or never About ¼ of the time About ½ of the time About ¾ of the time Almost always or always 13e. How often was the water you drank bottled, sweetened water (with low or no-calorie sweetener, including carbonated water)? Almost never or never About ¼ of the time About ¼ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time Almost always or always 13f. How often was the water you drank bottled, unsweetened water (including carbonated water)? |
| Almost never or never About 1/4 of the time About 1/2 of the time About 1/2 of the time Almost always or always 4. How often did you drink wine or wine coolers? NEVER (GO TO QUESTION 15) 1 time per month or less 1 time per day 2-3 times per month 2-3 times per day 1-2 times per week 4-5 times per day 3-4 times per week 6 or more times per day 5-6 times per week |

| Over the <u>past 12 months</u> | 16c. Each time you ate oatmeal, grits, or other cooked cereal, how much did you usually |
|---|---|
| 14a. Each time you drank wine or wine coolers,<br>how much did you usually drink? | eat?<br>□ Less than ¾ cup |
| ☐ Less than 5 ounces or less than 1 glass☐ 5 to 12 ounces or 1 to 2 glasses☐ More than 12 ounces or more than 2 glasses | ☐ 3/4 to 11/4 cups ☐ More than 11/4 cups |
| 15. How often did you drink liquor or mixed drinks? | 16d. How often was butter or margarine added<br>to your oatmeal, grits or other cooked<br>cereal? |
| ☐ NEVER (GO TO QUESTION 16) | ☐ Almost never or never<br>☐ About ¼ of the time |
| □ 1 time per month or less □ 1 time per day □ 2–3 times per month □ 2–3 times per day □ 1–2 times per week □ 4–5 times per day □ 3–4 times per week □ 6 or more times per day | ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 5–6 times per week | 17. How often did you eat cold cereal? |
| 15a. Each time you drank liquor or mixed drinks, how much did you usually drink? Less than 1 shot of liquor 1 to 3 shots of liquor More than 3 shots | NEVER (GO TO QUESTION 18) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 to 2½ cups More than 2½ cups More than 2½ cups More than 2½ cups Almost never or never About ¼ of the time About ¼ of the time About ¾ of the time Almost always or always 17c. How often was the cold cereal you ate All Bran, Fiber One, 100% Bran, or All-Bran Bran Buds? Almost never or never About ¼ of the time About ¼ of the time About ¼ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time Almost always or always Almost always Almost a |

| Over th | ne <u>past 12 months</u> | | 18a. | Each time you ate a | applesauce, how much |
|---|---|---|---|---|---|
| 17d. | How often was the cold cereal you ate some other bran or fiber cereal (such as Cheerios, Shredded Wheat, Raisin Bran, Bran Flakes, Grape-Nuts, Granola, Wheaties, or Healthy Choice)? | | | Less than ½ cup ½ to 1 cup More than 1 cup | |
| 17e. | □ Almost never or never □ About ¼ of the time □ About ¾ of the time □ About ¾ of the time □ Almost always or always How often was the cold cereal you ate any other type of cold cereal (such as Corn Flakes, Rice Krispies, Frosted Flakes, Special K, Froot Loops, Cap'n Crunch, or others)? □ Almost never or never □ About ¼ of the time □ About ⅓ of the time □ About ¾ of the time □ Almost always or always | | | w often did you eat a NEVER (GO TO QUES 1–6 times per year 7–11 times per year 1 time per month 2–3 times per month 1 time per week Each time you ate a you usually eat? Less than 1 apple 1 apple More than 1 apple | |
| 17f. | Was milk added to your cold cereal? | : | | w often did you eat p<br>zen)? | ears (fresh, canned, or |
| 17h. | What kind of milk was usually added? Whole milk 2% fat milk 1% fat milk Skim, nonfat, or ½% fat milk Soy milk Rice milk Other Each time milk was added to your cold cereal, how much was usually added? Less than ½ cup ½ to 1 cup More than 1 cup wo often did you eat applesauce? NEVER (GO TO QUESTION 19) 1–6 times per year 7–11 times per year 1 time per month 2–3 times per month 1 time per day 1 time per week 2 or more times per day | | 20a. | NEVER (GO TO QUEST—1–6 times per year 7–11 times per year 1 time per month 2–3 times per month 1 time per week Each time you ate pusually eat? Less than 1 pear In pear In pear In More than 1 pear woften did you eat be never week 1–6 times per year 1–11 times per year 1 time per month 2–3 times per month 1 time per week | 2 times per week 3-4 times per week 5-6 times per week 1 time per day 2 or more times per day pears, how many did you |
| <b>\</b> | | , | ļ | | |

| Over the past 12 months | 23c. Each time you ate peaches, nectarines, or plums, how much did you usually eat? |
|---|---|
| 21a. Each time you ate bananas, how many did you usually eat? ☐ Less than 1 banana ☐ 1 banana | ☐ Less than 1 fruit or less than ½ cup☐ 1 to 2 fruits or ½ to ¾ cup☐ More than 2 fruits or more than ¾ cup |
| ☐ More than 1 banana | 24. How often did you eat grapes? |
| 22. How often did you eat dried fruit (such as prunes or raisins)? (Please do not include dried apricots.) NEVER (GO TO QUESTION 23) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 22a. Each time you ate dried fruit, how much did you usually eat? Less than 2 tablespoons 2 to 5 tablespoons More than 5 tablespoons | NEVER (GO TO QUESTION 25) □ 1–6 times per year □ 2 times per week □ 7–11 times per year □ 3–4 times per week □ 1 time per month □ 5–6 times per week □ 2–3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day 24a. Each time you ate grapes, how much did you usually eat? □ Less than ½ cup or less than 10 grapes □ ½ to 1 cup or 10 to 30 grapes □ More than 1 cup or more than 30 grapes □ More than 1 cup or more than 30 grapes 25. Over the past 12 months, did you eat cantaloupe? |
| 23. Over the past 12 months, did you eat peaches, nectarines, or plums? | NO (GO TO QUESTION 26) YES 25a. How often did you eat fresh cantaloupe WHEN IN SEASON? |
| <b>↓</b> □YES | □ NEVER |
| 23a. How often did you eat fresh peaches, nectarines, or plums WHEN IN SEASON? NEVER 1-6 times per season 2 times per week 7-11 times per season 3-4 times per week | ☐ 1–6 times per season ☐ 2 times per week ☐ 7–11 times per season ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |
| ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | 25b. How often did you eat cantaloupe (fresh or frozen) DURING THE REST OF THE YEAR? |
| 23b. How often did you eat peaches, nectarines, or plums (fresh, canned, or frozen) DURING THE REST OF THE YEAR? NEVER 1-6 times per year | □ NEVER □ 1-6 times per year □ 2 times per week □ 7-11 times per year □ 3-4 times per week □ 1 time per month □ 5-6 times per week □ 2-3 times per month □ 1 time per day □ 1 time per week □ 2 or more times □ per day |
| po. 44, | |

| Over the <u>past 12 months</u> | 27. Over the <u>past 12 months</u> , did you eat<br>strawberries? |
|---|---|
| 25c. Each time you ate cantaloupe, how much did you usually eat? | NO (GO TO QUESTION 28) |
| Less than ¼ melon or less than ½ cup ¼ melon or ½ to 1 cup More than ¼ melon or more than 1 cup | YES 27a. How often did you eat fresh strawberries WHEN IN SEASON? |
| 26. Over the past 12 months, did you eat melon, other than cantaloupe (such as watermelon or honeydew)? NO (GO TO QUESTION 27) YES 26a. How often did you eat fresh melon, other than cantaloupe, WHEN IN SEASON? NEVER 1-6 times per season 7-11 times per season 1 time per month 1 time per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 26b. How often did you eat melon other than | NEVER 1–6 times per season 2 times per week 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 2 or more times per day 27b. How often did you eat strawberries (fresh or frozen) DURING THE REST OF THE YEAR? NEVER 1–6 times per year 2 times per week 1 time per month 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 2 or more times per day |
| cantaloupe (fresh or frozen) DURING THE REST OF THE YEAR? NEVER 1-6 times per year | 27c. Each time you ate strawberries, how much did you usually eat? Less than ¼ cup or less than 3 berries ¼ to ¾ cup or 3 to 8 berries More than ¾ cup or more than 8 berries 28. Over the past 12 months, did you eat oranges, tangerines, or clementines? NO (GO TO QUESTION 29) |
| 26c. Each time you ate melon other than cantaloupe, how much did you usually eat? Less than ½ cup or 1 small wedge More than 2 cups or 1 large wedge | YES 28a. How often did you eat fresh oranges, tangerines, or clementines WHEN IN SEASON? NEVER 1-6 times per season 7-11 times per season 1 time per month 2-3 times per week 1 time per week 1 time per week 2-3 times per week 1 time per week 1 time per week 2 or more times per day |

| Over the past 12 months | | 29c. | | grapefruit, how much did | | |
|---|---|---|---|---|---|---|
| | 28b. | How often did you eat or or clementines (fresh or THE REST OF THE YEAR | canned) <b>DURING</b> | | you usually eat? Less than ½ grapef ½ grapefruit More than ½ grape | |
| | | □ NEVER | | | ☐ More than ½ grape | truit |
| | 28c. | ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week Each time you ate orang clementines, how many | | | NEVER (GO TO QUES<br>1–6 times per year<br>7–11 times per year<br>1 time per month<br>2–3 times per month<br>1 time per week | |
| | | ☐ Less than 1 fruit☐ 1 fruit☐ More than 1 fruit | | | you usually eat? | less than 1 medium slice |
| 29 | | er the <u>past 12 months,</u> did<br>apefruit? | you eat | | 1/4 to 3/4 cup or 1 me | |
| Г | — | NO (GO TO QUESTION 30) | | 31. Ha | ow often did you eat <b>o</b> | ther kinds of fruit? |
| | $\Box$ | YES | | | NEVER (GO TO QUES | STION 32) |
| | <b>∀</b><br>29a. | How often did you eat fre WHEN IN SEASON? | esh grapefruit | | 1–6 times per year<br>7–11 times per year<br>1 time per month<br>2–3 times per month<br>1 time per week | ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 or more times per day |
| | | ☐ 1–6 times per season☐ 7–11 times per season☐ 1 time per month☐ 2–3 times per month☐ 1 time per week☐ | 2 times per week 3–4 times per week 5–6 times per week 1 time per day 2 or more times per day | 31a. | Each time you ate of much did you usuall Less than ¼ cup ¼ to ¾ cup More than ¾ cup | other kinds of fruit, how<br>ly eat? |
| | 29b. | How often did you eat grace canned) DURING THE RYEAR? | | as | ow often did you eat <b>C</b><br>spinach, turnip, colla<br>le)? | COOKED greens (such<br>rd, mustard, chard, or |
| | | □ NEVER | | | NEVER (GO TO QUES | STION 33) |
| | | ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week | ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 or more times per day | | 1–6 times per year<br>7–11 times per year<br>1 time per month<br>2–3 times per month<br>1 time per week | ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 or more times per day |

| Over the past 12 months | 35a. Each time you ate sauerkraut or cabbage, how much did you usually eat? |
|---|---|
| 32a. Each time you ate COOKED greens, how much did you usually eat? Less than ½ cup ½ to 1 cup | Less than ¼ cup ¼ to 1 cup More than 1 cup |
| More than 1 cup 33. How often did you eat RAW greens (such as spinach, turnip, collard, mustard, chard, or kale)? (We will ask about lettuce later.) NEVER (GO TO QUESTION 34) 1-6 times per year 2 times per week 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 33a. Each time you ate RAW greens, how much did you usually eat? Less than ½ cup ½ to 1 cup | 36. How often did you eat carrots (fresh, canned, or frozen)? NEVER (GO TO QUESTION 37) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 36a. Each time you ate carrots, how much did you usually eat? Less than ½ cup or less than 2 baby carrots ½ to ½ cup or 2 to 5 baby carrots More than ½ cup or more than 5 baby carrots |
| ☐ More than 1 cup ■ More than 1 cup ■ 34. How often did you eat coleslaw? | 37. How often did you eat string beans or green beans (fresh, canned, or frozen)? NEVER (GO TO QUESTION 38) |
| NEVER (GO TO QUESTION 35) 1–6 times per year | ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week ☐ 2 or more times per day ☐ 37a. Each time you ate string beans or green beans, how much did you usually eat? |
| 34a. Each time you ate coleslaw, how much did you usually eat? □ Less than ¼ cup □ ¼ to ¾ cup □ More than ¾ cup ■ Sauerkraut or cabbage (other than coleslaw)? □ NEVER (GO TO QUESTION 36) □ 1–6 times per year □ 7–11 times per year □ 1 time per month □ 1–6 times per week □ 1 time per month □ 1–6 times per week □ 1 time per month □ 1–6 times per week □ 1 time per week □ 2–3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day | Less than ½ cup ½ to 1 cup More than 1 cup 38. How often did you eat peas (fresh, canned, or frozen)? NEVER (GO TO QUESTION 39) 1–6 times per year 7–11 times per year 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day |
| T unite per week | |

| 38a. Each time you ate peas, how much did you usually eat? Less than ½ cup | Over the <u>past 12 months</u> | 40. How often did you eat <b>broccoli</b> (fresh or |
|---|---|---|
| Less than ¼ cup | | frozen)? — NEVER (GO TO QUESTION 41) |
| No (GO TO QUESTION 40) | ☐ Less than ¼ cup ☐ ¼ to ¾ cup ☐ More than ¾ cup | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day |
| you usually eat? YES 39a. How often did you eat fresh corn WHEN IN SEASON? NEVER | | 40a. Each time you ate broccoli, how much did |
| SEASON? % to 1 cup % to 2 cup % to 1 cup % to | | you usually eat? |
| 1-6 times per season 2 times per week 7-11 times per season 3-4 times per week 2-3 times per month 5-6 times per week 1 time per month 1 time per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 times per week 1 time per month 1 time per day 1 time per month 1 time per month 1 time per month 1 time per month 1 time per week 2 or more times per week 1-6 times per year 2 times per week 2 or more times per week 1 time per month 1 time per month 1 time per month 2-3 times per week 2 or more times per day 41a. Each time you ate cauliflower or Bruss sprouts, how much did you usually eat' 42. How often did you eat asparagus (fresh or frozen)? 42. How often did you eat asparagus (fresh or frozen)? 42. How often did you eat asparagus (fresh or frozen)? 42. How often did you eat asparagus (fresh or frozen)? 42. How often did you eat asparagus (fresh or frozen)? 43. Each time per week 2 or more times per week 1 time per month 1 time per day 42. How often did you eat asparagus (fresh or frozen)? 44. Each time per week 2 or more times per week 1 time per month 2 times per week 3 times per week 44. Each time per month 1 time per day 45. Times per year 2 times per week 45. Times per week 46. Times per year 2 times per week 46. Times per year 3 times per week 46. Times per year 3 times per week 47. Times per year 40. Times per year 40 | → 39a. How often did you eat fresh corn WHEN IN | ☐ ¼ to 1 cup |
| ☐ ⅓ to ⅔ cup or 4 to 7 spears | □ NEVER □ 1–6 times per season □ 2 times per week □ 7–11 times per season □ 3–4 times per week □ 1 time per month □ 5–6 times per week □ 2–3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day 39b. How often did you eat corn (fresh, canned, or frozen) DURING THE REST OF THE YEAR? □ NEVER □ 1–6 times per year □ 2 times per week □ 7–11 times per year □ 3–4 times per week □ 1 time per month □ 5–6 times per week □ 1 time per month □ 1 time per day □ 1 time per week □ 2 or more times per day 39c. Each time you ate corn, how much did you usually eat? □ Less than 1 ear or less than ½ cup □ 1 ear or ½ to 1 cup | 41. How often did you eat cauliflower or Brussels sprouts (fresh or frozen)? NEVER (GO TO QUESTION 42) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 41a. Each time you ate cauliflower or Brussels sprouts, how much did you usually eat? Less than ¼ cup ¼ to ½ cup More than ½ cup More than ½ cup More than ½ cup T-11 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 42a. Each time you ate asparagus, how much |
| | | 1/₃ to 3/₃ cup or 4 to 7 spears |

| Over the past 12 months | 46. Now think about all the <b>cooked vegetables</b> you ate in the past 12 months and how they were |
|---|---|
| 43. How often did you eat winter squash (such as pumpkin, butternut, or acorn)? | prepared. How often were your vegetables COOKED WITH some sort of fat, including oil spray? (Please do not include potatoes.) |
| ☐ NEVER (GO TO QUESTION 44) | r—☐ NEVER (GO TO QUESTION 47) |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day ☐ 2. Feels times year et a winter a graph here. | □ 1–6 times per year □ 2 times per week □ 7–11 times per year □ 3–4 times per week □ 1 time per month □ 5–6 times per week □ 2–3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day |
| 43a. Each time you ate winter squash, how much did you usually eat? | |
| ☐ Less than ½ cup<br>☐ ½ to ¾ cup<br>☐ More than ¾ cup | |
| 44. How often did you eat mixed vegetables? | |
| ☐ NEVER (GO TO QUESTION 45) | |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | 46a. Which fats were usually added to your vegetables DURING COOKING? (Please do not include potatoes. Mark all that apply.) |
| 44a. Each time you ate mixed vegetables, how much did you usually eat? | ☐ Margarine ☐ Corn oil |
| ☐ Less than ½ cup☐ ½ to 1 cup☐ More than 1 cup | (including low-fat) |
| 45. How often did you eat onions? | ☐ Olive oil |
| NEVER (GO TO QUESTION 46) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day | 47. Now, thinking again about all the cooked vegetables you ate in the past 12 months, how often was some sort of fat, sauce, or dressing added AFTER COOKING OR AT THE TABLE? (Please do not include potatoes.) |
| ☐ 1 time per week ☐ 2 or more times per day | ☐ NEVER (GO TO QUESTION 48) |
| 45a. Each time you ate onions, how much did you usually eat? Less than 1 slice or less than 1 tablespoon 1 slice or 1 to 4 tablespoons More than 1 slice or more than 4 tablespoons | ☐ 1–6 times per year ☐ 3–4 times per week ☐ 7–11 times per year ☐ 5–6 times per week ☐ 1 time per month ☐ 2–3 times per month ☐ 2 times per day ☐ 3 or more times per day |

♥ Question 46 appears in the next column

| Over the <u>past 12 months</u> | tomatoes (including those in salads)? |
|---|---|
| 47a. Which fats, sauces, or dressings were<br>usually added AFTER COOKING OR AT<br>THE TABLE? (Please do not include<br>potatoes. Mark all that apply.) | NO (GO TO QUESTION 50) YES 49a. How often did you eat fresh tomatoes |
| □ Margarine | (including those in salads) WHEN IN SEASON? |
| 47b. If margarine, butter, lard, fatback, or bacon fat was added to your cooked vegetables AFTER COOKING OR AT THE TABLE, how much did you usually add? | ☐ 1-6 times per season ☐ 2 times per week ☐ 7-11 times per season ☐ 3-4 times per week ☐ 1 time per month ☐ 5-6 times per week ☐ 2 or more times per day ☐ 1 time per day ☐ 2 or more times per day |
| <ul> <li>□ Did not usually add these</li> <li>□ Less than 1 teaspoon</li> <li>□ 1 to 3 teaspoons</li> <li>□ More than 3 teaspoons</li> </ul> | 49b. How often did you eat fresh tomatoes (including those in salads) DURING THE REST OF THE YEAR? |
| 47c. If salad dressing, cheese sauce, or white sauce was added to your cooked vegetables AFTER COOKING OR AT THE TABLE, how much did you usually add? | □ NEVER □ 1–6 times per year □ 2 times per week □ 7–11 times per year □ 3–4 times per weel □ 1 time per month □ 5–6 times per weel □ 2–3 times per month □ 1 time per day |
| ☐ Did not usually add these ☐ Less than 1 tablespoon ☐ 1 to 3 tablespoons ☐ More than 3 tablespoons | ☐ 1 time per week ☐ 2 or more times per day 49c. Each time you ate fresh tomatoes, how much did you usually eat? |
| <ul><li>48. How often did you eat sweet peppers (green, red, or yellow)?</li><li> NEVER (GO TO QUESTION 49)</li></ul> | ☐ Less than ¼ tomato ☐ ¼ to ½ tomato ☐ More than ½ tomato |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 1 time per day ☐ 2 or more times per day | 50. How often did you eat lettuce salads (with or without other vegetables)? |
| 48a. Each time you ate sweet peppers, how much did you usually eat? ☐ Less than ¼ pepper ☐ ⅓ to ¼ pepper | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |
| ☐ More than ¼ pepper | |
| | 1 |

| Over the <u>past 12 months</u> | 53. How often did you eat French fries, home fries,<br>hash browned potatoes, or tater tots? |
|---|---|
| 50a. Each time you ate lettuce salads, how much did you usually eat? | ☐ NEVER (GO TO QUESTION 54) |
| Less than ¼ cup ¼ to 1¼ cups More than 1¼ cups 50b. How often did the lettuce salads you ate include dark green lettuce? | ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 or more times per day |
| Almost never or never About 1/2 of the time About 3/2 of the time About 3/2 of the time About 3/2 of the time Almost always or always | 53a. Each time you ate French fries, home fries, hash browned potatoes, or tater tots how much did you usually eat? ☐ Less than 10 fries or less than ½ cup ☐ 10 to 25 fries or ½ to 1 cup ☐ More than 25 fries or more than 1 cup |
| 51. How often did you eat salad dressing (including low-fat) on salads? | ▼ 54. How often did you eat <b>potato salad</b> ? |
| ☐ NEVER (GO TO QUESTION 52) | NEVER (GO TO QUESTION 55) |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | ☐ 1–6 times per year ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per month ☐ 1 time per week ☐ 1 time per day ☐ 2 or more times per day |
| 51a. Each time you ate salad dressing on salads, how much did you usually eat? | 54a. Each time you ate <b>potato salad</b> , how much did you usually eat? |
| Less than 2 tablespoons 2 to 4 tablespoons More than 4 tablespoons | ☐ Less than ½ cup☐ ½ to 1 cup☐ More than 1 cup☐ |
| 52. How often did you eat sweet potatoes or yams? | 55. How often did you eat baked, boiled, or<br>mashed potatoes? |
| ☐ NEVER (GO TO QUESTION 53) | ☐ NEVER (GO TO QUESTION 56) |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | ☐ 1–6 times per year ☐ 2 times per week ☐ 3–4 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per week ☐ 1 time per day ☐ 2 or more times per day |
| 52a. Each time you ate sweet potatoes or yams, how much did you usually eat? | 55a. Each time you ate baked, boiled, or mashed potatoes, how much did you usually eat? |
| ☐ 1 small potato or less than ¼ cup ☐ 1 medium potato or ¼ to ¾ cup ☐ 1 large potato or more than ¾ cup | ☐ 1 small potato or less than ½ cup ☐ 1 medium potato or ½ to 1 cup ☐ 1 large potato or more than 1 cup |
| <b>♦</b> | ▼ |

Question 53 appears in the next column

| Over the <u>past 12 months</u> | 55h. Each time <b>cheese</b> or <b>cheese sauce</b> was added to your potatoes, how much was |
|---|---|
| 55b. How often was sour cream (including low-<br>fat) added to your potatoes, EITHER IN<br>COOKING OR AT THE TABLE? | usually added? Less than 1 tablespoon 1 to 3 tablespoons |
| COOKING OR AT THE TABLE? Almost never or never (GO TO QUESTION 55d) About ¼ of the time About ¼ of the time About ¾ of the time Almost always or always 55c. Each time sour cream was added to your potatoes, how much was usually added? Less than 1 tablespoon 1 to 3 tablespoons More than 3 tablespoons More than 3 tablespoons At THE TABLE? Almost never or never About ¼ of the time About ¼ of the time About ¼ of the time About ¾ of the time About ¾ of the time About ¼ of the time | |
| ☐ Almost always or always 55f. Each time margarine or butter was added to your potatoes, how much was usually added? | Less than 1 teaspoon 1 to 6 teaspoons More than 6 teaspoons |
| Never added Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons More than 3 teaspoons 55g. How often was cheese or cheese sauce added to your potatoes, EITHER IN COOKING OR AT THE TABLE? Almost never or never (GO TO QUESTION 56) About 1/2 of the time About 1/2 of the time Almost always or always | Very series of the per week |
| <u> </u> | ☐ More than 1 cup |

Question 62 appears in the next column

| Over the past 12 months | 64f. Each time <b>syrup</b> was added to your pancakes |
|---|---|
| 64. How often did you eat pancakes, waffles, or French toast? | waffles, or French toast, how much was usually added? |
| ☐ NEVER (GO TO QUESTION 65) | ☐ Less than 1 tablespoon ☐ 1 to 4 tablespoons ☐ More than 4 tablespoons |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | 65. How often did you eat lasagna, stuffed shells, stuffed manicotti, ravioli, or tortellini? (Please do not include spaghetti or other pasta.) |
| 64a. Each time you ate pancakes, waffles, or French toast, how much did you usually eat? Less than 1 medium piece 1 to 3 medium pieces More than 3 medium pieces 64b. How often was margarine (including low-fat) added to your pancakes, waffles, or French toast AFTER COOKING OR AT THE TABLE? Almost never or never About ½ of the time About ½ of the time About ¾ of the time Almost always or always 64c. How often was butter (including low-fat) added to your pancakes, waffles, or French toast AFTER COOKING OR AT THE TABLE? Almost never or never About ½ of the time About ½ of the time About ½ of the time About ¾ of the fime Figure 1 and 1 and 1 and 2 and 2 and 3 an | (Please do not include spaghetti or other pasta.) NEVER (GO TO QUESTION 66) □ 1-6 times per year □ 2 times per week □ 7-11 times per year □ 3-4 times per week □ 1 time per month □ 5-6 times per week □ 2-3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day 65a. Each time you ate lasagna, stuffed shells, stuffed manicotti, ravioli, or tortellini, how much did you usually eat? □ Less than 1 cup □ 1 to 2 cups □ More than 2 cups 66. How often did you eat macaroni and cheese? □ NEVER (GO TO QUESTION 67) □ 1-6 times per year □ 2 times per week □ 7-11 times per year □ 3-4 times per week □ 1 time per month □ 5-6 times per week □ 2-3 times per month □ 1 time per day □ 1 time per week □ 2 or more times per day 66a. Each time you ate macaroni and cheese, how much did you usually eat? □ Less than 1 cup □ 1 to 1½ cups |
| Never added Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons 64e. How often was <b>syrup</b> added to your pancakes, waffles, or French toast? Almost never or never (GO TO QUESTION 65) About ⅓ of the time | More than 1½ cups 67. How often did you eat pasta salad or macaroni salad? NEVER (GO TO QUESTION 68) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week |
| ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |

Question 65 appears in the next column

| Over the <u>past 12 months</u> | <ol> <li>How often did you eat bagels or English<br/>muffins?</li> </ol> |
|---|---|
| 67a. Each time you ate pasta salad or macaroni | mullins? |
| salad, how much did you usually eat? | ☐ ☐ NEVER (GO TO INTRODUCTION TO QUESTION 70) |
| ☐ Less than ½ cup ☐ ½ to 1 cup ☐ More than 1 cup | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 1 time per week ☐ 2 or more times per day ☐ 2 or more times per day |
| 68. Other than the pastas listed in Questions 65, 66, and 67, how often did you eat pasta, spaghetti, or other noodles? | 69a. How often were the bagels or English muffins you ate whole wheat? |
| ☐ NEVER (GO TO QUESTION 69) | ☐ Almost never or never |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day | ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| ☐ 1 time per week ☐ 2 or more times per day 68a. Each time you ate pasta, spaghetti, or | 69b. Each time you ate bagels or English muffins, how many did you usually eat? |
| other noodles, how much did you usually eat? | ☐ Less than 1 bagel or English muffin ☐ 1 bagel or English muffin ☐ More than 1 bagel or English muffin |
| Less than 1 cup 1 to 3 cups More than 3 cups | 69c. How often was <b>margarine</b> (including low-fat) added to your bagels or English muffins? |
| 68b. How often did you eat your pasta, spaghetti, or other noodles with tomato sauce or spaghetti sauce made WITH meat? ☐ Almost never or never | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | 69d. How often was <b>butter</b> (including low-fat) added to your bagels or English muffins? ☐ Almost never or never |
| 68c. How often did you eat your pasta, spaghetti, or other noodles with tomato sauce or spaghetti sauce made WITHOUT meat? | ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| About ¼ of the time About ¼ of the time About ½ of the time Almost always or always | 69e. Each time margarine or butter was added to your bagels or English muffins, how much was usually added? |
| 68d. How often did you eat your pasta, spaghetti, or other noodles with margarine, butter, oil, or cream sauce? | |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | |
| <b>↓</b> | ↓ |

| Over the past 12 months | 70c. How often was mayonnaise or<br>mayonnaise-type dressing (including low- |
|---|---|
| 69f. How often was <b>cream cheese</b> (including low-fat) spread on your bagels or English muffins? | fat) added to the breads or rolls used for your sandwiches? |
| Almost never or never (GO TO INTRODUCTION TO QUESTION 70) About 1/4 of the time About 1/4 of the time About 1/4 of the time Almost always or always 69g. Each time cream cheese was added to your bagels or English muffins, how much was usually added? Less than 1 tablespoon 1 to 2 tablespoons More than 2 tablespoons | Almost never or never (GO TO QUESTION 70e) About 1/4 of the time About 1/4 of the time About 1/4 of the time About 1/4 of the time About 1/4 of the time Almost always or always 70d. Each time mayonnaise or mayonnaise-type dressing was added to the breads or rolls used for your sandwiches, how much was usually added? Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons |
| The next questions ask about your intake of breads other than bagels or English muffins. First, we will ask about bread you ate as part of sandwiches only. Then we will ask about all other bread you ate. 70. How often did you eat breads or rolls AS PART OF SANDWICHES (including burger and hot dog rolls)? (Please do not include fast food sandwiches.) NEVER (GO TO QUESTION 71) 1–6 times per year | → 70e. How often was margarine (including low-fat) added to the breads or rolls used for your sandwiches? Almost never or never |

Question 71 appears in the next column

| Over th | ne <u>past 12 months</u> | 71g. | Each time <b>cream cheese</b> was added to your breads or rolls, how much was usually added? |
|---|---|---|---|
| 71a. | Each time you ate breads or dinner rolls, NOT AS PART OF SANDWICHES, how much did you usually eat? | | Less than 1 tablespoon 1 to 2 tablespoons More than 2 tablespoons |
| | 1 slice or 1 dinner roll 2 slices or 2 dinner rolls More than 2 slices or 2 dinner rolls | | ow often did you eat jam, jelly, or honey on<br>gels, muffins, bread, rolls, or crackers? |
| 71b. | How often were the breads or rolls you ate white bread? | | NEVER (GO TO QUESTION 73) |
| | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About % of the time ☐ Almost always or always | | 1–6 times per year 7–11 times per year 1 time per month 2–3 times per week 3–4 times per week 5–6 times per week 1 time per day 1 time per day 2 or more times per day |
| 71c. | How often was margarine (including low-fat) added to your breads or rolls? | 72a. | Each time you ate <b>jam, jelly,</b> or <b>honey</b> , how much did you usually eat? |
| | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | | Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons wo often did you eat peanut butter or other |
| 71d. | How often was <b>butter</b> (including low-fat) added to your breads or rolls? | | t butter? NEVER (GO TO QUESTION 74) |
| | ☐ Almost never or never ☐ About 1/4 of the time ☐ About 1/2 of the time ☐ About 1/4 of the time ☐ Almost always or always | | 1–6 times per year 7–11 times per year 1 time per month 2–3 times per week 5–6 times per week 1 time per week 1 time per day 2 or more times per day |
| 71e. | Each time margarine or butter was added to your breads or rolls, how much was usually added? | 73a. | Each time you ate <b>peanut butter</b> or <b>other nut butter</b> , how much did you usually eat? |
| | □ Never added □ Less than 1 teaspoon □ 1 to 2 teaspoons □ More than 2 teaspoons | <b>↓</b> 74 Ho | ☐ Less than 1 tablespoon ☐ 1 to 2 tablespoons ☐ More than 2 tablespoons ow often did you eat roast beef or steak IN |
| 71f. | How often was cream cheese (including low-fat) added to your breads or rolls? | SA | ANDWICHES? NEVER (GO TO QUESTION 75) |
| | — Almost never or never (GO TO QUESTION 72) ☐ About ¼ of the time ☐ About ¾ of the time ☐ About ¾ of the time ☐ Almost always or always | | 1–6 times per year 7–11 times per year 1 time per month 2–3 times per week 1 time per month 1 time per week 2 or more times per day |
| <b>↓</b> | | ţ | |

| Over the past 12 months | 77. How often did you eat other cold cuts or |
|---|---|
| 74a. Each time you ate roast beef or steak IN SANDWICHES, how much did you usually eat? | luncheon meats (such as bologna, salami,<br>corned beef, pastrami, or others, including low-<br>fat)? (Please do not include ham, turkey, or<br>chicken cold cuts.) |
| ☐ Less than 1 slice or less than 2 ounces ☐ 1 to 2 slices or 2 to 4 ounces ☐ More than 2 slices or more than 4 ounces | ☐ NEVER (GO TO QUESTION 78) |
| 75. How often did you eat turkey or chicken COLD CUTS (such as loaf, luncheon meat, turkey ham, turkey salami, or turkey pastrami)? (We will ask about other turkey or chicken later.) NEVER (GO TO QUESTION 76) 1-6 times per year 2 times per week 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day | 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 5–6 times per week 1 time per month 1 time per day 1 time per week 2 or more times per day 77a. Each time you ate other cold cuts or luncheon meats, how much did you usually eat? Less than 1 slice 1 to 3 slices 1 to 4 times per week 3 dimes per week 3 dimes per week 5 times per week 1 times per week 1 time per day 1 time |
| ☐ 1 time per week ☐ 2 or more times per day 75a. Each time you ate turkey or chicken COLD CUTS, how much did you usually eat? ☐ Less than 1 slice ☐ 1 to 3 slices ☐ More than 3 slices ▼ 76. How often did you eat luncheon or deli-style ham? (We will ask about other ham later.) | |
| NEVER (GO TO QUESTION 77) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 76a. Each time you ate luncheon or deli-style ham, how much did you usually eat? Less than 1 slice 1 to 3 slices More than 3 slices More than 3 slices Almost never or never About ¼ of the time About ¼ of the time Almost always or always | 78. How often did you eat canned tuna (including in salads, sandwiches, or casseroles)? NEVER (GO TO QUESTION 79) 1–6 times per year |
| Question 77 appears in the next column | ↓ Question 79 appears on the next page 2 |

| Over the past 12 months 78c. How often was the canned tuna you ate | 80b. Each time you ate beef hamburgers or cheeseburgers from a FAST FOOD or | |
|---|---|--|
| prepared with mayonnaise or other<br>dressing (including low-fat)? | OTHER RESTAURANT, how much did you usually eat? | |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time | ☐ Less than 1 burger<br>☐ 1 burger<br>☐ More than 1 burger | |
| ☐ About ¾ of the time ☐ Almost always or always | 80c. How often did you have <b>cheeseburgers</b> rather than <b>hamburgers</b> ? | |
| 79. How often did you eat GROUND chicken or turkey? (We will ask about other chicken and turkey later.) □ NEVER (GO TO QUESTION 80) | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day | 81. How often did you eat beef hamburgers or cheeseburgers that were NOT FROM A FAST FOOD or OTHER RESTAURANT? | |
| ☐ 1 time per week ☐ 2 or more times per day | □ NEVER (GO TO QUESTION 82) | |
| 79a. Each time you ate GROUND chicken or turkey, how much did you usually eat? Less than 2 ounces or less than ½ cup 2 to 4 ounces or ½ to 1 cup More than 4 ounces or more than 1 cup 80. How often did you eat beef hamburgers or cheeseburgers from a FAST FOOD or OTHER RESTAURANT? | 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2 -3 times per month 1 time per day 2 or more times per day 2 or more times per day 2 or more times per day 4 times per week 2 or more times per day 5 times per week 2 or more times per day 4 times per week 5-6 times per week 5 | |
| NEVER (GO TO QUESTION 81) 1–6 times per year | □ Less than 1 patty or less than 2 ounces □ 1 patty or 2 to 4 ounces □ More than 1 patty or more than 4 ounces 81b. How often were these beef hamburgers or cheeseburgers made with lean ground beef? □ Almost never or never □ About ¼ of the time □ About ¾ of the time □ About ¾ of the time □ Almost always or always 82. How often did you eat ground beef in mixtures (such as meatballs, casseroles, chili, or meatloaf)? □ NEVER (GO TO QUESTION 83) □ 1-6 times per year □ 2 times per week □ 7-11 times per year □ 3-4 times per week □ 1 time per month □ 5-6 times per week | |
| | 2-3 times per month | |
| Over the past 12 months | 85. How often did you eat roast beef or pot roast? (Please do not include roast beef or pot roast in |
|---|---|
| 82a. Each time you ate ground beef in | sandwiches.) |
| mixtures, how much did you usually eat? | ─ □ NEVER (GO TO QUESTION 86) |
| ☐ Less than 3 ounces or less than ½ cup ☐ 3 to 8 ounces or ½ to 1 cup ☐ More than 8 ounces or more than 1 cup | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day |
| 83. How often did you eat hot dogs or<br>frankfurters? (Please do not include sausages<br>or vegetarian hot dogs.) | ☐ 1 time per week ☐ 2 or more times per day 85a. Each time you ate roast beef or pot roast, |
| ■ NEVER (GO TO QUESTION 84) | how much did you usually eat? |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day | ☐ Less than 2 ounces ☐ 2 to 5 ounces ☐ More than 5 ounces |
| ☐ 1 time per week ☐ 2 or more times per day | <ol> <li>How often did you eat steak (beef)?</li> <li>(Please do not include steak in sandwiches)</li> </ol> |
| 83a. Each time you ate hot dogs or frankfurters, how many did you usually eat? | NEVER (GO TO QUESTION 87) |
| Less than 1 hot dog 1 to 2 hot dogs More than 2 hot dogs | □ 1–6 times per year □ 7–11 times per year □ 1 time per month □ 2–3 times per month □ 2–3 times per month □ 1 time per day □ 1 time per day □ 2 or more times per day |
| 83b. How often were the hot dogs or frankfurters you ate <b>light</b> or <b>low-fat</b> ? | 86a. Each time you ate <b>steak</b> (beef), how much |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | did you usually eat? Less than 3 ounces 3 to 7 ounces More than 7 ounces |
| 84. How often did you eat <b>beef mixtures</b> (such as beef stew, beef pot pie, beef and noodles, or | 86b. How often was the steak you ate lean steak? |
| beef and vegetables)? NEVER (GO TO QUESTION 85) | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 1 time per day | ☐ About ¾ of the time ☐ Almost always or always ▼ 87. How often did you eat pork or beef spareribs? |
| 1 time per week 2 or more times per day | ☐ NEVER (GO TO QUESTION 88) |
| 84a. Each time you ate beef mixtures, how much did you usually eat? Less than 1 cup 1 to 2 cups More than 2 cups | ☐ 1–6 times per year ☐ 2 times per week ☐ 3–4 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |

Question 85 appears in the next column

| Over the past 12 months | 90. How often did you eat baked, broiled, roasted, |
|---|---|
| 87a. Each time you ate pork or beef spareribs, how much did you usually eat? | stewed, or fried chicken (including nuggets)? (Please do not include chicken in mixtures.) |
| Less than 4 ribs 4 to 12 ribs More than 12 ribs | □ NEVER (GO TO QUESTION 91) □ 1–6 times per year □ 2 times per week □ 7–11 times per year □ 3–4 times per week |
| 88. How often did you eat roast turkey, turkey cutlets, or turkey nuggets (including in | 1 time per month 5–6 times per week 2–3 times per month 1 time per day 2 or more times per day 2 or more times per day |
| sandwiches)? NEVER (GO TO QUESTION 89) | 90a. Each time you ate baked, broiled, roasted, stewed, or fried chicken (including nuggets), how much did you usually eat? |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day 88a. Each time you ate roast turkey, turkey | Less than 2 drumsticks or wings, less than 1 breast or thigh, or less than 4 nuggets 2 drumsticks or wings, 1 breast or thigh, or 4 to 8 nuggets More than 2 drumsticks or wings, more than 1 breast or thigh, or more than 8 nuggets |
| cutlets, or turkey nuggets, how much did<br>you usually eat? (Please note: 4 to 8 turkey<br>nuggets = 3 ounces.) | 90b. How often was the chicken you ate fried chicken (including deep fried) or chicken nuggets? |
| ☐ Less than 2 ounces ☐ 2 to 4 ounces ☐ More than 4 ounces ▼ | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time |
| 89. How often did you eat <b>chicken mixtures</b> (such as salads, sandwiches, casseroles, stews, or other mixtures)? | ☐ Almost always or always 90c. How often was the chicken you ate WHITE meat? |
| NEVER (GO TO QUESTION 90) 1–6 times per year | ☐ Almost never or never ☐ About 1/2 of the time ☐ About 1/2 of the time ☐ About 1/2 of the time ☐ Almost always or always 90d. How often did you eat chicken WITH skin? ☐ Almost never or never ☐ About 1/2 of the time |
| ☐ Less than ½ cup<br>☐ ½ to 1½ cups<br>☐ More than 1½ cups | ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| | 91. How often did you eat baked ham or ham steak? |
| | NEVER (GO TO QUESTION 92) |
| | ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week ☐ 2 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 or more times per day |
| <b>\</b> | <b>↓</b> |

| Over the past 12 months | 94a. Each time you ate liver or liverwurst, how |
|---|---|
| 91a. Each time you ate baked ham or ham steak, how much did you usually eat? Less than 1 ounce 1 to 3 ounces More than 3 ounces | much did you usually eat? Less than 1 ounce 1 to 4 ounces More than 4 ounces 95. How often did you eat bacon (including low-fat)? |
| 92. How often did you eat pork (including chops, roasts, and in mixed dishes)? (Please do not include ham, ham steak, or sausage.) NEVER (GO TO QUESTION 93) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 92a. Each time you ate pork, how much did you usually eat? Less than 2 ounces or less than 1 chop 2 to 5 ounces or 1 chop More than 5 ounces or more than 1 chop 93. How often did you eat gravy on meat, chicken, potatoes, rice, etc.? NEVER (GO TO QUESTION 94) 1–6 times per year 2 times per week 2 times per week | NEVER (GO TO QUESTION 96) 1–6 times per year |
| 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 1 time per month 1 time per day 1 time per week 2 or more times per day 93a. Each time you ate gravy on meat, chicken, potatoes, rice, etc., how much did you usually eat? Less than 1/2 cup 1/2 to 1/2 cup More than 1/2 cup More than 1/2 cup Well to 1/2 cup 1-6 times per year 2 times per week 1 time per month 1 time per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per day 2 or more times per day 2 or more times per day 2 or more times per day 3 or more times | NEVER (GO TO QUESTION 97) 1–6 times per year |

Question 95 appears in the next column

| Over the past 12 months | 100. How often did you eat fish sticks or other fried fish (not including shellfish)? |
|---|---|
| 97. How often did you eat fried shellfish (such as crab, lobster, shrimp)? | TIST (flot including shellish)? ☐☐ NEVER (GO TO QUESTION 101) |
| NEVER (GO TO QUESTION 98) 1–6 times per year 2 times per week 7–11 times per year 3-4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 97a. Each time you ate fried shellfish, how much did you usually eat? Less than 2 ounces 2 to 4 ounces More than 4 ounces More than 4 ounces NEVER (GO TO QUESTION 99) 1–6 times per year 2 times per week 1 time per month 5–6 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day 98a. Each time you ate shellfish that was NOT FRIED, how much did you usually eat? | 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 100a. Each time you ate fish sticks or other fried fish, how much did you usually eat? Less than 2 ounces or less than 1 fillet 2 to 7 ounces or 1 fillet More than 7 ounces or more than 1 fillet 101. How often did you eat other fish that was NOT FRIED (not including shellfish)? NEVER (GO TO INTRODUCTION TO QUESTION 102) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 101a. Each time you ate other fish that was NOT FRIED, how much did you usually eat? Less than 2 ounces or less than 1 fillet |
| Less than 1 ounce 1 to 4 ounces More than 4 ounces | 2 to 5 ounces or 1 fillet More than 5 ounces or more than 1 fillet |
| | Now think about all the meat, poultry, and fish you ate in the past 12 months and how they were prepared. 102. How often was oil, butter, margarine, or other fat used to FRY, SAUTE, BASTE, OR MARINATE any meat, poultry, or fish you ate? (Please do not include deep frying.) NEVER (GO TO QUESTION 103) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day |

Question 100 appears in the next column

| Over the past 12 months | 104c. Each time you ate <b>soup</b> , how much did you |
|---|---|
| 102a. Which of the following fats were regularly used to prepare your meat, poultry, or fish? (Mark all that apply.) | usually eat? ☐ Less than 1 cup ☐ 1 to 2 cups ☐ More than 2 cups |
| ☐ Margarine (including ☐ Corn oil ☐ low-fat) ☐ Canola or rapeseed oil ☐ Oil spray (such as Pam or others) ☐ Lard, fatback, or ☐ Other kinds of oils ☐ Oilve oil ☐ None of the above ☐ Oilve oil ☐ Corn oil ☐ Canola or rapeseed oil ☐ Oil spray (such as Pam or others) ☐ Other kinds of oils ☐ None of the above ☐ Oilve oil ☐ Oilve oilve oil | □ More than 2 cups 104d. How often were the soups you ate bean soups? □ Almost never or never □ About 1/4 of the time □ About 1/4 of the time □ About 1/4 of the time |
| 103. How often did you eat tofu, soy burgers, or soy meat-substitutes? | ☐ Almost always or always 104e. How often were the soups you ate cream |
| ☐ NEVER (GO TO QUESTION 104) | soups (including chowders)? |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 3–4 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 103a. Each time you ate tofu, soy burgers, or soy meat-substitutes, how much did you usually eat? | 104f. How often were the soups you ate <b>tomato</b> or <b>vegetable soups</b> ? ☐ Almost never or never |
| ☐ Less than ¼ cup or less than 2 ounces ☐ ¼ to ½ cup or 2 to 4 ounces ☐ More than ½ cup or more than 4 ounces | ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 104. Over the past 12 months, did you eat soups? NO (GO TO QUESTION 105) | 104g. How often were the soups you ate broth<br>soups (including chicken) with or without<br>noodles or rice? |
| r□ yes | ☐ Almost never or never |
| ↑ 104a. How often did you eat soup IN THE WINTER? □ NEVER | ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| ☐ 1–6 times per winter ☐ 2 times per week | 105. How often did you got nive? |
| 7-11 times per winter 3-4 times per week 5-6 times per week 1 time per month 1 time per week 2 or more times per day 2 or more times per day | 105. How often did you eat pizza? NEVER (GO TO QUESTION 106) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week |
| 104b. How often did you eat soup DURING THE REST OF THE YEAR? | ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |
| □ NEVER | |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | |

Question 105 appears in the next column

| Over the past 12 months | 108. How often did you eat biscuits? |
|---|---|
| 105a. Each time you ate <b>pizza</b> , how much did you<br>usually eat? | ☐ NEVER (GO TO QUESTION 109) |
| Less than 1 slice or less than 1 mini pizza 1 to 3 slices or 1 mini pizza More than 3 slices or more than 1 mini pizza | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day |
| 105b. How often did you eat pizza with pepperoni, sausage, or other meat? | 108a. Each time you ate <b>biscuits</b> , how many did you usually eat? |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | Fewer than 1 biscuit 1 to 2 biscuits More than 2 biscuits |
| 106. How often did you eat crackers? | 109. How often did you eat potato chips (including low-fat, fat-free, or low-salt)? |
| ☐ NEVER (GO TO QUESTION 107) | ☐ NEVER (GO TO QUESTION 110) |
| ☐ 1–6 times per year ☐ 7–11 times per year ☐ 1 time per month ☐ 2–3 times per month ☐ 1 time per week ☐ 2 times per week ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per day ☐ 2 times per week ☐ 2 or more times per day | ☐ 1–6 times per year ☐ 2 times per week ☐ 3–4 times per week ☐ 3 –4 times per week ☐ 5–6 times per week ☐ 1 time per week ☐ 1 time per day ☐ 2 or more times per day |
| 106a. Each time you ate <b>crackers</b> , how many did you usually eat? | 109a. Each time you ate <b>potato chips</b> , how much did you usually eat? |
| ☐ Fewer than 4 crackers ☐ 4 to 10 crackers ☐ More than 10 crackers | ☐ Fewer than 10 chips or less than 1 cup ☐ 10 to 25 chips or 1 to 2 cups ☐ More than 25 chips or more than 2 cups |
| 107. How often did you eat corn bread or corn muffins? | 109b. How often were the potato chips you ate fat-<br>free? (Please do not include reduced-fat<br>chips.) |
| NEVER (GO TO QUESTION 108) 1-6 times per year | Almost never or never About 1/4 of the time About 1/2 of the time About 1/2 of the time About 1/2 of the time Almost always or always 110. How often did you eat corn chips or tortilla chips (including low-fat, fat-free, or low-salt)? NEVER (GO TO QUESTION 111) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 2 or more times per day 2 or more times per day 3 description 3 description 3 description 4 time per week 2 or more times per day 3 description 4 time per week 2 or more times per day 3 description 4 time per week 2 or more times per day 3 description 4 time per week 2 or more times per day 3 description 4 time per week 2 or more times per day 4 times per week 4 times per w |

Question 108 appears in the next column

| Over the past 12 months | 113. How often did you eat peanuts, walnuts, seeds. or other nuts? |
|---|---|
| 110a. Each time you ate <b>corn chips</b> , how much did you usually eat? | NEVER (GO TO QUESTION 114) |
| ☐ Fewer than 10 chips or less than 1 cup ☐ 10 to 25 chips or 1 to 1½ cups ☐ More than 25 chips or more than 1½ cups 110b. How often were the corn chips or tortilla chips you ate fat-free? (Please do not include reduced-fat chips.) | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 1 time per day ☐ 1 time per week ☐ 2 or more times per day 113a. Each time you ate peanuts, walnuts, seeds, or other nuts, how much did you usually eat? |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | Less than ¼ cup ¼ to ½ cup More than ½ cup |
| 111. How often did you eat <b>popcorn</b> (including low-fat)? | 114. How often did you eat energy, high-protein, or<br>breakfast bars (such as Power Bars, Balance,<br>Clif, or others)? |
| ☐ NEVER (GO TO QUESTION 112) | ☐ NEVER (GO TO QUESTION 115) |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per week ☐ 2 or more times per day |
| 111a. Each time you ate <b>popcorn</b> , how much did you usually eat? | 114a. Each time you ate energy, high-protein, or breakfast bars, how much did you usually eat? |
| ☐ Less than 2 cups, popped<br>☐ 2 to 5 cups, popped<br>☐ More than 5 cups, popped | ☐ Less than 1 bar<br>☐ 1 bar<br>☐ More than 1 bar |
| 112. How often did you eat pretzels? | <b>♦</b><br>115. How often did you eat <b>yogurt</b> (NOT including<br>frozen yogurt)? |
| 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 112a. Each time you ate pretzels, how many did you usually eat? Fewer than 5 average twists 5 to 20 average twists More than 20 average twists | NEVER (GO TO QUESTION 116) 1-6 times per year |

| Over the past 12 months | 118. How often did you eat frozen yogurt, sorbet, or ices (including low-fat or fat-free)? |
|---|---|
| 115b. How often was the <b>yogurt</b> you ate <b>low-fat</b> or fat-free? | NEVER (GO TO QUESTION 119) |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 5–6 times per week ☐ 1 time per week ☐ 1 time per day ☐ 2 or more times per day |
| 116. How often did you eat cottage cheese (including low-fat)? | 118a. Each time you ate frozen yogurt, sorbet, or ices, how much did you usually eat? |
| NEVER (GO TO QUESTION 117) 1–6 times per year 2 times per week 7–11 times per year 3–4 times per week 1 time per month 5–6 times per week 2–3 times per month 1 time per day 1 time per week 2 or more times per day | Less than ½ cup or less than 1 scoop ½ to 1 cup or 1 to 2 scoops More than 1 cup or more than 2 scoops 119. How often did you eat ice cream, ice cream bars, or sherbet (including low-fat or fat-free)? |
| 116a. Each time you ate cottage cheese, how much did you usually eat? Less than ¼ cup ¼ to 1 cup More than 1 cup | NEVER (GO TO QUESTION 120) 1–6 times per year |
| 117. How often did you eat cheese (including low-fat; including on cheeseburgers or in sandwiches or subs)? | 119a. Each time you ate ice cream, ice cream bars, or sherbet, how much did you usually eat? |
| NEVER (GO TO QUESTION 118) 1–6 times per year | Less than ½ cup or less than 1 scoop ½ to 1½ cups or 1 to 2 scoops More than 1½ cups or more than 2 scoops 119b. How often was the ice cream you ate light, low-fat, or fat-free ice cream or sherbet? |
| 117a. Each time you ate cheese, how much did you usually eat? ☐ Less than ½ ounce or less than 1 slice ☐ ½ to 1½ ounces or 1 slice ☐ More than 1½ ounces or more than 1 slice | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 117b. How often was the cheese you ate low-fat or fat-free? | 120. How often did you eat <b>cake</b> (including low-fat or fat-free)? |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | NEVER (GO TO QUESTION 121) 1–6 times per year |
| <b>↓</b> | ▼ |

| Over the past 12 months | 123a. Each time you ate sweet muffins or dessert<br>breads, how much did you usually eat? |
|---|---|
| 120a. Each time you ate cake, how much did you usually eat? Less than 1 medium piece 1 medium piece More than 1 medium piece | Less than 1 medium piece 1 medium piece More than 1 medium piece 124. How often did you eat fruit crisp, cobbler, or strudel? |
| 121. How often did you eat cookies or brownies (including low-fat or fat-free)? | □ NEVER (GO TO QUESTION 125) |
| NEVER (GO TO QUESTION 122) | 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 1 time per day 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 1 time per week 2 or more times per day 124a. Each time you ate fruit crisp, cobbler, or strudel, how much did you usually eat? Less than ½ cup ½ to 1 cup More than 1 cup 125. How often did you eat pie? 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 1 time per month 1 time per day 1 time per week 2 or more times per day 125a. Each time you ate pie, how much did you usually eat? Less than ½ of a pie More than ½ of the time About ¾ of the time About ¾ of the time Almost always or always |

Question 124 appears in the next column

| Over the <u>past 12 months</u> | 128. How often did you eat eggs, egg whites, or egg |
|---|---|
| 125c. How often were the pies you ate cream, pudding, custard, or meringue pie? | substitutes (NOT counting eggs in baked<br>goods and desserts)? (Please include eggs in<br>salads, quiche, and soufflés.) |
| Almost never or never About 1/2 of the time About 1/2 of the time Almost always or always 125d. How often were the pies you ate pumpkin or sweet potato pie? Almost never or never About 1/2 of the time About 1/2 of the time About 1/2 of the time Almost always or always 125e. How often were the pies you ate pecan pie? | NEVER (GO TO QUESTION 129) 1-6 times per year |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | ☐ Almost never or never ☐ About 1/4 of the time ☐ About 1/4 of the time ☐ About 1/4 of the time ☐ Almost always or always |
| 126. How often did you eat chocolate candy? □ NEVER (GO TO QUESTION 127) | 128c. How often were the eggs you ate <b>regular</b> whole eggs? |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| 126a. Each time you ate <b>chocolate candy</b> , how much did you usually eat? | 128d. How often were the eggs you ate cooked in oil, butter, or margarine? |
| Less than 1 average bar or less than 1 ounce 1 average bar or 1 to 2 ounces More than 1 average bar or more than 2 ounces 127. How often did you eat other candy? | ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always |
| ☐ NEVER (GO TO QUESTION 128) | |
| ☐ 1–6 times per year ☐ 2 times per week ☐ 7–11 times per year ☐ 3–4 times per week ☐ 1 time per month ☐ 5–6 times per week ☐ 2–3 times per month ☐ 1 time per day ☐ 2 or more times per day | COCCE |
| 127a. Each time you ate other candy, how much did you usually eat? | |
| ☐ Fewer than 2 pieces ☐ 2 to 9 pieces ☐ More than 9 pieces | |

Question 128 appears in the next column

| Over the past 12 months | 130b. How often was the cold or iced tea you |
|---|---|
| 128e. How often were the eggs you ate part of egg salad? | drank presweetened with either sugar or<br>artificial sweeteners (such as Splenda,<br>Equal, Sweet'N Low or others)? |
| ☐ Almost never or never ☐ About ¼ of the time ☐ About ½ of the time ☐ About ¾ of the time ☐ Almost always or always | ☐ Almost never or never (GO TO QUESTION 131) ☐ About 1/4 of the time ☐ About 1/2 of the time ☐ About 1/4 of the time ☐ Almost always or always |
| 129. How many cups of coffee, caffeinated or decaffeinated, did you drink (including coffee drinks such as Latte, Mocha, Frappuccino, etc.)? NONE (GO TO QUESTION 130) Less than 1 cup per 5–6 cups per week month 1 cup per day 1–3 cups per month 2–3 cups per day 4–5 cups per day 2–4 cups per week 6 or more cups per day 129a. How often was the coffee you drank decaffeinated? Almost never or never About ½ of the time About ½ of the time Almost always or always 130. How many glasses, cans, or bottles of COLD or ICED tea, caffeinated or decaffeinated, did you drink? NONE (GO TO QUESTION 131) Less than 1 glass, can 5–6 glasses, cans or bottle per month 1–3 glasses, cans or bottles per week 2–4 glasses, cans or bottles per day 4–5 glasses, cans or bottles per week 2–4 glasses, cans or bottles per day 6 or more glasses, cans or bottles per day 130a. How often was the cold or iced tea you drank decaffeinated or herbal? Almost never or never About ½ of the time About ½ of the time About ¾ of the time Almost always or always | 130c. What kind of sweetener was added to your presweetened cold or iced tea most of the time? Sugar or honey |
| Question 131 appears in the next column | Question 133 appears on the next page<br>34 |

| Over the <u>past 12 months</u> | 133b. Each time <b>non-dairy creamer</b> was added to your coffee or tea, how much was usually |
|---|---|
| 132b. Each time sugar or honey was added to your<br>coffee or tea, how much was usually added? | used? |
| ☐ Less than 1 teaspoon ☐ 1 to 3 teaspoons ☐ More than 3 teaspoons | Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons |
| 132c. How often did you add artificial sweetener (such as Splenda, Equal, Sweet'N Low or others) to your coffee or tea? Almost never or never (GO TO QUESTION 133) About 1/4 of the time About 1/4 of the time | 133c. What kind of <b>non-dairy creamer</b> did you usually use? Regular powdered Low-fat or fat-free powdered Regular liquid Low-fat or fat-free liquid |
| ☐ About ¾ of the time<br>☐ Almost always or always | 133d. How often was cream or half and half<br>added to your coffee or tea? |
| 132d. What kind of artificial sweetener did you usually use? | ☐ Almost never or never (GO TO QUESTION 133f) ☐ About ¼ of the time ☐ About ½ of the time |
| ☐ Equal or aspartame ☐ Sweet'N Low or saccharin ☐ Splenda or sucralose | ☐ About % of the time ☐ Almost always or always |
| Herbal extracts or other kind 132e. Each time artificial sweetener was added to your coffee or tea, how much was usually added? Less than 1 packet or less than 1 teaspoon | 133e. Each time cream or half and half was added to your coffee or tea, how much was usually added? Less than 1 tablespoon 1 to 2 tablespoons More than 2 tablespoons |
| ☐ 1 packet or 1 teaspoon ☐ More than 1 packet or more than 1 teaspoon | →133f. How often was milk added to your coffee or tea? |
| 133. Over the <u>past 12 months</u> , did you add whiteners (such as cream, milk, or non-dairy creamer) to your tea or coffee? | ☐ Almost never or never (GO TO QUESTION 134) ☐ About 1/4 of the time ☐ About 1/4 of the time ☐ About 1/4 of the time |
| NO (GO TO QUESTION 134) | ☐ Almost always or always |
| YES 133a. How often was non-dairy creamer added to your coffee or tea? | 133g. Each time milk was added to your coffee or tea, how much was usually added? Less than 1 tablespoon |
| Almost never or never (GO TO QUESTION 133d) About ¼ of the time About ½ of the time | ☐ 1 to 3 tablespoons☐ More than 3 tablespoons☐ |
| ☐ About % of the time ☐ Almost always or always | 133h. What kind of <b>milk</b> was usually added to your coffee or tea? |
| ▼ Question 133d appears in the next column Question 134 appears on the next page | Question 134 appears on the next page |
| Queenon 134 appears on the next page | quodion 134 appears on the next page |

Question 134 appears on the next page

| Over the past 12 months | 137. Over the past 12 months, did you eat |
|---|---|
| 134. How often was <b>sugar</b> or <b>honey</b> added to foods you ate? (Please do not include sugar in coffee, tea, other beverages, or baked goods.) | mayonnaise or mayonnaise-type dressing? NO (GO TO QUESTION 138) T YES |
| NEVER (GO TO INTRODUCTION TO QUESTION 135) 1-6 times per year 2 times per week 7-11 times per year 3-4 times per week 1 time per month 5-6 times per week 2-3 times per month 1 time per day 1 time per week 2 or more times per day 134a. Each time sugar or honey was added to foods you ate, how much was usually added? Less than 1 teaspoon 1 to 3 teaspoons More than 3 teaspoons More than 3 teaspoons The following questions are about the kinds of margarine, mayonnaise, sour cream, cream cheese, and salad dressing that you ate. If possible, please check the labels of these foods to help you answer. | 137a. How often was the mayonnaise you ate light, low-fat or fat-free? Almost never or never About ½ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time Almost always or always 138. Over the past 12 months, did you eat sour cream? NO (GO TO QUESTION 139) YES 138a. How often was the sour cream you ate light, low-fat, or fat-free? Almost never or never About ¼ of the time About ¾ of the time About ¾ of the time About ¾ of the time Almost always or always |
| NO (GO TO QUESTION 136) YES 135a. How often was the margarine you ate light, low-fat, or fat-free (stick or tub)? Almost never or never About ½ of the time About ½ of the time Almost always or always 136. Over the past 12 months, did you eat butter? NO (GO TO QUESTION 137) YES 136a. How often was the butter you ate light or low-fat? Almost never or never About ½ of the time About ½ of the time About ¾ of the time Almost always or always | 139. Over the past 12 months, did you eat cream cheese? NO (GO TO QUESTION 140) YES 139a. How often was the cream cheese you ate light, low-fat, or fat-free? Almost never or never About ½ of the time About ½ of the time About ¾ of the time Almost always or always |

Question 140 appears on the next page 36

Question 137 appears in the next column

| Over the <u>past 12 months</u> | 143. Over the <u>past month</u> , which of the following foods did you eat AT LEAST THREE TIMES? |
|---|---|
| 140. Over the <u>past 12 months</u> , did you eat salad dressing? | (Mark all that apply.) |
| NO (GO TO INTRODUCTION TO QUESTION 141) YES 140a. How often was the salad dressing you ate light, low-fat or fat-free? Almost never or never About ½ of the time About ¾ of the time About ¾ of the time About ¾ of the time About ¾ of the time Summarize your usual intake of vegetables and fruits. Please do not include salads, potatoes, or | Avocado, guacamole Cheesecake Chocolate, fudge, or butterscotch toppings or syrups Chow mein noodles Croissants Dried apricots Egg rolls Granola bars Hot peppers Jell-O, gelatin Mangoes Milkshakes or ice-cream sodas Choesecake Oysters Oysters Pickles or pickled vegetables or fruit Plantains Pork neck bones, hock, head, feet Pudding or custard Veal, venison, lamb Whipped cream, regular Whipped cream, substitute None None |
| juices. | followed any type of vegetarian diet? |
| 141. Over the past 12 months, how many servings of vegetables (not including salad or potatoes) did you eat per week or per day? Less than 1 per week | NO (GO TO INTRODUCTION TO QUESTION 145) YES 144a. Which of the following foods did you TOTALLY EXCLUDE from your diet? (Mark all that apply.) Meat (beef, pork, lamb, etc.) Poultry (chicken, turkey, duck) Fish and seafood Eggs Dairy products (milk, cheese, etc.) |

| pills or other supplements. 145. Over the past 12 months, did you take any | ninese last questions are about the vitamins, minerals, or herbal supplements you took that are NOT part of a One-a-day-, Theragran-, or Centrum-type of multivitamin. |
|---|---|
| multivitamins, such as One-a-Day-, Theragran-,<br>Centrum-, or Prenatal-type multivitamins (as pills,<br>liquids, or packets)? | Over the past 12 months |
| ── NO (GO TO INTRODUCTION TO QUESTION 147) | Tums or Rolaids? |
| liquids, or packets)? NO (GO TO INTRODUCTION TO QUESTION 147) YES 146. How often did you take One-a-day-, Theragran-, Centrum- or Prenatal-type multivitamins? Less than 1 day per month 1-3 days per month 1-3 days per week 4-6 days per week Every day 146a. Did your multivitamin usually contain minerals (such as iron, zinc, etc.)? NO YES Don't know 146b. For how many years have you taken multivitamins? Less than 1 year 1-4 years 5-9 years 10 or more years 146c. Over the past 12 months, did you take any vitamins, minerals, or other herbal supplements other than your multivitamin? NO Thank you very much for completing this questionnaire! Because we want to be able to use all the information you have provided, we would greatly appreciate it if you would please take a moment to | 147. How often did you take Antacids such as Tums or Rolaids? NEVER (GO TO QUESTION 148) Less than 1 day per month 1-3 days per week 4-6 days per week Every day 147a. When you took Antacids such as Tums or Rolaids, about how many tablets or lozenges did you take in one day? Less than 1 1 2 3 4 or more Don't know Don't know 147b. Was your antacid usually "extra strength"? NO YES Don't know 147c. For how many years have you taken Antacids such as Tums or Rolaids? Less than 1 year 1-4 years 5-9 years 10 or more years 148. How often did you take Calcium (with or without Vitamin D) (NOT as part of a multivitamin in Question 146 or antacid in Question 147)? NEVER (GO TO QUESTION 149) Less than 1 day per month |
| review each page making sure that you: Did not skip any pages and Crossed out the incorrect answer and circled the correct answer if you made any changes. | ☐ 1-3 days per month ☐ 1-3 days per week ☐ 4-6 days per week ☐ Every day |
| ☐ YES (GO TO INTRODUCTION TO QUESTION 147 | |

Introduction to Question 147 appears in the next column

| Over the past 12 months | 150. How often did you take Vitamin C (NOT as part of a multivitamin in Question 146)? |
|---|---|
| 148a. When you took Calcium, about how much elemental calcium did you take in one day? (If possible, please check the label for elemental calcium.) Less than 500 mg 500–599 mg 600–999 mg 1,000 mg or more Don't know | NEVER (GO TO QUESTION 151) Less than 1 day per month 1-3 days per month 4-6 days per week Every day 150a. When you took Vitamin C, about how much |
| DOPT KNOW 148b. Did your Calcium usually contain Vitamin D? NO | did you take in one day? Less than 500 mg 500-999 mg 1,000-1,499 mg 1,500-1,999 mg 2,000 mg or more Don't know 150b. For how many years have you taken Vitamin C? Less than 1 year 1-4 years 5-9 years 10 or more years NEVER (GO TO INTRODUCTION TO QUESTION 152) Less than 1 day per month 1-3 days per week 4-6 days per week 4-6 days per week Every day 151a. When you took Vitamin E, about how much did you take in one day? Less than 400 IU 400-799 IU 800-999 IU 1,000 IU or more Don't know 151b. For how many years have you taken Vitamin E? Less than 1 year 1-4 years 5-9 years 10 or more years |

Question 150 appears in the next column

| Over the past 12 months | |
|---|---|
| The last two questions ask you about other supplements you took more than once per week. | Thank you <u>very much</u> for completing this questionnaire! Because we want to be able to use all the information you have provided. |
| 152. Please mark any of the following single supplements you took more than once per week (NOT as part of a multivitamin in Question 147): | we would greatly appreciate it if you would<br>please take a moment to review each page<br>making sure that you: |
| □ B-6 □ Occu-vite/Eye health □ B-complex □ Potassium □ B-12 □ Selenium □ Beta-carotene □ Vitamin A □ Folic acid/folate □ Vitamin D □ Magnesium □ Zinc | <ul> <li>Did not skip any pages and</li> <li>Crossed out the incorrect answer and circled the correct answer if you made any changes.</li> </ul> |
| 153. Please mark any of the following herbal,<br>botanical, or other supplements you took<br>more than once per week. | |
| □ Chondroitin □ Ginseng □ Coenzyme Q-10 □ Glucosamine/ □ Echinacea chondroitin □ Energy supplements □ Peppermint □ Fish oil/omega 3's □ Probiotics □ Flaxseed/oil □ Saw palmetto □ Garlic □ Soy supplement □ Ginger □ Sports supplements □ Ginkgo biloba □ St. John's wort □ Other | |

### 26 Appendix O: Automated Self-Administered 24-hour Recall (ASA24)



# Overview of the ASA24™ Respondent Web sites and Considerations Related to Data Security and Participant Confidentiality

Extensive evidence has demonstrated that 24-hour dietary recalls provide the highest quality, least biased dietary data. Traditional 24-hour recalls, however, are expensive and impractical for large-scale research because they rely on trained interviewers and multiple administrations to estimate usual intakes. As a result, researchers often make use of food frequency questionnaires, which are less expensive but contain substantial error.

To address this challenge, investigators at NCI created the Automated Self-administered 24-hour Recall (ASA24™) system, a freely-available, web-based tool that enables multiple automated self-administered 24-hour recalls. ASA24™ was developed under contract with Westat®, a social science research firm located in Rockville, MD, and builds on the Food Intake Recording Software System (FIRSSt) developed by Dr. Tom Baranowski of the Baylor College of Medicine. An External Working Group provided advice about the needs and interests of potential users.

ASA24™ consists of a Respondent Web site used to collect recall data and a Researcher Web site used to manage study logistics and obtain data analyses. Two Respondent Web sites are currently available in English and Spanish: ASA24™-2014 and ASA24™-Kids-2014. This document provides an overview of the methodology and main features of the ASA24™ Respondent sites, as well as information on security of the data collected and protections to the confidentiality of the participants of studies that make use of ASA24™. Images of the main Respondent site screens are also included.

#### ASA24™ Respondent Web site Methodology

Respondents are guided through the 24-hour recall interview using a modified version of the USDA's Automated Multiple-Pass Method (AMPM). The steps in the interview process include:

- 1. Meal-based Quick List
- 2. Meal Gap Review
- 3. Detail Pass
- 4. Forgotten Foods
- 5. Final Review
- 6. Last Chance
- 7. Usual Intake Question
- 8. Supplement Module (if selected by the researcher)

#### Meal-based Quick List

During the first pass of the interview, respondents are asked to provide a list of the foods and drinks consumed at each meal occasion for one of two possible 24-hour time periods, depending on the preference of the researcher: yesterday, from midnight to midnight; or, the past 24-hours based on the time of participant login. Respondents are able to browse food group categories to find their foods and drinks or search for a particular item. Foods and drinks



reported at each meal are recorded in the My Foods and Drinks panel within the instrument. This initial step is called the meal-based Quick List. In addition to selecting an eating occasion (e.g., breakfast, lunch, snack), respondents are also prompted to specify the time of the occasion before reporting the foods and drinks consumed. The researcher can opt to collect additional contextual information including where meals were eaten, television and computer use during meals, and whether the meal was eaten alone or with others.

#### Meal Gap Review

Once respondents finish creating their My Foods and Drinks list at the end of the Quick List step, they are asked if they consumed anything during any 3-hour gaps between eating occasions, and, for the midnight to midnight version, between midnight and the first eating occasion, and between the last eating occasion and midnight. A response of "Yes" to any gap will return the respondent to the Quick List to add the appropriate food(s) or drink(s).

#### **Detail Pass**

Respondents are asked for details about the foods and drinks they recorded during the Quick List, including form (e.g., raw), preparation methods (e.g., grilled or roasted), the amount eaten, and any additions (e.g., sugar, coffee cream, salad dressing). Researchers can also opt to ask the source (grocery store, farmer's market, vending machine, etc.) of each food reported.

#### **Forgotten Foods**

Following the Detail Pass, a pop-up window appears with questions probing about the consumption of commonly forgotten foods and drinks (e.g., snack foods, fruits, vegetables, cheese, water, coffee, tea). Respondents must check either "Yes" or "No" for each food or drink probed. For any "Yes" response, the respondent will be returned to the Quick List to add the forgotten item(s).

#### **Final Review**

Respondents are prompted to review all of the foods and drinks reported for the intake day, and make edits and add meals, foods and drinks as necessary.

#### **Last Chance**

After the Final Review, a pop-up screen appears with an option to add food or drink items if respondents have still forgotten any. Again, respondents will be brought back to the Quick List to add more items; otherwise, they will move forward to the final question in the food and drink module.

#### **Usual Intake Question**

The final question asks: Was the amount of food that you are yesterday more than usual, usual, or less than usual? This question probes whether this was a typical day's intake.



#### Supplement Module (if selected by the researcher during study set-up)

Respondents are asked to provide information about the type and dose of supplements consumed by completing a Quick List, a Detail Pass, and a Final Review. Supplements include vitamins, minerals, and other supplements including prescription supplements. Respondents are able to browse supplement categories (e.g., Multi-Vitamin/Mineral, Calcium products, Herbal/Botanicals) or search for a particular supplement. The supplements included are based on those reported in the National Health and Nutrition Examination Survey.

#### ASA24™ Respondent Web Site Features

The ASA24™ Respondent Web site guides the participant through the completion of a 24-hour recall for the previous day, from midnight to midnight, using a dynamic user interface. The instrument:

- provides an animated guide and audio and visual cues to instruct participants and enhance use in low-literacy populations and with children (with options to turn off the guide and/or the audio);
- · asks respondents to report eating occasion and time of consumption;
- includes optional modules to query where meals were eaten, whether meals were
  eaten alone or with others, and television and computer use during meals;
- · flows as per modified USDA Automated Multiple-Pass Method (AMPM) 24-hour recall;
- allows respondents to report foods and drinks by browsing by category or searching from a list of food and drink terms derived from the National Health and Nutrition Examination Survey (NHANES);
- asks detailed questions about food preparation, portion size, and additions so that food
  codes from USDA's Food and Nutrient Database for Dietary Studies (FNDDS) can be
  assigned; it also provides an option to query respondents about food source;
- · uses images to assist respondents in reporting portion size;
- allows the respondent to add or modify food and drink choices at multiple points during the interview;
- includes an optional module to query dietary supplement intake based on supplements reported in NHANES;
- · is available in English and Spanish; and
- is compliant with Section 508 of the 1973 Rehabilitation Act.

The Respondent Web sites do not provide any direct feedback to respondents. Instead, researchers can obtain analysis files from the Researcher Web site and contact respondents with any findings they choose to share.

#### Data Security and Protections to Confidentiality of Participants using ASA24™

Researchers using ASA24<sup>™</sup> do not provide the National Cancer Institute, Westat (the research firm that developed and maintains ASA24<sup>™</sup>), or the ASA24<sup>™</sup> system with any identifying data for participants of their studies. Rather, researchers specify an identifier for each respondent and download system-generated usernames and encrypted passwords that they provide to respondents so that they may access the application.



ASA24™ also does not collect any identifying data directly from respondents. However, IP address information is accessed for the purpose of routing information between the server and the respondent's computer—often the IP address is that of the user's Internet Service Provider (ISP). IP addresses are not stored or tracked by ASA24™. However, logs of connections are kept in the hosting environment for audit trail purposes. This information is not mined in any way but would be available if there were a legal obligation to release it.

Response data are secured at the hosting site using industry standard security controls, including firewalls and encryption. All data entered into ASA24™ at the respondent's computer is encrypted by the internet browser (e.g., Internet Explorer, Firefox) before they are transmitted to our servers using Secure Socket Layer (SSL) Technology. SSL allows for the authentication of the sending and receiving computers.

Only a particular study's investigator(s) and the ASA24 $^{\rm m}$  operations team can access response data. Access is gained through usernames and strong passwords.

#### ASA24 Respondent Web site Screen Shots

Figure 1: The participant can choose to complete ASA24 in either English or Spanish.



Figure 2: An introductory screen prompts the participant to report everything that she or he had to eat or drink yesterday.





Figure 3: The main ASA24 screen is used to select foods and drinks to be added to My Foods and Drinks during the Quick Pass, and to add details and make changes. The animated guide provides an overview of the main ASA24 screen and gives instructions on how to report all foods, drinks, and supplements (if the optional Supplement Module is selected by the researcher) consumed either from midnight to midnight yesterday or for the past 24 hours, starting at the time of login (depending on the researcher preferences).



Figure 4: The meal details screen collects information on the eating occasion and time, and displays optional modules that can be selected by the researcher to query where meals were eaten, whether meals were eaten alone or with others, and television and computer use during meals. This is the first step in the meal-based Quick List.





Figure 5: Participants complete the Quick List pass by browsing categories or searching for the foods and drinks they consumed. The food and drink terms are based on the National Health and Nutrition Examination Survey.



Figure 6: The foods and drinks that the participant reports during the Quick List are displayed in the My Foods and Drinks panel on the right of the main screen.





Figure 7: After the participant reports the foods and drinks consumed yesterday and selects Done entering all meals and snacks, the Meal Gap Review is displayed.



Figures 8a-c: The detail pass prompts the participant to report the details of each food and drink, including the specific type or how it was prepared, anything added to it, and the amount that was consumed.

Figure 8a.





Figure 8b.



Figure 8c.





Figure 9: Once the Detail Pass is complete, the Final Review begins. The participant can make changes to the details for a given food or drink and add more foods and drinks if necessary.



Figure 10: The forgotten foods pass queries the participant about frequently forgotten foods.

Responding yes to one or more categories will result in a prompt to add the forgotten foods or drinks.





Figure 11: The final question in the food and drink module asks the participant whether the amount of foods and drinks consumed yesterday was usual.



Figure 12: If the Supplement Module is selected by the researcher during study set up, the participant will also be asked about the supplements, if any, that he or she took either from midnight to midnight yesterday or for the past 24 hours, starting at the time of login (depending on researcher preferences).





Figure 13: The Supplement Module collects details about each supplement reported.



Figure 14: Once the participant completes the food and drink module and the supplement module, if selected by the researcher during study set up, his or her responses are saved in the secure database and he or she can exit ASA24. Only the researcher(s) who are registered to that study and the ASA24 operations team can access the response data.



### 27 Appendix P: qADAM Questionnaire

#### Questions Used as Part of the qADAM Questionnaire

- How would you rate your libido (sex drive)?
   (terrible) 2(poor) 3(average) 4(good) 5(excellent)
- 2. How would you rate your energy level?

  1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- How would you rate your strength/endurance?
   1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- How would you rate your enjoyment of life?
   1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- How would you rate your happiness level?
   1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- 6. How strong are your erections?(1= extremely weak 5= extremely strong)1 2 3 4 5
- How would you rate your work performance over the past 4 weeks?
   1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- How often do you fall asleep after dinner?
   1(never) 2(1-2/week) 3(3-4/week) 4(5-6/week) 5(every night)
- How would you rate your sports ability over the past 4 weeks?
   1(terrible) 2(poor) 3(average) 4(good) 5(excellent)
- 10. How much height have you lost? 1(2" or more) 2(1.5-1.9") 3(1-1.4") 4(0.5-0.9") 5(none-0.4")

The quantitative ADAM questionnaire. Int J Impot Res. 2010 Jan; 22(1): 20-24.

O Mohamed, <sup>1</sup> R E Freundlich, <sup>1</sup> H K Dakik, <sup>1</sup> E D Grober, <sup>2</sup> B Najari, <sup>3</sup> L I Lipshultz, <sup>1</sup> and M Khera<sup>1,\*</sup>

Published online 2009 Aug 6. doi: 10.1038/ijir.2009.35

PMCID: PMC2834355

# 28 Appendix Q: Psychosexual Daily Questionnaire

| Please rate your overall level of sex | ual desire today by circling the appropriate nu | mber below: |
|---|---|---|
| | 0-1-2-3- | 4 — 5 — 6 — 7<br>very high |
| | very low | very riigir |
| 2. Please rate highest level of enjoym | ent or pleasure of any sexual activity that you | experienced today. |
| | pationI sexual fantasies) and/or (b) with a part | ner (e.g., kissing, intercourse) by circling |
| the appropriate number below. (a) Without a partner | | |
| (a) Williout a partier | 0 — 1 — 2 — 3 — 4 —<br>none | —5 ——6 ——7<br>very high enjoyment/pleasure |
| (b) With a partner | 0 — 1 — 2 — 3 — 4 —<br>none | 567<br>very high enjoyment/pleasure |
| (c) Please indicate if partner is availab | le yes no | |
| <ol><li>Please rate your mood by writing the solution is not at all true;</li><li>indicates that the d</li></ol> | | w. For each item 0 indicates that the descriptor |
| | not at all true 0 — 1 — 2 — 3 — 4 | 5 6 7 very true |
| (a) Angry? | (d) Full of pep/energetic? | (g) Friendly? |
| (b) Alert? | (e) Sad or Blue? | (h) Nervous? |
| (c) Irritable? | (f) Tired? | (i) Well/good? |
| 4. For all of the items below check yes | s if you have experienced (or are experiencing | j) today, otherwise check no. |
| Yes No | Yes No | Yes No |
| (a) sexual daydreams | (e) orgasm | (i) masturbation |
| (b) anticipation of sex | (f) flirting (by others toward you) | (j) night spontaneous erection |
| (c) sexual interactions with partner | (g) ejaculation | (k) day spontaneous erection |
| (d) flirting (by you) | (h) intercourse | (I) erection in response to sexual activity |
| Answer the following two question | s only if you experienced an erection as | shown in No. 4. j-l above. |
| 5. If you experienced an erection toda<br>(make a reasonable estimate): | ay, indicate the % full erection that you experi- | enced by circling the appropriate number below |
| %= 0 | 10 20 30 40 50 60 70 | 80 90 100 |
| If you experienced an erection toda<br>number below: | ay, indicate whether it was maintained for a sa | atisfactory duration by circling the appropriate |
| not satisfact | ory 0 — 1 — 2 — 3 — 4 — 5 — | 6 — 7 very satisfactory |

A Simple Self-Report Diary for Assessing Psychosexual Function in Hypogonadal Men Ka Kui Lee<sup>1,2</sup>, Nancy Berman<sup>3</sup>, Gerianne M. Alexander<sup>4</sup>, Laura Hull<sup>1</sup>, Ronald S. Swerdloff<sup>1</sup> and Christina Wang<sup>1,\*</sup>

Article first published online: 2 JAN 2013 DOI: 10.1002/j.1939-4640.2003.tb02728.x

| 29 A | opendix R: Sun Exposure and Benaviour Inventory (SEBI V2) |
|---|---|
| Subje | ct ID: Survey Administration: 1 <sup>st</sup> / 2 <sup>nd</sup> Date: |
| For <b>e</b> a | ach question listed, please check off the ONE answer that is the BEST response to the question. |
| A sur | <b>aburn</b> is defined as skin redness or pain which lasts at least <u>one day after sun exposure</u> . |
| 1. Wh | ich of the following BEST describes your skin's reaction to one hour of summer sun without reen? |
| | Always burns, never gets darker /tans (Very light |
| | skin, Caucasian) Always burns at first, but sometimes gets darker/tans with continued sun exposure (Light skin, Caucasian) |
| | Sometimes burns first, but always gets darker/tans with continued sun exposure (Medium skin, usually Caucasian) |
| | Rarely burns, gets darker/tans easily with sun exposure (Olive skin, may be of many race/ethnic backgrounds) |
| (Brown | Never burns, skin gets darker with sun exposure n to dark-brown skin, may be of many race/ethnic backgrounds) |
| | Never burns, no darkening of skin color with sun exposure (Black skin, African ancestry) |
| | w many times <u>in your life</u> have you had a <b>SUNBURN?</b> None |
| | 1-10 |
| | 11-20<br>More than 20 |
| 3. Ho | w many times in your life have you had a SUNBURN that BLISTERED? |
| | None<br>1-3 |
| | 4-10<br>More than 10 |
| | IVIOIC MAII IV |
| 4. Ho | w many times in your life have you used a tanning bed/booth/sunlamp? |
| | None<br>1-10 |
| | 11-50 |
| | 51-100 |

| | 101-500<br>More than 500 | | | | | |
|---|---|---|---|---|---|---|
| 5. Hav<br>□ | re you lived in an area with a <b>significantly s</b><br>Yes<br>No | sunnier clim | ate than Bo | oston for <u>six</u> | months or | more? |
| IF yes, | what city/state or country? | | F | or how long | <u>;</u> ? | |
| | Less than 5 years<br>6-10 years<br>11-20 years<br>More than 20 years | | | | | |
| 6. Plea | se rate your <u>lifetime</u> sun exposure | | | | | |
| | | Very low | Low | Moderate | High | Very high |
| TOT | AL sun exposure | , | | | | <u> </u> |
| | sure from OUTDOOR RECREATION | | | | | |
| Expo | sure from your <b>JOB</b> | | | | | |
| | ich of the following <b>BEST</b> describes your adult (18-25)? Light skin, red or red-blonde hair Light skin, blonde or light brown hair Light skin, brown or black hair Medium-tone skin, brown or black hair Brown skin, dark brown or black hair Black skin, dark brown or black hair | NATURA | <b>L</b> skin and | hair color w | hen you w | ere a |
| 8. Wha | at is your eye color? Brown Blue, green, gray Hazel (brownish green) | | | | | |
| Now, | think about your current lifestyle to answ | ver the rema | nining ques | tions. | | |
| 9. Thii | nk about what you do when you are outsion | de <u>during th</u> | e summer o | on a warm su | ınny day. | |
| | | Never | Rarely | Sometimes | Often | Always |
| How | often do you wear SUNSCREEN? | | | | | |

| SLEI | EVES that cover you | ur shoulders? | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | often do you wear a | | | | | | | |
| | face, ears, and neck | | | | | | | |
| How | often do you stay in | the SHADE or | | | | | | |
| | ER AN ÚMBRÉLL | | | | | | | |
| How | often do you wear SI | UNGLASSES? | | | | | | |
| | · · | | l . | | | l. | | I |
| | nat is the Sun Protec | ction Factor (SPF) | of the su | nscreen | that you us | se most ofte | en'? | |
| | Less than SPF 15 | | | | | | | |
| | SPF 15 or higher | | | | | | | |
| | Don't know | | | | | | | |
| | I don't use sunscre | een | | | | | | |
| 11 Do | as vous sunsaraan h | ove both IIVA on | a HWD n | mataatia | m? | | | |
| | es your sunscreen h<br>Yes | ave dom U V A and | <b>и () у Б</b> р | iolectic | )11 <b>(</b> | | | |
| | No | | | | | | | |
| | □ Don't know | | | | | | | |
| | I don't use sunscre | | | | | | | |
| | low often do you sp | end time <u>in the sur</u> | n or in a t | anning | bed/booth | in order to | get a <u>tan</u> | or to feel |
| good | | | | | | | | |
| | Never | | | | | | | |
| | Rarely | | | | | | | |
| | Sometimes | | | | | | | |
| | Often | | | | | | | |
| | Always | | | | | | | |
| 13. H | lave you been tan in | the last 12 month | s? | | | | | |
| | Yes | | | | | | | |
| | No | | | | | | | |
| | 1 0111011111111111111111111111111111111 | <b>.</b> | | | | | | |
| | n the <b>SUMMER</b> (Ju | | on avera | ge, hov | v many hou | ırs per day | are you c | <u>utside</u> |
| betwo | een 10am and 4pm? | | | | | | | |
| | | Less than 1hour | 1hour | 2hour | s 3hours | 4hours | 5hours | 6 hours |
| On W | VEEKDAYS | | | | | | | |
| | day-Friday) | | | | | | | |
| | VEEKENDS | | | 1 | | | | |
| | rday and Sunday) | | | | | | | |
| Sara | | l | l | 1 | | 1 | I | 1 |

15. In **NON-SUMMER** months (September to May), on average, how many hours per day are you **outside** between 10am and 4pm?

How often do you wear a **SHIRT WITH** 

| | Less than 1hour | 1hour | 2hours | 3hours | 4hours | 5hours | 6 hours |
|---|---|---|---|---|---|---|---|
| On WEEKDAYS | | | | | | | |
| (Monday-Friday) | | | | | | | |
| On WEEKENDS | | | | | | | |
| (Saturday and Sunday) | | | | | | | |

### **Investigator Signature of Agreement**

The Eunice Kennedy Shriver National Institute of Child Health and Human Development

Reproductive Medicine Network

| <u>Title:</u> Males, Antioxidants, and Infertility (MOXI) Tr | ial |
|---|---|
| Version: 4.0 | |
| Principal Investigator: | |
| I, [Insert PI's name] , the Principal Investigator for agree to conduct this study in accordance with this protocol o site. | [Insert Institute Name], hereby certify that I have read an<br>n behalf of all RMN Investigators and research staff from m |
| I will conduct the clinical study as described and will adher<br>25, Part 46, Good Clinical Practices (GCP), International C<br>Declaration of Helsinki. I have read and understood the co | Conference on Harmonisation (ICH), and the |
| The signature of the investigator below indicates acceptance o investigator commitments as outlined in Form FDA 1572, State | |
| Principal Investigator's Signature | <br>Date |
| Printed Name | Date |

### DATA AND SAFETY MONITORING BOARD (DSMB) CHARTER

### Males, Antioxidants, and Infertility (MOXI) Trial

### 1. Purpose and Responsibilities of the DSMB

The members of the Data and Safety Monitoring Board (DSMB) identified in this Charter for the MOXI study are responsible for safeguarding the interests of study participants, assessing the safety and efficacy of all study procedures, and shall monitor the overall conduct of the MOXI trial. This Committee will serve as an independent advisory group to the Director of NICHD, and is required to provide recommendations about starting, continuing, and stopping the MOXI trial.

This Committee is responsible for identifying mechanisms to complete various tasks that will impact the safety and efficacy of all study procedures, and overall conduct. The table below identifies the key areas where oversight is necessary and the ways in which the Committee for the MOXI trial will complete those tasks.

| Basic Responsibility of DSMB | Method DSMB for MOXI will use to complete task |
|---|---|
| Familiarize themselves with the study protocol | · Review study protocols and informed consent forms. |
| Monitor adverse events | <ul> <li>Adverse Event: Review quarterly progress reports prepared by the DCC on behalf of RMN.</li> <li>Serious Adverse Events: Review report submitted by the DCC on behalf of RMN within one week of the event if life threatening or fatal, or within two weeks otherwise. The DSMB will submit a report of their review to the NICHD Committee Coordinator within 7 business days if the SAE is life threatening or fatal, or within two weeks otherwise.</li> </ul> |
| Monitor data quality | · Conduct interim evaluations of the data. |
| Oversee participant recruitment and enrollment | Review interim progress reports prepared by the DCC on behalf of RMN. |
| Develop an understanding of the Study's risks and benefits | <ul> <li>Review study protocols and related literatures.</li> <li>Review interim reports of subject accrual and outcome measures provided by the DCC.</li> <li>Assess the need to perform further in-depth evaluation of the benefits and risks of the study after reviewing each report.</li> </ul> |
| Ensure the proper reporting occurs | Review and approve the meeting and reporting schedule listed in Section 5 of this DSMB charter. |
## 2. Contacts

#### **NICHD**

Louis DePaolo, PhD, Program Officer Charisee Lamar, PhD, MPH, RRT, Committee Coordinator Esther Eisenberg, MD, MPH, Project Scientist

#### **Data Coordination Center (DCC)**

Heping Zhang, PhD, DCC Principal Investigator Hao Huang, MD, DCC Data Manager

The Data Manager at the DCC will prepare and review the DSMB reports prior to submission to the DSMB, and will not be blind to treatment condition.

#### **Lead Investigator**

Anne Z. Steiner, MD, MPH

## 3. DSMB Members, Organizational Chart, & Communications

#### **Members**

The DSMB for the MOXI trial is comprised of the members listed in the table below. In addition, their high level roles and responsibilities are identified in the table.

| Name of Member | Role on DSMB | High Level Responsibilities |
|---|---|---|
| Frank Witter, MD | Chair of DSMB Voting member | <ul> <li>Chair the DSMB discussion and prepare written recommendations to NICHD.</li> <li>Ensure the safety of study subjects, the integrity of the research data.</li> <li>Provide NICHD with advice on the ethical and safe progression of studies conducted in the RMN.</li> <li>Advises on research design issues, data quality and analysis, and research participant protection for each prospective and on-going study.</li> </ul> |
| Robert E. Brannigan, MD | Voting member | Ensure the safety of study subjects, the integrity of the research data. Provide NICHD with advice on the ethical and safe progression of |
| Rev. Phillip Cato, PhD | Voting member | |
| PonJola Coney, MD | Voting member | <ul> <li>studies conducted in the RMN.</li> <li>Advises on research design issues, data quality and analysis, and research participant protection for each prospective and on-going study.</li> </ul> |
| Lurdes Y.T. Inoue, PhD | Voting member | |
| Stacey A. Missmer, ScD | Voting member | |

Only Voting members for this DSMB may attend closed sessions for this Committee. In addition, only Voting members will have access to unblinded data points for this Committee.

#### **Organizational Chart**

The following diagram illustrates the relationship between the DSMB and other entities in the MOXI study.



#### Communication

Communication for members of this DSMB will be primarily through the NICHD Program Office and, where applicable, the Data Coordination Center (DCC). Investigators from the MOXI study will not communicate directly with DSMB members about the study, except when making presentations or responding to questions at DSMB meetings or during scheduled conference calls.

# 4. Conflict of Interest and Compensation

It is extremely important that all members of the DSMB state any real or apparent conflicts of interests at the onset of the study. Members of the DSMB shall read the NICHD Clinical Research Guidance Document regarding Conflict of Interest and provide their signed summary of any COI for the study, at its onset, to the NICHD Committee Coordinator, Dr. Charisee Lamar. A table summarizing any COI within the DSMB is provided in the Appendix.

Prior to each meeting, all members of the RMN DSMB will have an opportunity to state whether they have developed any new conflicts of interest since the meeting. As a new COI is identified it must be documented in the table in the Appendix and a new signed summary of the COI should be provided to the NICHD Committee Coordinator. The Coordinator will forward the COI documentation to the DCC for record-keeping purposes.

If a new conflict is reported, the Coordinator and staff will determine if the conflict limits the ability of the DSMB member to participate in the discussion.

All DSMB members will be compensated for their role in supporting the committee. Compensation will include an honorarium for meeting attendance and any travel costs.

## 5. Meeting Schedule

DSMB meetings will be conducted quarterly. However, the DSMB may hold a meeting at any time in accordance with their mission. The NICHD Committee Coordinator will notify the DCC of any change in schedule.

# 6. Blinding

All summaries for DSMB reports will be presented in a blinded fashion, unless specified by the DSMB Chair.

# 7. Report Schedule and Content

The type of reports (full or brief) is indicated below, followed by a description of the contents of each type.

| DSMB Report | Report Submission Date | Type of Report |
|-------------|------------------------|----------------|
| 1. | tbd | Brief |
| 2. | tbd | Brief |
| 3. | tbd | Brief |
| 4. | tbd | Full |
| 5. | tbd | Brief |
| 6. | tbd | Full |
| 7. | tbd | Brief |
| 8. | tbd | Full |
| 9. | tbd | Brief |
| 10. | tbd | Full |
| 11. | tbd | Brief |

## **Brief DSMB reports** will include the following summaries:

- overall actual versus projected enrollment accrual
- overall randomization update
- overall study drop-out rate
- serious adverse events
- primary outcome measures update

### Full DSMB reports will include the following summaries:

• recruitment update (number screened) overall and by site

- enrollment update (enrolled defined as randomized to a treatment) overall and by site
- accrual status including actual enrollment compared to projections overall and by site
- randomization update (i.e., number assigned to each treatment arm)
- study drop-out rate for enrolled patients (number, reason, time point) overall and by site)
- pre-specified subset of baseline demographic data for enrolled patients
- safety data, adverse events, and serious adverse events
- number of case report forms expected
- number/percentage of expected case report forms received overall and by site
- number of case report forms that are query clean
- primary outcome measures update

## References

NIH Policy for Data and Safety Monitoring http://grants.nih.gov/grants/guide/notice-files/NOT98-084.html

Guidance on Reporting Adverse Events to Institutional Review Boards for NIH-supported Multi-center Clinical Trials <a href="http://grants.nih.gov/grants/guide/notice-files/not99-107.html">http://grants.nih.gov/grants/guide/notice-files/not99-107.html</a>.

# Appendix: Summary of COI within the DSMB

| DSMB Member Name | Date Submitted<br>Signed COI | Was a COI<br>Identified? | Will the Member Remain part of the Committee? |
|---|---|---|---|
| Robert E. Brannigan, MD | | | |
| Rev. Phillip Cato, PhD | | | |
| PonJola Coney, MD | | | |
| Lurdes Y.T. Inoue, PhD | | | |
| Stacey A. Missmer, ScD | | | |
| Frank Witter, MD | | | |





# **Reproductive Medicine Network**

Funded by Eunice Kennedy Shriver NICHD

# **Conflict of Interest Statement**

# Males, Antioxidants, and Infertility (MOXI) Trial

| ĺ, | assuming the role of |
|---|---|
| | (insert role, for example: DSMB member) |
| for the | |
| | (insert project or study name) |
| agree to th | e following statements. |
| □ I agree to | 0: |
| : | protect the interests and safety of study participants; uphold the integrity of the research process including data collection and analysis to be as free from bias and preconception as I am able; adhere to the highest scientific and ethical standards, to comply with all relevant regulations and to eliminate or disclose, during my involvement with the proposed clinical research project, any real or apparent conflicts of interest. |
| In addition | ı: |
| financial ir<br>monetary v | that I, my spouse or dependent children, or organization with which I am connected, do/does not have any nterest in the study, where financial interested is defined by the DHHS, as anything of value, including but not limited to, salary or other payments for services (for example, consulting fees or |
| | ; equity interests (for example, stocks, stock options or other ownership interests); and intellectual property |

The financial interest term does not include various items which can be found in The Federal regulation, PHS, DHHS Part 50--Policies of General Applicability; Subpart F- Responsibility of Applicants for Promoting Objectivity in Research for Which PHS Funding Is Sought.

For Federal employees, financial interests that are allowable and require disclosure are:

Financial Interest Disclosure: Financial interest that require disclosure are stock holdings in pharmaceutical firms, medical device manufacturers, and biotechnology companies

Allowable Financial Interests: In a company that produces a product that is being evaluated by a study, participants may hold up to \$15,000 of stock: and up to an aggregate of \$25,000 of the stock of that company and its competitors who produce that (or a similar) product. As an alternative to individual stock holdings, participants may hold up to an aggregate of \$50,000 in sector mutual funds-including pharmaceutical/health care sectors.

For holdings in excess of these *de minimus* levels, a conflict of interest analysis needs to be conducted by NIH regarding the holding, the company producing the product being evaluated under the study, and its competitors, and, if a conflict

exists, could lead to the need to withdraw from the study.

I agree to not withhold any data related to the \_\_\_\_\_\_ study or to interfere with the analysis or publication of the study's results.

I will not engage in activities that could be viewed as real or apparent COI, including but not limited to:

having a part-time, full-time, paid, or unpaid employee status of any organizations that are: (a) involved in the study under review; (b) whose products will be used or tested in the study under review, or whose products or services would be directly and predictably affected in a major way by the outcome of the study;

being an officer, member, owner, trustee, director, expert advisor, or consultant of such organizations;

being a current collaborator or associate of the principal investigator (applicable to potential members of data safety and monitoring boards);

having a scientific interest beyond that required for my role, where scientific interest is defined as having

influence over the protocol, the study design, conducting the study analysis or any reporting related to the

investigation (applicable to potential members of data safety and monitoring boards).

#### 8.2 Data Collection and Management (including quality assurance/compliance measures)

#### 8.2.1 Data Entry and Forms

Case Report Forms (CRFs) will be developed as the protocol is developed. They will also be implemented in a Web-based Oracle data management system. The Web data entry forms will be similar to the paper forms with the same questions. However, the Web forms usually have more flexibility than the paper forms, such as pull-down menus.

#### 8.2.2 Features of Data Management System

Features of the data management system include study definition; different types of data entry (including double entries and complete audit trail); forms control; query capture, reporting, and resolution; dictionary coding of Adverse Events (AEs) and medical terms; and clinical data review Tools; and prepares data and CRF images to FDA e-Submission Standards. The enduser/reporting/ad hoc query front-end uses a standard Web browser, so that data entry and browsing can be done from any machine with Internet access, without purchase of special software. Login to this system will be through a secured Web server with the security under the protection of Yale Center for Clinical Investigations.

#### 8.2.3 Data Security

A data server and Web server will be used. The data server will be managed by YNHH IT center and the website two servers will be separated and managed by Forte Research Systems. The web server will be accessible through a secured login, but the data server can only be accessed through the web server. For security purposes, no login to the data server will be permitted, and access to the back end is limited to authorized individuals. PHI, including patient names and addresses, will be locked and secured at the participating sites, and data will be linked through a unique identification number, which will be assigned after a patient is screened or enrolled. Access will be limited to authorized individuals (21 CFR 11.10(d)). Each user of the system will have an individual account. The user will log into the account at the beginning of a data entry session, input information (include changes) on the electronic record, and log out at the completion of the data entry session. The system will be designed to limit the number of log-in attempts and record unauthorized access log-in attempts. Individuals will work only under their own access key, and not share these with others. The system will not allow an individual to log onto the system to provide another person access to the system. Access key Users will be asked to change their passwords at established intervals commensurate with a documented risk assessment. This plan has been adapted from the guidelines for computerized systems used in clinical investigations established by the U.S. Department of Health and Human Services Food and Drug Administration.

#### 8.2.4 Data Quality Control

#### Competency to perform procedure/tests in the protocol

The site PI will be responsible for ensuring that study related tests are performed by competent personnel. The criteria for determination of competency may vary between sites in the study.

biostatistics, epidemiology, infertility, gynecology, andrology and ethics. The NICHD Committee Coordinator is responsible for scheduling regular committee meetings, recording all meeting minutes and summarizing the committee recommendations for the Steering Committee and NICHD. Steering Committee members are prohibited from attending closed sessions of the DSMB. Open sessions may be attended by Steering Committee members or Chairperson when requested by NICHD and the DSMB.

The DSMB has quarterly teleconferences to review Network randomized trial protocols with respect to ethical and safety standards, monitors the safety of on-going clinical trials, monitors the integrity of the data with respect to original study design, and provides advice on study conduct. The DSMB periodically monitors data quality, including protocol adherence and adverse events. As outlined in the protocols, the DSMB will conduct interim evaluations of the data. It may recommend protocol modifications based on concern for subject welfare and scientific integrity.

#### 8.5 Reporting

Administrative Reports will be prepared by the DCC - which include monthly and quarterly reports on accrual, data quality and study compliance - and presented to the Steering Committee and DSMB. Statistical reports include reports to the SC, DSMB and AB from the data analysis, and special reports for scientific manuscripts.

Statistical Reports will be generated in SAS. Reports are provided for DSMB reviews, and for final analysis of study results in preparation for scientific publications. The content of the interim reports will be very complete, and will serve as the template for the final report of each study, which in turn will form the basis of the publication of the results. Our proposed reports to the DSMB would include the following: a protocol description and history; accrual rates; site performance in terms of accrual; eligibility; protocol violations; data accuracy and minority representation; patient characteristics by treatment and site; and the rate of adverse experiences.

## 8.6 Obligation of the Investigator

#### 8.6.1 IRB Review

The site PI is responsible for submitting the approved protocol and consent form to the IRB for review. The IRB must approve all aspects of the study as detailed in the protocol, including the patient informed consent form. It is anticipated that there will be minor site-specific changes in the consent form. The IRB must periodically review the status of the study at appropriate intervals not exceeding one year. The site PI will also be responsible for submitting revisions to the protocol to the IRB, as directed by the DCC, and promptly communicating serious adverse events that result during the study, to both the local IRB and the DCC. After the approval, the informed consent and IRB approval (or amendment) letters must be forwarded to the DCC.

#### 8.6.2 Maintenance/Retention of site records

In order to comply with Good Clinical Practice (GCP) requirements, the investigators must maintain the master patient log that identifies all patients entered into the study for a period of

## 9 RMN Publications Policy

The publications policy proposes guidelines for publications that originate from our collaborative Reproductive Medicine Network. Decisions concerning publications shall be determined by consensus (majority vote) of the collaborating Principal Investigators (or designees) noted below as the "Network." This policy is designed to promote prompt, exact, quality publications and presentations of Network studies with appropriate academic recognition of those with significant contributions. Protocols are classified into three types: 'Main Study' (which may include major and minor publications), "Ancillary Study', and 'Pilot Study'. Additionally, there may be publications from concepts or ideas generated by the RMN ("Related Publications") or from other groups utilizing RMN data and/or specimens, known as "Outside Studies" (those utilizing data and/or specimens from the RMN studies). Abstract submissions to national meetings will also follow the publications policy below. The progress of publications (including presentations) will be a standing agenda note on all teleconferences and meetings. The Steering Committee will make the final decision regarding disputes with respect to analysis request approval, prioritization, presentation, authorship and/or manuscript submission.

#### 9.1 Main Study

A Main Study is a Network study designed prospectively by an investigator independent of other studies. Generally, that investigator becomes Lead Investigator of the protocol and Chair of the Protocol Subcommittee. At the end of each Main Study, a primary analysis resulting in the primary manuscript and a number of secondary analyses is produced based on the research questions stated in the protocol. The Protocol Subcommittee Chair is the primary author of the primary analysis. A Main Study can generate major (related to the major hypotheses) and minor publications (relating to secondary hypotheses).

#### 9.1.1 Major Publications

A major publication is defined as one reporting results of the major hypotheses tested. (For example: Does hMG/IUI increase cyclic fecundity in couples with unexplained or male factor infertility?)

#### **a.** Authorship

Publications will include the names of investigators from each RMU and the DCC rather than merely identify the "Reproductive Medicine Network". Each RMU and the DCC will have up to two authors per publication, ordinarily the PI and the Co-PI, but this may at times involve another investigator who has contributed to the study at his/her site, in lieu of the PI or Co-PI. The Principal Investigator at each RMU will be responsible for submitting the names of the two authors from that unit and designating them as either the primary and secondary authors of the unit. No more than 2 authors may represent a RMN site. An ancillary site (such as a SCCPIR) may only have 1 investigator. The Steering Committee Chair and NICHD Project Scientist will be authors. Occasionally, additional authors, both within and outside the RMN

It is anticipated that there will be up to 18-25 authors per major manuscript. The authorship order of the RMUs and outside sites will be based upon subject recruitment, data accuracy and promptness of data report according to the chart below:

Data accuracy will be ranked according to the rate of missing or false data entries/randomized subjects at each site. Inquiries that show data was accurately entered will not count against this rate of data inaccuracy. Each site's PI will be responsible for documenting the contributions to the study of that site's authors. In the event the journal editor requires fewer authors even after written documentation of the authors' contribution has been provided, the Steering Committee will vote on the authorship order which will include at a minimum the Lead Investigator and PI of the DCC (or his/her designee) in the positions listed above with the authorship order ending with the footnoted statement "for the Reproductive Medicine Network". The other authors will be referenced in the footnote and listed in the title page.

#### d. Acknowledgement Section

The acknowledgement section will include other investigators and study personnel who contributed substantially to the study by site, as well as members of the Advisory Board and the Data and Safety Monitoring Board. The designation will list the initials of the individuals followed by their highest degree (e.g. C. L. Gnatuk, J.A. Ober, R.N., etc.).

Significant contributions include but are not limited to protocol review, initiation and participation at each site, subject recruitment and enrollment, study conduct, data analysis, and preparation of the manuscript.

#### 9.1.2 Minor Publications

Minor studies are defined as those in which the hypotheses would not be the main elements of Network studies, but in which the study data base would be utilized to test secondary hypotheses. (One example would be testing whether metformin use spares the dose of clomiphene resulting in lower dose needs.) Ideas for "minor studies" will, in general, be proposed by a single individual, who would direct all efforts leading to publication and representation. The results from minor studies would be handled similarly to those from major studies. The "Protocol" is defined as the Concept Protocol/study design of the hypothesis resulting in the publication.

Authorship will follow the Major Publications guidelines above with the exception that the individual leading the minor study would be the first author, followed by the ranked primary RMN investigators involved in developing the Concept Protocol. The Lead Investigator of the minor publication can propose additional investigators who contributed to the study, whose inclusion in the authorship will be voted on by the Steering Committee (majority vote of SC required for inclusion in authorship). Centers may wish to withdraw inclusion from authorship of publications

of minor studies in which only data are contributed, and this will be the decision of the individual site (RMU) PI.

#### 9.2 Ancillary Study

An Ancillary Study is an observational study, conducted as a supplement to a Main Study. By definition, an Ancillary Study involves all or a subset of patients enrolled in a Main Study. An Ancillary Study does not involve any additional participants. To be defined as an Ancillary Study, there must be a need for collection of additional data not already collected in the Main Study. An Ancillary Study may also be designed by another Network investigator, who would serve as the lead investigator and primary author of the paper. Ancillary Studies may be a "single-center" or "multi-center".

A "single-center" Ancillary Study is a study in which all data are collected, stored and analyzed at a single center. The center bears the additional cost of such a study. The study requires approval of the Main Study Protocol Subcommittee and the Steering Committee. The center conducting the study is responsible for the analysis and reporting of the results. Abstracts and manuscripts resulting from data from the single-center Ancillary Study are not subject to the RMN Publications Policies.

A "multi-center" Ancillary Study is defined as one for which data or material (such as specimens) are collected at more than one center, or additional funds for conduct of the study are provided by the NICHD RMN and the DCC provides data analysis. Multi-center Ancillary Studies require the approval of the Main Study Protocol Subcommittee and the Steering Committee.

Authorship will be as per Major Publications above with the exception that the individual leading the Ancillary Study and writing the paper would be the first author, followed by ranked RMN primary investigators, etc. A center not participating in the Ancillary Study would not receive authorship unless by majority vote of the Steering Committee.

#### 9.2.1 Publication Policy on Ancillary Papers

#### <u>Authorship</u>

- 1. RMN will be included as the group author and the acknowledgement will define the entire RMN roster as provided by all PIs.
- 2. The SC Chair, the NICHD Project Scientist, and all PIs will be co-authors upfront. The order will be recommended by the lead author(s).
- 3. Based on the ICJME statement for authorship (http://www.icmje.org/ethical\_1author.html), anyone who makes additional contributions that are documented and substantive will be co-authors. Correcting typos and making grammar suggestions may be below the threshold.
- 4. The responsibilities of the lead authors and the DCC: